

### STATISTICAL ANALYSIS PLAN

Protocol Number P261-401

Protocol Number P261-401

Protocol Number P261-401

Pate of P

Date of P A Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Intranasal Midazolam (USL261) in the Outpatient **Treatment of Subjects with Seizure Clusters** ARTEMIS-1: Acute Rescue Therapy in Epilepsy with Midazolam

Date of Plan: April 14, 2017 (Final v2.9)

### STATISTICAL ANALYSIS PLAN

### Final 2.9

A Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Intranasal Midazolam (USL261) in the Outpatient **Treatment of Subjects with Seizure Clusters** ARTEMIS-1: Acute Rescue Therapy in Epilepsy with Midazolam Intranasal Spray-1



## TABLE OF CONTENTS

| LIST OF A | ABBREVIATIONS | 7 |
|---|---|---|
| 1. | INTRODUCTION | 8 |
| 2. | STUDY DESIGN | 8 |
| 2.1. | General Study Design and Plan | 8 |
| 2.1.1. | Screening. | (10) |
| 2.1.2. | Test-Dose Phase | 10 |
| 2.1.3. | Comparative Phase | 10 |
| 2.2. | Randomization and Method of Treatment Assignment | 11 |
| 2.3. | Study Procedures | 12 |
| 3. | STUDY OBJECTIVES | 15 |
| 3.1. | Primary Efficacy Objective | 15 |
| 3.2. | Secondary Efficacy Objectives | 15 |
| 3.3. | Exploratory Efficacy Objectives | 15 |
| 3.4. | Safety Objectives | 15 |
| 3.5. | Pharmacokinetic Objectives | 16 |
| 4. | STUDY DESIGN General Study Design and Plan Screening. Test-Dose Phase Comparative Phase Randomization and Method of Treatment Assignment Study Procedures STUDY OBJECTIVES. Primary Efficacy Objective Secondary Efficacy Objectives Exploratory Efficacy Objectives Safety Objectives Pharmacokinetic Objectives ANALYSIS POPULATIONS Screened Population Safety Population Randomized Population Randomized Safety Population Randomized Safety Population | 16 |
| 4.1. | Screened Population | 16 |
| 4.2. | Safety Population. | 16 |
| 4.3. | Randomized Population | 16 |
| 4.4. | Randomized Safety Population | 17 |
| 4.5. | Modified Intent-to-Treat Population (mITT) | 17 |
| 4.6. | Per Protocol Population | 17 |
| 4.7. | Pharmacokinetic Population | 17 |
| 5. | GENERAL STATISTICAL CONSIDERATIONS | |
| 5.1. | Vevel of Significance | 18 |
| 5.2. ann <sup>O</sup> | Handling of Missing Data | 18 |
| 5.1.<br>5.2.<br>5.3<br><b>5.3.1.</b> | Interim Analyses | 19 |
| 5.3.1. | Early Success | 19 |
| 5.3.2. | Early Futility | 20 |
| 5.3.3. | Early Termination not related to Success or Futility | 20 |
| 5.3.4. | Logistical details for interim analyses | 20 |

| 5.4. | Examination of Subgroups. | 21 |
|---|---|---|
| 5.5. | Data Collected from Unscheduled Visits. | 21 |
| 6. | DESIGN OPERATING CHARACTERISTICS | 21 |
| 6.1. | Simulation Scenarios | 21 |
| 6.2. | Operating Characteristics | 22 |
| 7. | STATISTICAL ANALYSIS | 22 |
| 7.1. | Subject Disposition | 23 |
| 7.2. | Protocol Deviations | 23 |
| 7.3. | Demographics and Baseline Characteristics | 24 |
| 7.4. | Medical and Surgical History | 24 |
| 7.5. | Prior and Concomitant Medications | 25 |
| 7.6. | Analyses of Efficacy Endpoints | 26 |
| 7.6.1. | Primary Efficacy Endpoint | 26 |
| 7.6.1.1. | Derivation of Treatment Success Endpoint | 27 |
| 7.6.1.2. | Analysis of the Primary Endpoint | 28 |
| 7.6.2. | Secondary Efficacy Endpoints | 29 |
| 7.6.2.1. | Operating Characteristics STATISTICAL ANALYSIS Subject Disposition Protocol Deviations Demographics and Baseline Characteristics Medical and Surgical History Prior and Concomitant Medications Analyses of Efficacy Endpoints Primary Efficacy Endpoint Derivation of Treatment Success Endpoint Analysis of the Primary Endpoint Secondary Efficacy Endpoints Proportion of Subjects with Recurrence of Seizure(s) Beginning 10 Minutes after Administration of Double-Blind Study Drug to 4 Hours after Double-Blind Study Drug Administration | 29 |
| 7.6.2.2. | Time to Next Seizure with a Start Time >10 Minutes after Double-Blind Study Drug Administration | 30 |
| 7.6.3. | Exploratory Efficacy Analyses | 30 |
| 7.6.3.1. | Proportion of Subjects with Recurrence of Seizure(s) Beginning 10 Minutes after Study Drug Administration to 24 Hours after Study Drug Administration | |
| 7.6.3.2. | Return to Full Baseline Functionality within 24 Hours after Study Drug Administration (as determined by the caregiver) | 31 |
| 7.6.3.3. | Analyses for Subjects Receiving 2 Doses of Study Drug | 31 |
| 7.6.3.4 | Treatment Success of all Dose of Study Drug | 32 |
| 7.6.3.4<br>7.6.3.5. | Subject and Caregiver Outcome Assessments | 33 |
| .7.7. | Safety Analyses | 34 |
| 7.7.1. | Adverse Events (AEs) | 34 |
| 7.7.1.1. | Pre-treatment AEs | 34 |
| 7.7.1.2. | Treatment-emergent AEs (TEAEs) | 34 |

| 7 <b>.</b> 7 <b>.2</b> . | Observer's Assessment of Alertness/Sedation (OAA/S) | 37 |
|---|---|---|
| 7.7.2.1. | Composite Score. | 37 |
| 7.7.2.2. | Sum Score | 37 |
| 7.7.2.3. | Pharmacodynamic (PD) Parameters | 37 |
| 7.7.3. | Requirement for Unscheduled ER or EMS Visit | 38 |
| 7.7.4. | Brief Smell Identification Test (B-SIT; United States only) | 38 |
| 7.7.5. | Columbia-Suicide Severity Rating Scale (C-SSRS) | 38 |
| 7.7.5.1. | Suicidal Ideation | 39 |
| 7.7.5.2. | Suicidal Behavior | 39 |
| <b>7.7.6.</b> | Suicidal Ideation Suicidal Behavior Physical, Nasal, and Complete Neurological Examinations Laboratory Parameters Vital Signs and Oxygen Saturation Electrocardiogram (ECG) OTHER PLANNED ANALYSES Pharmacokinetic (PK) Analyses Pharmacokinetic/Pharmacodynamic Variables and Analyses | 40 |
| 7.7.7. | Laboratory Parameters | 40 |
| <b>7.7.8.</b> | Vital Signs and Oxygen Saturation | 40 |
| <b>7.7.9.</b> | Electrocardiogram (ECG) | 41 |
| 8. | OTHER PLANNED ANALYSES | 41 |
| 8.1. | Pharmacokinetic (PK) Analyses | 41 |
| 8.2. | Pharmacokinetic/Pharmacodynamic Variables and Analyses | 42 |
| 9. | CHANGES TO THE PLANNED ANALYSIS | 42 |
| 10. | MOCK TABLES, FIGURES, AND DATA LISTINGS | 44 |
| 11. | REFERENCES | |
| APPEND | IX 1. POTENTIALLY CLINICALLY SIGNIFICANT LABORATORY VALUES | 45 |
| APPEND | | |
| APPEND | IX 3. LIST OF AE TERMS OF SPECIAL INTEREST | 49 |
| | LIST OF TABLES Schedule of the Study Procedures | |
| Table 1: | Schedule of the Study Procedures | 12 |
| Table 2: | Required p-values for declaring success according to Lan-DeMets Pocock Approximation Spending Function | |
| Table 3: | Study Phases Start and End. | 22 |
| Table 4: | Classification of Prior and Concomitant Medications | 25 |
| Table 5: | Search Strategy for AESI | 36 |
| Table 6: | Pharmacodynamic Parameters | 38 |
| Table 7: | Suicidal Ideation Scores. | 39 |

| Table 8: | Potentially Clinically Significant Laboratory Values | 45 |
|---|---|---|
| Table 9: | Listing of Non-Enzyme Inducing AEDs | 46 |
| Table 10: | List of Enzyme Inducing AEDs | 46 |
| Table 11: | Abuse-related AEs (MedDRA Preferred Term) | 49 <sub>ill</sub> ere |
| Table 12: | AEs Related to Acute Central Respiratory Depression (SMQ) | 516 <sup>5</sup> |
| Table 13: | AEs Related to Acute Central Respiratory Depression (SMQ) | 60 |
| Table 14: | AEs Related to Route of Administration-Respiratory Disorders NEC (HLT) | 68 |
| Table 15: | AEs Related to Route of Administration-Upper Respiratory Tract Disorders (HLT) (Exclude Infections). | 77 |
| Table 16: | (HLT) (Exclude Infections). AEs Related to Taste and Smell Disorders (SMQ). | 92 |
| Table 17: | AEs Related to Depression and Suicidality/Self-Injury-Depression (SMQ) (Exclude Suicide/Self-Injury) | 93 |
| Table 18: | AEs Related to Depression and Suicidality/Self-Injury-Suicide/Self-Injury (SMQ) | |
| | LIST OF FIGURES | |
| Figure 1: | Study Design | 9 |
| Figure 2: | Study Design Disposition Flow Chart Possible Scenarios for Seizure Data Start and Stop Times Within the 6 Hour | 23 |
| Figure 3: | Period Following the First Dose of Study Drug Are Displayed Below, Along | |
| | with the Treatment Success Endpoint Derivation (Assuming No Second Dose was given) | 28 |
| This document cannot | | |
| This do | | |

Statistical Analysis Plan for Protocol No.: P261-401

### LIST OF ABBREVIATIONS

**Definition** Abbreviation μL

**ACLS** 

ΑE **AED** 

ATC **B-SIT** 

C-SSRS

**CFR** 

CI

CRO DSMB

**ECG** 

**EMS** 

ER ET **GCP** 

**IAMC** 

**ICF** 

**ICH** 

ΙN

IRB IRT ITI

ITIO

ITT

Legally acceptable representative LAR

MCS Mental Health Component Score (SF-12v2)

Midazolam **MDZ** Milligram Mg

Medical Dictionary for Regulatory Activities MedDRA

mITT Modified intent-to-treat

Observer's Assessment of Alertness/Sedation

Intravenous

Physical Health Component Score (SF-12v2)

Pharmacokinetic

PT RSAP THOU BE USED TO Patient Management Plan Preferred Term in MedDRA KSA SAS SAS U'' Randomized Safety Population Statistical Analysis Software

Standard deviation

Upsher-Smith Laboratories, Inc.

USL261 Midazolam Nasal Spray, study drug (formally ITI-111)

System Organ Class in MedDRA **TEAE** Treatment-emergent adverse event

**TSQM** Treatment Satisfaction Questionnaire for Medication

WHO World Health Organization

#### INTRODUCTION 1.

Acute repetitive seizures and seizure clusters occur in a subset of epilepsy patients. Seizure clusters have distinguishable characteristics that are easily recognized by patients, caregivers, and physicians and include a consistent onset (auras, prodrome) that may be indicative of convulsive or non-convulsive symptoms. Although patients typically recover between seizures, these seizure can last anywhere from minutes to hours. When a cluster of seizures occurs outside a hospital, the patient must often be transported to an acute care facility so medical personnel can administer intravenous (IV) therapy to stop the seizure(s).<sup>2</sup>

The primary goals of seizure cluster treatment are seizure cessation and prevention of seizure recurrence. Acute benzodiazepine treatment is effective for seizure control and often results in rapid seizure cluster termination; however, most treatment options rely on intervention by emergency medical personnel and, therefore, delay treatment while the patient is transported to a medical facility.<sup>3</sup> The development of an easily administered outpatient treatment of seizure clusters may reduce emergency medical intervention and decrease seizure cluster duration.

This statistical analysis plan covers the detailed procedures for performing statistical analyses and producing tables, listings, and figures of the Phase 3 study Protocol P261-401 (Fifth Issue, Amendment 4, 20 May 2015).

### 2.

### 2.1.

General Study Design and Plan design and Plan an This is a Phase 3 multicenter study, with 2 distinct phases and 4 study center visits as depicted in Figure 1. The first phase is the Test-Dose Phase where subjects will receive 2 doses of openlabel 5.0 mg USL261 10 minutes apart at the study center. The Test-Dose Phase is designed to assess the safety, tolerability and pharmacokinetics of USL261 in a monitored setting and provide the caregivers with training on the study procedures. The Test-Dose Phase will be followed by an outpatient, double-blind, placebo-controlled, parallel-group phase, referred to as the Comparative Phase. In the Comparative Phase, all subjects will be randomized 2:1 to receive 5.0 mg USL261 or placebo. The subject's caregiver will administer the double-blind study drug at the time of a seizure cluster that meets the study criteria, according to the subject's individualized Patient Management Plan (PMP). The double-blind dose of study medication may be followed by an open-label single dose of 5.0 mg USL261 if any of the following occurs:

- The treated seizure cluster has not terminated within 10 minutes after the initial drug administration or
- Another seizure occurs between 10 minutes and 6 hours after administration of the study drug, and the subject does not have <8 breaths per minute, does not require emergency rescue treatment and assisted breathing intubation, and does not have excessive uncharacteristic sedation

Anytime between 24 to 120 hours after study drug administration, subjects and caregivers will return to the study center for a post-dose study visit (Visit 4).

A maximum of approximately 350 subjects, aged 12 years and older, with a documented history of seizure clusters and on a stable AED regimen (no change in type[s] of drug) will be enrolled in the Test-Dose Phase in order to achieve a maximum of 240 subjects completing the Comparative Phase. Before any subject continues to the Comparative Phase, safety data from at least 25 subjects in the Test-Dose Phase will be reviewed by an independent Data and Safety Monitoring Board (DSMB). Enrollment will temporarily halt once approximately 25 subjects complete the Test-Dose Phase, to allow the DSMB to review the safety data. If the safety data from this initial cohort supports continuation of the trial according to the DSMB, enrollment into the Test-Dose Phase will resume and the initial 25 subjects will proceed to the Comparative Phase. All subsequent subjects will progress directly from Test-Dose Phase to the Comparative Phase.

A classic group sequential design, with 3 interim analyses and a maximum sample size of 240 subjects who have completed the Comparative Phase is utilized in order to reach sufficient overall power (approximately 90%) for this study with possible study stopping at interims for efficacy or futility. In this group sequential design, interim analyses will occur after 132, 165, and 204 subjects have completed the Comparative Phase.

Figure 1 shows the overall study scheme with regard to screening. Test-Dose Phase, and Comparative Phase.



### 2.1.1. Screening

After subjects and caregivers have provided informed consent (and assent, where appropriate), subjects will undergo screening procedures at Visit 1 (see Table 1). At Visit 1, training will be provided to the caregivers for self-study, which will be completed at or before Visit 2. The screening period (time between Visit 1 and 2) will be a maximum of 28 days. The screening period may be extended in certain cases; however, the extension of the screening period must be approved by the Sponsor or CRO designee. If a screening period extension is granted for a given subject, that subject will have to undergo repeat screening laboratory and ECG assessments within 28 days before Visit 2.

#### 2.1.2. **Test-Dose Phase**

The Test-Dose Phase, which occurs at Visit 2, will take place at the study center under the supervision of the study investigator within 28 days of Visit 1. The investigator, or other

Subjects who meet eligibility criteria at Visit 2 will receive a test dose of 5.0 mg USL261 administered by a member of the study center personnel followed by a second dose of 5.0 mg USL261 to minutes later administered by the caregiver under the supervision period for at least 4.7 outlined. outlined in Table 1 will be performed. After 132 subjects have completed the Comparative Phase, for all new test dosed subjects, caregivers and study center personnel will monitor the subject during the observation period for at least 1 hour after test dose administration. A subject who experiences signs or symptoms at Visit 2 that are concerning in the investigator's judgment or are exclusionary per exclusion criterion number 22 must be monitored until resolved or longer as deemed appropriate by the investigator.

At least one study center personnel who is trained and qualified to perform airway assessment and management, including endotracheal intubation (or local country /site equivalent) and Advanced Cardiac Life Support (ACLS) (or local country/site equivalent), will be available at the site for the entire observation period following the administration of the first test dose.

#### 2.1.3. **Comparative Phase**

Subjects and caregivers will return to the study center for Visit 3 within 24 hours to 28 days of Visit 2 (unless DSMB review of first 25 subjects is not yet completed). At Visit 3, the investigator, or other qualified study personnel, will review, assess, and (if needed) re-instruct caregivers on the information provided in the self-study training. Before subjects are randomized, caregivers must have demonstrated hands-on competence in administering the study drug, performing timed respiration rate measurements and recording them in the practice Subject Worksheet, as well as airway management techniques.

If the subject continues to meet eligibility criteria at Visit 3, he/she will be randomized to receive either USL261 5.0 mg or placebo. Caregivers will receive a study materials kit, which includes the Subject Workbook, the subject's Patient Management Plan (PMP), and the study drug kit. The PMP will specify the criteria for seizure cluster recognition, the procedure for contacting the central study nurse hotline after study drug administration, the requirements for administering a second dose of study drug (active USL261), and a rescue protocol individualized for the subject.

During the Comparative Phase, caregivers will administer the double-blind study medication at the time of a seizure cluster that meets study criteria (according to the subject's individualized PMP) and call the central study nurse hotline as soon as possible following study drug administration. If the treated seizure has not terminated within 10 minutes after the initial drug administration or another seizure occurs between 10 minutes and 6 hours after administration of the study drug, and the subject does not have < 8 breaths per minute, does not require emergency

rescue treatment with assisted breathing or intubation, and does not have excessive uncharacteristic sedation (as defined by the investigator in the PMP), the second dose of study drug (ie, 5.0 mg dose of USL261) may be administered. If the second dose of study drug is

If the subject encounters persistent seizure cluster activity or seizure recurrence (as defined in the subject's PMP), has < 8 breaths per minute, or is excessively and uncharacteristically sedet. Will outline rescue instruction. EMS (or local equivalent).

Subjects and caregivers will return to the study center 24 to 120 hours after study drug administration for Visit 4. Subjects who are prematurely discontinued from study participation or terminate their participation should return to the study center for Visit 4 (Early Termination). The subject or caregiver will report to the investigator (or his/her designee) as soon as possible any significant medical event (including events that are life-threatening or that result in death, hospitalization or prolonged hospitalization, persistent or significant disability, or incapacity of the subject) that occurs to the subject from the time written informed consent is obtained until completion of the final study visit (Visit 4 [Post-Dose Assessment or ET]) or 7 days after last administration of study drug, whichever is later. The subject or caregiver may also call the central study nurse hotline at any time during the study for help or advice regarding study procedures.

This study will be conducted in accordance with International Conference on Harmonization (ICH) E6. Guidelines for Good Clinical Practice (GCP) and applicable regulatory requirements including the US Code of Federal Regulations dealing with clinical studies (21 Code of Federal Regulations [CFR] including § 50 and \$6 concerning informed consent and Institutional Review Board [IRB] regulations, respectively).

#### 2.2. Randomization and Method of Treatment Assignment

A stratified, blocked randomization schema will be generated by an unblinded statistician and used to assign subjects to treatment. Treatment assignments will be assigned and kept strictly confidential by the Interactive Response Technology (IRT) System. Randomization will be stratified by age  $(< 18 \text{ vs.} \ge 18)$ . Within each stratum, subjects will be randomized in a 2:1 ratio of USL261 5.0 mg nasal spray (active) or matching placebo nasal spray using an appropriate randomly permuted block.

Subjects who meet eligibility requirements at Visit 3 will be randomized to treatment. At the time of randomization, subjects will be assigned unique subject identification numbers. Numbers will be assigned in consecutive increasing order without replacement or reuse of any assigned number. The study will be double-blinded to the treatment group assignment accessible only to authorized persons per sponsor's (or designee's) Standard Operating Procedures (SOPs) until the time of unblinding.

### 2.3. Study Procedures

The schedule of study procedures and evaluations is summarized in Table 1.

**Table 1:** Schedule of the Study Procedures

| Phase | Screening | Test-Dose<br>Phase | | Comparative Ph | ase |
|---|---|---|---|---|---|
| Visit Number | 1 | 2[a] | 3[b] | Treatment[c] | 4 or ET[d] |
| Study Assessments | | | | 1 | aillo |
| Informed consent[e] | X | | | | 1 10 |
| Register subject with IRT | X | | | | 60, |
| Inclusion/Exclusion evaluation | X | X | X | . ( | 103 |
| Caregiver training[f] | X | X | X | 25 | |
| Demographics | X | | | 10 | |
| Medical/surgical history[g] | X | | | et | |
| Concomitant medication review | X | X | X | kn. | X |
| ER and EMS Visit Review[h] | X | | | 70 | X |
| Physical exam[i] | X | X | X c | 100 | X |
| Neurological exam[j] | X | X | X | <i>y</i> - | X |
| B-SIT | | X | X | | X |
| Clinical laboratory testing[k] | X | 4 | 1100 | | X |
| FSH level (females only) | X | 07.0 | 5, | | |
| Pregnancy testing[1] (all females) | X | cOx o | X | | X |
| Drug screen[m] | X | C XOV | Λ | | Λ |
| | | ) 0° | 37 | | |
| Patient Management Plan (PMP)[n] | X | oli X | X | | |
| Central review of seizure cluster | W S | | | | |
| description[o] Treatment administration | | V[] | | X | |
| | K. 1100 | X[p] | | X | |
| Call central study nurse hotline [q] | NO. | 77 | | Λ | |
| Pharmacokinetic blood sampling[r] | SI, | X | | | |
| Observer's Assessment of | | X | | | |
| Alertness/Sedation (OAA/S)[s] | v | 37[4] | | | |
| 12-lead ECG | X<br>X | X[t]<br>X | X | | X |
| Body weight | X | Λ | Λ | | X |
| Height Vital signs[u] | X | X | X | | X |
| Caregiver-recorded respiration rate[v] | Λ | X | Λ | X | Λ |
| Pulse oximetry[u] | | X | | Λ | |
| Report test dose information on IRT | | X | | | |
| Columbia- Suicide Severity Rating | | | | | |
| Scale [w] | X | X | X | | X |
| Outcome Assessments | | X | | | X |
| Randomization using IRT | | 21 | X | | 71 |
| Dispense study materials kit [x] | | | X | | |
| Record seizure activity in Subject | | | Λ | | |
| Workbook | | | | X | |
| Evaluate subject's return to baseline | | | | | |
| functionality [y] | | | | X | |
| Adverse event collection | X | X | X | X | X |
| Collect study drug containers, used and | | | | | |
| unused | | | | | X |

14 April 2017 12

Statistical Analysis Plan for Protocol No.: P261-401

| Review/collect Subject Workbook | | X |
|---------------------------------|------|---|
| Telephone follow-up | X[z] | |

- [a] Visit 2 assessments occurring at the same time should be completed in the following order: ECG, OAA/S, vitals, pulse oximetry, PK blood draw, and second dose; Visit 2 will occur within 28 days of Visit 1. If necessary, assessments may be performed up to 1 minute before or 1 minute after the scheduled time.
- [b] For patients enrolled in the study after the initial DSMB review, Visit 3 will occur a minimum of 24 hours and a maximum of 28 days after Visit 2.
- [c] These assessments will be performed by the caregiver.
- [d] Visit 4 will occur between 24 and 120 hours after double-blind study drug administration. Any subject who has not treated a seizure cluster meeting the study criteria within 6 months of Visit 3 (Randomization) will return to the study center for Visit 4 (Early Termination).
- [e] Informed consent provided by subject (or subject's LAR) and caregiver before any other study-specific procedures; assent may also be required for some subjects
- [f] Caregiver training includes, but is not limited to, providing self-study training to the caregiver and review of that training by the study center personnel. It also includes CPR and airway management training for caregivers.
- [g] Includes seizure history and current/past medication use; complete at Visit.
- [h] At Visit 1, collect number of calls to EMS and ER visits for a seizure cluster or other seizure emergency in the year prior to screening. At Visit 4, collect number of calls to EMS and ER visits for a seizure cluster or other seizure emergency since last visit or follow-up phone call. Number of calls to EMS and ER visits for a seizure cluster or other seizure emergency since last visit or follow-up phone call will also be collected on each monthly telephone follow-up call between Visit 3 and Visit 4 or ET.
- [i] Physical examination includes assessments of the skin, head, eyes, ears, nose, throat, neek, thyroid, lungs, heart, abdomen, lymph nodes, and extremities, and a nasal cavity examination using a nasal speculum.
- [j] A complete neurological examination will be performed at Visits 1 and 4/ET. A partial neurological examination will be performed at Visits 2 and 3.
- [k] Includes hematology, serum chemistry, and urinalysis; phenobarbital levels will be assessed at Visit 1 for subjects taking phenobarbital and in subjects for which the investigator deems it necessary.
- [1] Serum pregnancy test at Visit 1, urine pregnancy tests at Visits 2, 3, and 4/ET.
- [m] Includes barbiturates, benzodiazepines, cocaine, marijuana, methamphetamine, opiates, and phencyclidine (all in urine) and alcohol (blood).
- [n] PMP preparation begins at Visit 1. PMP should be completed before a subject receives the first test dose of USL261 at Visit 2. PMP provided to and reviewed with subject and caregiver at Visit 3.
- [o] Approval of each subject's seizure cluster pattern by central reviewer is required for study inclusion
- [p] At Visit 2, subjects will receive a test dose of 5.0 mg USL261 administered by a member of the study center personnel followed by a second dose of 5.0 mg USL261 10 minutes later administered by the caregiver under the supervision of study center personnel.
- [q] Caregivers to call the central study nurse hotline as soon as possible after administering study drug.
- [r] Blood samples for PK assessment will be collected before and at 5, 10, 20, 30 minutes and 1, 2, and 4 hours after the first test dose. After 132 subjects have completed the Comparative Phase, for all new test dosed subjects, blood samples will be collected before and at 5, 10, 20, 30 minutes and 1 hour after administration of the first 5.0 mg test dose of USL261 at Visit 2.
- [s] At Visit 2, the OAA/S will be administered before and at 5, 10, 20, 30 minutes and 1, 2, and 4 hours after the first test dose by a trained member of the study center personnel. After 132 subjects have completed the Comparative Phase, for all new test dosed subjects, the OAA/S will be administered before and at 5, 10, 20, 30 minutes and 1 hour after the first test dose by a trained member of the study center personnel.
- [t] ECG will be performed twice at Visit 2: once before and once 15 minutes after the first test dose
- [u] Vital signs include blood pressure (BP), heart rate (HR), respiration rate (RR), and temperature. At Visit 2, BP, HR, RR, and pulse oximetry are recorded before and at 5, 10, 15, 20, 30, 45 minutes and 1, 1.5, 2, 3 and 4 hours after the first test dose. After 132 subjects have completed the Comparative Phase, for all new test dosed subjects, BP, HR, RR, and pulse oximetry will be recorded before and at 5, 10, 15, 20, 30, 45 minutes and 1 hour after the first test dose. Temperature will be measured only at the pre-dose time point.
- [v] Caregiver counts the number of breaths taken by the subject during a 30-second interval. At Visit 2, caregivers will measure respiration rate before and at 5, 10, 15, 20, 30, 45 minutes and 1, 1.5, 2, 3 and 4 hours after the first test dose. After 32 subjects have completed the Comparative Phase, for all new test dosed subjects, caregivers will measure respiration rate before and at 5, 10, 15, 20, 30, 45 minutes and 1 hour after the first test dose. On the day of treatment, caregivers will measure respiration rate at approximately 15 and 30 minutes and 1, 2, and 4 hours after study drug administration.
- [w] Baseline/Screening version of the C-SSRS is administered at Visit 1. The Since Last Visit version is administered at Visits 2, 3 and 4/ET.
- [x] The study materials kit will include at a minimum: Individualized PMP, summary of the PMP, Subject Workbook (used for collecting and recording seizure activity information, study drug administration, respiration rate, and other observations made by the caregiver), study drug kit, and dosing instructions.

Statistical Analysis Plan for Protocol No.: P261-401

quality of quality of property of the property

### 3. STUDY OBJECTIVES

### 3.1. Primary Efficacy Objective

The primary efficacy objective is to evaluate the efficacy of USL261 compared with placebo for the outpatient treatment of seizure clusters based on Treatment Success, which is defined as achieving both of the following:

- Termination of seizure(s) within 10 minutes after study drug administration, and
- No recurrence of seizure(s) beginning 10 minutes after study drug administration to 6 hours after study drug administration.

### 3.2. Secondary Efficacy Objectives

The secondary efficacy objectives of this study are to evaluate the efficacy of USL261 compared with placebo for the outpatient treatment of seizure clusters using the following:

- Time to next seizure with a start time >10 minutes after the study drug administration
- Proportion of subjects with recurrence of seizure(s) beginning 10 minutes after study drug administration to 4 hours after study drug administration

## 3.3. Exploratory Efficacy Objectives

The exploratory efficacy objectives of this study are detailed for the comparison of USL261 and placebo for the outpatient treatment of seizure clusters.

- Proportion of subjects with recurrence of seizure(s) beginning 10 minutes after study drug administration to 24 hours after study drug administration.
- Time to return to full baseline functionality (as determined by the caregiver)
- Analyses for subjects receiving 2 doses of study drug
- Subject and caregiver outcome assessments
  - SF-12v2 for both subject and caregiver
  - Treatment Satisfaction Questionnaire for Medication (TSQM)
  - Infranasal Therapy Impact Questionnaire (ITIQ)

### 3.4. Safety Objectives

The safety objectives are to evaluate the safety and tolerability of USL261 for the treatment of seizure clusters using the following assessments:

- Adverse events (AEs)
- Caregiver-recorded respiration rate at 15 minutes, 30 minutes, 1 hour, 2 hours and 4 hours after study drug administration in the Comparative phase
- Requirement for unscheduled emergency room (ER) or emergency medical service (EMS) visit within 24 hours after study drug administration

- Brief Smell Identification Test (B-SIT; United States only)
- Columbia-Suicide Severity Rating Scale (C-SSRS)

### 3.5.

Vital signs (systolic and diastolic blood pressure, heart rate, respiration rate and temperature) as recorded by the study center personnel

Pharmacokinetic Objectives

acokinetic (PK) objective is to evaluate the PK profile of USL261 after administration and the study center personnel

AUC<sub>0-last</sub> – the area under the ineasurable The Pharmacokinetic (PK) objective is to evaluate the PK profile of USL261 after administration of USL261 using the following PK parameters.

- measurable concentration. Estimation by the linear-up/log-down trapezoidal method is preferred.
- $AUC_{0-x}$  the area under the plasma concentration-time curve from time 0 to time x, where x = 1. 2 and 4 hours
- C<sub>max</sub> the maximum plasma concentration
- t<sub>max</sub> the time to maximum plasma concentration
- $t_{lag}$  the time before the first measurable plasma concentration

#### **ANALYSIS POPULATIONS** 4.

#### **Screened Population** 4.1.

The Screened Population includes all subjects who signed an Informed Consent Form (ICF) or assent form.

#### 4.2. Safety Population

The Safety Population includes all subjects who received at least 1 dose of study drug even if they were not randomized. Therefore, this population includes all treated subjects, including those who terminate following the test dose (Visit 2), but before randomization (Visit 3), as well as subjects who are randomized.

### **Randomized Population**

The Randomized Population includes all subjects who are randomized to receive double-blind treatment. The Randomized Population is also the Intent-to-treat (ITT) Population.

#### 4.4. **Randomized Safety Population**

The Randomized Safety Population (RSAF) is the group of subjects who are randomized and USL261 5 mg: USL261 group who received only the first dose of double-blind study drug
 USL261 5 mg: USL261 group who received only the first dose of double-blind study drug and the second dozen. receive at least one dose of double-blind study drug. If a subject received the wrong treatment in the double-blind period or until discontinuation, the safety data for that subject will be summarized under the actual treatment group received. The demographic, baseline characteristics and safety data will be summarized under the following treatment groups:

- Placebo: Placebo group who received only the first dose of double-blind study drug
- Placebo + USL261 5 mg: Placebo group who received the first dose of double-blind study drug and the second dose of open-label USL261

#### **Modified Intent-to-Treat Population (mITT)** 4.5.

The mITT Population includes all subjects in the Randomized Population who received at least 1 dose of study drug during the Comparative Phase, who had post-treatment efficacy assessment (ie, with any seizure diary data). This mITT definition was chosen because Randomized subjects may be discontinued from the study prior to treatment in the Comparative Phase. Following the intent-to-treat principle, all efficacy analyses will be conducted using the mITT Population, analyzed according to the randomized treatment assignment. The potential biases arising from excluding randomized subjects who did not receive study medication are negligible since exclusion is not influenced by knowledge of whether being assigned to USL261 or placebo.

#### 4.6. Per Protocol Population

The Per Protocol Population includes all subjects in the mITT Population who did not discontinue study participation or have any excludable protocol deviations (see Section 7.2).

All protocol deviations will be reviewed in a blinded manor prior to DB lock and it will be determined prior to DB lock if a patient should be excluded from the Per Protocol population. The Per Protocol population will be used for supportive analysis to assess robustness of the primary analysis.

#### Pharmacokinetic Population 4.7.

The PK Population includes all subjects who received a test dose of USL261 in the Test-Dose Phase, have at least one quantifiable post-dose concentration and have no excludable protocol deviations (see Section 7.2). All protocol deviations will be reviewed in a blinded manor prior to DB lock and it will be determined prior to DB lock if a patient should be excluded from the PK population.

#### **5.** GENERAL STATISTICAL CONSIDERATIONS

#### 5.1. **Level of Significance**

analysis section.

To control Type I error for the primary and secondary efficacy endpoints, a statistical gate-keeping procedure will be applied to control for multiplicity. The primary and secondary efficacy endpoints will be tested individually using the following hierarchical procedure:

First step: The proportion of subjects that are classified as T Comparative Phase (two sided not in the control of the primary and secondary efficacy endpoints will be tested individually using the following hierarchical procedure:

To proceed to the next step in the hierarchy, the previous step must be statistically significant (ie, two sided p-value is significant favoring USL261).

Second step: Time to next seizure following first dose of study drug (p-value from the log-rank test) will be determined.

Third step: The proportion of subjects with recurrence of seizure(s) beginning at 10 minutes after to 4 hours following the first dose of study drug.

All null hypotheses will be defined as no treatment difference

#### **Handling of Missing Data** 5.2.

Any specific imputation procedures for missing or incomplete data will be discussed in the section describing analytic methods for the efficacy/safety variable in question. Unless otherwise stated, observed data will be presented in tables and listings without imputation of missing values.

AEs with non-complete start dates and complete stop dates after the first double-blind study drug administration will be considered TEAEs during the Test Dose Phase if:

- Time is missing and the date is equal to or after the date of test-dose administration and is equal to or before the date of the first double-blind study drug administration:
- Day and month are missing and the year is equal to or after the year of test-dose administration but is equal to or before the year of the first double-blind study drug administration;
- Day is missing and the year is equal to or after the year of test-dose administration but is equal to or before the year of the first double-blind study drug administration;
- Day is missing, the year is equal to the year of test-dose administration, and the month is equal to or after the month of test-dose administration but is equal to or before the month of the first double-blind study drug administration;
- Year is missing;
- Complete date is missing.

Upsher-Smith Laboratories, Inc. Statistical Analysis Plan for Protocol No.: P261-401

AEs with partial start dates and complete stop dates after administration of the first double-blind study drug will be considered TEAEs during the Comparative Phase if:

- Time is missing and the date is after the date of the first double-blind study drug

- Day is missing and the year is after the year of the first double-blind administration;

  Day is missing, the year is equal to the year of the first double-blind study drug administration, and the month is after the administration.

Missing AE relationships will be presented as 'related' in tables but missing in listings. Missing AE intensity will be considered as 'severe' in tables but will be reported as missing in listings.

Medications with non-complete dates will be considered concomitant if partial dates show that medications were taken between the day of first dose of study drug at Visit 2 and the end of study. Medications will be considered prior if partial dates show that medications were taken within 30 days prior to the first dose of study drug at Visit 2 Medications can be categorized as both prior and concomitant.

### 5.3.

**5.3. Interim Analyses**Three interim analyses will be conducted to evaluate the treatment success rate for possible early stopping for success or futility. The interim analyses will occur after 132, 165, and 204 subjects complete the Comparative Phase (ie, subjects have received at least 1 dose of study drug during the Comparative Phase). All interim analyses will be performed on the mITT population, ie, subjects that are randomized and experience a cluster seizure event during the comparative phase. Subjects lost to follow-up or with missing primary outcome information will be considered treatment failures.

Treatment success is defined in Section 7.6.1.1.

#### 5.3.1. **Early Success**

Early success will be declared as shown in Table 2. A group sequential design is used to allow for multiple interim analyses for efficacy, yet control the type I error rate at 2.5%. The Lan-DeMets spending function approximation of the Pocock boundary, is used for the efficacy boundary. The critical values for this efficacy boundary were obtained using R package gsDesign (version 2.8-8).

At each interim analysis, a one-sided Fisher's Exact test on the two proportions will be performed and compared to the Lan-DeMets Pocock approximation boundary critical values. For the three planned interim analyses and the final analysis, the critical values are presented in Table 2.

Required p-values for declaring success according to Lan-DeMets Pocock Table 2: **Approximation Spending Function** 

| Interim | P-value |
|----------|---------|
| Analysis | |
| 132 | 0.0166 |
| 165 | 0.0094 |
| 204 | 0.0089 |
| 240 | 0.0085 |

#### 5.3.2. **Early Futility**

, sions or variations thereof. Also at each of the pre-specified interim analyses (N=132, 165, 204), the predictive probability of success at the maximum sample size is computed (futility is not applicable to the final analysis at 240 subjects). The predictive probability calculation begins by assuming non-informative uniform prior distributions. Beta(1,1), on the treatment success rates for the placebo/control arm  $(p_C)$  and the probability of treatment success in the treatment arm  $(p_T)$ , and computing the posterior distribution with the currently available data. The predictive distribution of the final data assuming the maximal sample size of N=240 is then computed. The number of future treatment successes for each arm has a Beta-Binomial distribution which is then added to the fixed number of current treatment successes in each arm. We may then compute the predictive probability that a trial success is reached at N=240 subjects. If this predictive probability is less than 10%, the trial is stopped for futility. Note that the success boundaries are computed assuming no futility stopping, and thus controls type I error regardless of the method used for futility stopping.

### Early Termination not related to Success or Futility 5.3.3.

If the trial has not crossed a boundary for early success or early futility and yet is stopped early before reaching the pre-specified maximum sample size of 240 subjects, the final analysis will be conducted with the enrolled patients in the mITT population. The p-value required for study success will remain as the p-value required at the final analysis according to the pre-specified Lan-DeMets Pocock boundary as if the trial had performed all planned interim analyses and continued to the maximum sample size. Therefore the p-value required for success will be p=0.0085 as described in Table 2 (Section 5.3.1).

#### Logistical details for interim analyses 5.3.4.

The interim analyses will be conducted by an unblinded statistician and reviewed by an unblinded interim analysis monitoring committee (IAMC), both independent of the sponsor. The IAMC will consist of two individuals with adaptive design expertise to ensure the pre-specified adaptations are performed as planned, and to react to any unanticipated issues. The IAMC will be independent of the DSMB. IAMC membership, responsibilities, timelines, and communication channels will be clearly specified in a charter. In particular, the IAMC communication channels with the sponsor will be limited to maintain the blind of the sponsor study team in order to minimize the chance of operational bias. To this end, the IAMC will inform senior management first of the decision to continue the trial or stop according to the

statistical analysis plan. The senior management will in turn inform the team to continue or not to continue the study only with no further information on the interim analysis.

#### 5.4. **Examination of Subgroups**

JORS OF Variations thereof. Further analysis of the primary and secondary endpoints may be examined for consistency across the subgroups listed below. Any subgroup analyses will be exploratory in nature.

- Age (< 18 years,  $\ge$  18 < 65 years,  $\ge$  65 years)
- Sex (male/female)
- Race (white/non-white)
- Enzyme-inducing AEDs used within 14 days before the study drug administration (see Appendix 2) vs. others
- Weight categories (</\ge Median weight of the safety population)
- Region (North America and similar [this includes USA, Canada, Australia and New Zealand], Eastern Europe [Hungary, Poland, Ukraine], and Western Europe [Spain, Germany, Italy, and Israel])
- BMI standardized categories (underweight/normal [<25], overweight [\ge 25-<30], and obese 1-3 categories combined [≥30])

#### Data Collected from Unscheduled Visits 5.5.

The data collected from the unscheduled visits are excluded from the by visit summary analysis.

However, when defining baseline for each assessment, the data collected from the unscheduled visits are still included.

#### **DESIGN OPERATING CHARACTERISTICS 6.**

#### Simulation Scenarios 6.1.

The estimated placebo treatment success rate is 0.40. The study is powered under the hypothesis that the USL261 treatment will lead to a clinically meaningful odds ratio of 2.9. With these assumptions, the sample size of 240 subjects who have completed the Comparative Phase (160 USL261/80 placebo) is sufficient to obtain approximately 90% power.

We examined a range of odds ratios/treatment success rates for placebo treatment success rates of 40% and performed 10,000 simulations to determine the power and average sample size (type I error is controlled analytically through the group sequential design). Simulations were performed using R version 3.1.0. For a given set of data we computed the success and futility criteria analytically. To simulate an individual trial, placebo and treatment data were simulated from the appropriate Binomial distributions (using the required sample sizes and placebo and treatment rates) and compared to the success and futility bounds. Trials that continued at an interim had additional data simulated, and so on until the trial reached completion. After

simulating 10,000 trials, the overall power, expected sample size, and other operating characteristics were computed by taking the observed mean values throughout the simulations.

### **6.2.** Operating Characteristics

Assuming treatment success rates of 0.40 for the placebo arm, and Odds Ratio of 2.9, the power of this design is approximately 90% while maintaining at most 2.5% type I error. The expected (average) sample size will be approximately 150.

### 7. STATISTICAL ANALYSIS

Categorical variables will be summarized using counts and percentages. Continuous variables, including the change from baseline, will be summarized using descriptive statistics [n, mean, standard deviation (SD), minimum, median, maximum]. For modeling results, least squares means and standard errors will be presented.

Unless otherwise stated, all summaries will be presented by treatment group (USL261 or Placebo).

The Test Dose Phase is defined as the period of time from the date of first dose of study drug administration at Visit 2 up to, but not including, the date of randomization. The Comparative Phase is defined as the period of time from the date of randomization to the date of the last assessment in the study.

Table 3: Study Phases Start and End

| <b>Epoch Name</b> | Start Date | End Date |
|---|---|---|
| Before Screening (BS) | Birth date | Date of Screening – 1 day |
| Screening (SC) | Date of screening | Date of Visit 2 – 1 day |
| Test-Dose (TD) | Visit 2 | Visit 3 (not including the date |
| | 4 | of randomization) |
| Double-blind (DB) | Visit 3 day | Visit 4 |
| Post Treatment but in Study | Study drug discontinuation | Visit 4 |
| (PD) | visit +1 day | |
| Post Study Follow-up (PS) | If enter Double-blind: Visit 4 | Open ended |
| USE | +1 day | |
| not blady romes up (18) | If failed during TD: Visit 3 + | |
| anor | 1 day | |

Baseline values are the last available values before Test-Dose administration. For rescreened subject who underwent two Test-Dose administration, the last available values before the later Test-Dose administration will be defined as Baseline values.

Data listings will include all subjects with at least one applicable value. Listings will be sorted by treatment group, site, subject number, and date (if applicable).

14 April 2017 22

All datasets and output will be produced using SAS® Version 9.1.3 or higher (SAS Institute, Inc., Cary, North Carolina, USA).

#### 7.1. **Subject Disposition**

All individual subject disposition data will be listed by clinic/investigator site for screen failures separately, and for subjects in the Safety Population separately.

The primary reason for screen failure will be listed for all screen failed subjects.

Subject disposition will be presented by the primary reason for early withdrawal for the Safety Population during the Test Dose Phase. The number and percent of subjects who completed the study and the number and percent of subjects who discontinued the study along with the distribution of the reasons for study discontinuation will be presented in total and by phases for all study populations wherever applicable (see Figure 2).



Completer

### **Protocol Deviations**

All instances of protocol non-compliance will be tracked during the study and CSR Reportable protocol deviations will be finalized by a blinded Sponsor review prior to database lock. CSR Reportable deviations are deviations that materially affect the evaluation of efficacy or safety. CSR Reportable deviations will be reviewed in a blinded manner to determine if the data should

Completer

be excluded from an analysis population. A subject with a CSR Reportable protocol deviation will not necessarily be excluded from the analysis populations. The excludable protocol deviations will be classified by the sponsor for each population. Protocol deviation categories

Demographics and Baseline Characteristics

Demographics and baseline Characteristics

Demographics and baseline characteristics will be presented for the Safety Ropulation and repeated for the Randomized Safety and mITT Populations. Subject demographics include age gender, weight, height, BMI, race, clinical site region, and ethnicity. Weight recorded will be converted to kilograms, and height recorded in inches will be converted to kilograms.

In addition subject age (years) will be categorized as follows:

- < 18 years
- $\geq 18 < 65 \text{ years}$
- > 65 years

Subject baseline characteristics will include: IQ (if available), epilepsy type, developmentally delayed status, EEG history, CT scan and/or MRI history, previous and current seizure types, seizure etiology including primary cause of epilepsy, and seizure cluster episode history. For seizure cluster episodes, if duration are collected in free-text which covers a period of time, average of the upper bound and the lower bound will be used for the analysis.

Subject demographics will additionally be presented for the mITT Population by the Treatment Success status of their first double-blind dose of study drug (see Section 7.6.1 for the definition of treatment success). These data presentations will include columns for "Treatment Success of first dose and "Not Treatment Success of first dose" for each treatment group.

Comparability of treatment groups will be evaluated using descriptive statistics.

### **Medical and Surgical History**

This docur?.4. Medical and surgical history will be coded using the MedDRA coding dictionary version 14.1. Coded medical history terms will be summarized by MedDRA system organ class (SOC) and preferred term (PT) for the Safety, Randomized Safety and mITT Populations. SOC will be sorted alphabetically and then preferred term will be sorted in order of frequency of the total

column within each SOC. At each level of summarization, a subject will be counted only once for each medical and surgical history he/she has within that level. Subject listings of coded medical history terms will be provided.

For subjects who were rescreened after study drug exposure and have two subject identifiers, all medical and surgical history data will be combined into one subject identifier.

### 7.5. Prior and Concomitant Medications

Prior medications are defined as medications taken within 30 days prior to the first dose of study drug at Visit 2. Concomitant medication is defined as any medication taken between the day of first dose of study drug at Visit 2 and the end of study.

The World Health Organization Drug Dictionary (WHO Drug) of version December 2011 will be used to classify prior and concomitant by therapeutic class and preferred name based on ATC code level 4. Medication start and end dates will be compared with the start date of study drug and classified as per Table 4.

In case of partial or missing dates, comparisons will be made based on the level of detail available. For example, if start date of study drug administration is 04Jan2013, and a medication has a start date of Jan2013 but missing date the medication will be classified as concomitant.

| End<br>date<br>Start<br>date | Before start of<br>study drug<br>administration at<br>Visit 2 | On or after start of study drug administration at Visit 2 | Missing |
|---|---|---|---|
| Before start of study<br>drug administration at<br>Visit 2 | Prior | Prior/Concomitant | Prior/Concomitant |
| On or after start of study drug administration at Visit 2 | - | Concomitant | Concomitant |
| Missing | Prior | Prior/Concomitant | Prior/Concomitant |

Prior medications will be summarized for the Safety, Randomized, and Randomized Safety Populations. Concomitant medications will be presented for the Safety Population during the Test Dose Phase and for the Randomized and Randomized Safety Populations during the Comparative Phase. Levels of summarization will include global, WHO Anatomic Therapeutic Chemical (ATC) Classification System level 3 drug class, ATC level 4 drug class, and WHO preferred term.

At each level of summarization, a subject will be counted only once for each concomitant medication he/she has within that level. The percentage of subjects having had at least one medication at each level will be calculated

14 April 2017 25

Upsher-Smith Laboratories, Inc. Statistical Analysis Plan for Protocol No.: P261-401

Prior/Concomitant medications excluding AEDs, prior/concomitant AEDs, prior/concomitant AEDs used for epilepsy, and prior/concomitant AEDs used for indications other than epilepsy will be summarized separately and similar to concomitant medications. AEDs will be further classified as enzyme-inducing and non-inducing AEDs.

Listings will be provided for prior/concomitant medications and prior/concomitant AEDs for all subjects. AEDs collected from AED page on CRF will be presumed to have 'Epilepsy' as indication. AEDs collected from concomitant medication page will be listed by indication captured on CRF.

For subjects who were rescreened after study drug exposure and have two subject identifiers, all medication data will be combined into one subject identifier.

#### 7.6. **Analyses of Efficacy Endpoints**

Information recorded by the caregiver in the Subject Workbook will be used for analysis of the primary, secondary, and exploratory efficacy endpoints. Any seizures occurring within 24 hours after administration of study drug will be recorded. Subjects without any recurrent seizures recorded with a start time >10 minutes after administration of study drug will be considered seizure-free in all analyses.

The following covariates will be used in the analyses of efficacy endpoints, where specified:

- Age (< 18 years, 18 <65 years, ≥65 years)

- Sex (male/female)
  Weight (kg)
  BMI standardized categories (underweight/normal [<25], overweight [≥25-<30], and</li> obese 1-3 categories combined  $[\geq 30]$ )
- Geographic region of clinical site (North America and similar [this includes USA, Canada, Australia and New Zealand], Eastern Europe [Hungary, Poland, Ukraine], and Western Europe [Spain, Germany, Italy, and Israel])
- Enzyme-inducing AEDs used within 14 days before the study drug administration (see Appendix 2) vs others

Additional covariates may also be explored.

#### **Primary Efficacy Endpoint** 7.6.1.

All statistical analyses of the primary efficacy endpoint will be conducted for the mITT Population and analyzed as described in Section 5.3. The primary efficacy endpoint analyses will also be conducted on the Per Protocol Population as supportive analyses. The following null (H<sub>0</sub>) and alternative (H<sub>a</sub>) hypotheses will be evaluated:

- H<sub>o</sub>: The proportion of subjects who meet the criteria for Treatment Success is not different between the USL261 and the placebo groups in the Comparative Phase;
- H<sub>a</sub>: The proportion of subjects who meet the criteria for Treatment Success is different between the USL261 and the placebo groups in the Comparative Phase.

Upsher-Smith Laboratories, Inc. Statistical Analysis Plan for Protocol No.: P261-401

Treatment Success is a composite measure of efficacy that will be assessed based upon the first seizure cluster treated with study drug during the Comparative Phase. Treatment Success is defined as achieving the following:

- Termination of seizure(s) within 10 minutes after the double-blind study drug
- No recurrence of seizure(s) beginning 10 minutes after study drug administration to 600 hours after the double-blind study drug administration

  Derivation of Treatment Succession.

Treatment Success Endpoint

Treatment Success will be determined based on data reported in the CRFs and derived programmatically. An imputation will be conducted first for the seizure start time.

If the end time of a seizure is missing imputition if the two selections in the selection is the two selections.

time if the two aforementioned seizures occrurred within the same date; otherwise, the missing end time will be imputed as 23:59.

If the start time of a seizure is missing, impute the start time to the previous seizure's end time if the two aforementioned seizures occurred within the same date; otherwise, the missing start time will be imputed as 00:00.

There are three components to be assessed in the programmatic derivation:

- 1. Termination of seizure(s) within 10 minutes: The initial seizure stopped within (<) 10 minutes from the time of dosing and any subsequent seizures also stopped within 10 minutes of dosing. Data used in this derivation includes the time of first dose as recorded on the "Study Drug Administration (First Dose)" CRF, and seizure data recorded on the "Report All Seizures for 24 Hours" and the "Seizure Diary" CRFs.
- 2. No recurrence of seizure(s) beginning 10 minutes after study drug administration to 6 hours after study drug administration. The times of reported seizures will be used to assess if there are any seizures with start time from >10 minutes up to  $(\leq)$  6 hours after the first dose of study drug. Data used in this derivation includes seizure data recorded on the "Report All Seizures for 24 Hours" CRF.
- 3. No second dose given within 6 hours of the first dose of study drug administration as receiving the second dose within  $(\leq)$  6 hours confounds the efficacy evaluation of the first dose. Data used in this derivation include the time of second dose as recorded on the "Study Drug Administration (Second Dose)" CRF.

Subjects who meet all three of these components will be defined as a "Treatment Success." If a subject does not meet all three of these components, (which may or may not be due to missing data), they will be defined as "Not a Treatment Success."

Possible scenarios for seizure data start and stop times within the 6 hour period following the first dose of study drug are displayed below in Figure 3, along with the treatment success endpoint derivation (assuming no second dose was given):

Figure 3: Possible Scenarios for Seizure Data Start and Stop Times Within the 6 Hour Period Following the First Dose of Study Drug Are Displayed Below, Along with the Treatment Success Endpoint Derivation (Assuming No Second Dose was given)



## 7.6.1.2. Analysis of the Primary Endpoint

Treatment Success will be analyzed by Fisher's Exact test. The 95% confidence intervals (CIs), using normal approximation around the proportions, will be presented. In addition, each component (seizure termination and recurrence) of treatment success will be summarized by treatment group. Chi-squared test will be performed as a sensitivity analysis. Results from both tests (Fisher and Chi-squared) will be presented together. In addition, the Cochran-Mantel-Haenszel (CMH) test, stratified by age (< 18 years,  $\ge 18$  - <65 years,  $\ge 65$  years) will be used to analyze Treatment Success.

Subjects who do not have sufficient available data to confirm whether they can be classified either as "Treatment Success" or as "Not a Treatment Success" as described in Section 7.6.1.1 are considered to have missing data. For the primary analysis of Treatment Success, subjects with missing data impacting the Treatment Success endpoint described above will be considered as "Not a Treatment Success."

Similarly, for each component of the Treatment Success endpoint (seizure termination and recurrence), when available data do not allow to determine the classification, subjects with

14 April 2017 28

missing data will be considered as having an unfavorable outcome for the corresponding component. Sensitivity analysis will be conducted for the Treatment Success endpoint in order to assess robustness of study conclusions to missing data using a tipping point approach.<sup>4</sup> This mong subjects with missing data in the USL261 and Placebo treatment groups. Clinical interpretation of the plausibility of different combination of outcomes will be provided in the Clinical Study Report. The tipping point analysis will be conducted as follows. Let  $n_{1m}$  and  $n_{2m}$  be the number of subjects with missing data in the USL261 and Placebo treatment groups respectively.

Step 1: Let  $k_1$ =0.

Step 2: Let  $k_2$ =0.

Step 3: Repeat the analysis of the primary endpoint as described above by considering 1 subjects from the USL261 treatment group as "Not a Taxable Considering 1 as "Treatment States".

as "Treatment Success," while considering k2 subjects from the Placebo treatment group as "Not a Treatment Success" and (n<sub>2m</sub> - k<sub>2</sub>) subjects as "Treatment Success."

Step 4: Let  $k_2 = k_2 + 1$ . Repeat Steps 3 - 4 while  $k_2 \le n_{2m}$ .

Step 5: Let  $k_1 = k_1 + 1$ . Repeat Steps 2 - 5 while  $k_1 \le n_{1m}$ .

The results of the analysis for each possible combination of outcomes for subjects with missing data (k<sub>1</sub> and k<sub>2</sub>) will be presented in a table. Additionally, a graph will be produced presenting the number of subjects with missing data considered as "Not a Treatment Success" on the X and Y axes for the USL261 and Placebo treatment groups respectively, and dots marking the combinations of X- and Y-axis values for which the null hypothesis was not rejected in favor of the USL261 treatment.

An additional exploratory logistic regression on Treatment Success will include the covariates specified in Section 7.6. A backward selection of covariates will be used to obtain the final model. All covariates with a p>0.10 will be dropped from the model. The covariates remaining in the final model that are identified as having significant association with the outcome (p<0.05) may be explored in a subgroup analysis. The odds ratio between USL261 and Placebo and its associated 95% confidence intervals will be reported. This analysis will be conducted considering all subjects with missing data as "Not a Treatment Success", similar to the primary analysis.

#### **Secondary Efficacy Endpoints** 7.6.2.

All secondary efficacy analyses will be based on the mITT population. Multiplicity adjustments are described in Section 5.1).

# This documation. Proportion of Subjects with Recurrence of Seizure(s) Beginning 10 Minutes after Administration of Double-Blind Study Drug to 4 Hours after Double-Blind **Study Drug Administration**

The proportion of subjects with recurrence of seizure(s) recorded in the diary with start time >10 minutes and \( \leq 4 \) hours after the administration of double-blind study drug will be analyzed using Fisher's Exact test. The 95% CIs will be presented for the proportion. In addition, Chi-squared

test will be performed as a sensitivity analysis. Subjects who have been administered the second dose of study drug (ie, 5.0 mg dose of USL261) within 4 hours of double-blind study drug administration will be derived as if they had a recurrence of seizure. Subjects who do not have a seizure recorded, or whose first seizure occurs >4 hours after study drug administration, will be counted as not having a seizure.

# 7.6.2.2.

Time to Next Seizure with a Start Time >10 Minutes after Double-Blind Study
Drug Administration
eier estimates will be used to summarize the time-to-next seizure after de la description administration. Subjects who do not be Kaplan-Meier estimates will be used to summarize the time-to-next seizure after double-blind study drug administration. Subjects who do not have another seizure before the end of the 24hour observation period, and have not been administered the second dose of study drug (ie, 5.0) mg dose of USL261) will be censored at the end of the observation period. Subjects administered the second dose of study drug (ie, 5.0 mg dose of USL261) who did not have a seizure before the administration of the second dose will be censored at the time of the second dose (5.0 mg USL261) administration. The time-to-next seizure percentiles (defined based on the data) with associated 95% CIs will be displayed. The probabilities of experiencing the next seizure after double-blind study drug administration at each hour with associated standard error and 95% confidence intervals will be presented. The log-rank test will be used to compare the time to next seizure after double-blind study drug administration between treatment groups. In addition, the hazard ratio for treatment (USL261: placebo) and its 95% CI will be calculated from a Cox proportional hazards model. Kaplan-Meier curves by treatment group will also be presented.

Additional analysis will be conducted based on a different censoring method that subjects administered the second dose of study drug (ie, 5.0 mg dose of USL261) who did not have a seizure before the administration of the second dose will be considered as events (failure).

The Cox proportional hazards regression model will be used to evaluate the difference between treatment groups adjusting for the covariates specified in Section 7.6. Interactions between treatment and each covariate will be evaluated at the 0.10 significance level; if not significant, they will be removed from the final model.

#### **Exploratory Efficacy Analyses** 7.6.3.

Exploratory efficacy analyses will be conducted using the mITT population. All tests performed will test a two-sided hypothesis of no difference between groups at a significance level of 0.05 for all exploratory outcome measures.

### Proportion of Subjects with Recurrence of Seizure(s) Beginning 10 Minutes after 7.6.3.1. Study Drug Administration to 24 Hours after Study Drug Administration

The proportion of subjects with recurrence of seizure(s) with a start time >10 minutes and ≤24 hours after study drug administration will be analyzed using Fisher's Exact Test. The 95% CIs will be presented for the proportion. In addition, Chi-squared test will be performed as a sensitivity analysis. Subjects who do not have a seizure recorded with a start time >10 minutes and ≤24 hours after the administration of double-blind study drug will be counted as not having a seizure. Subjects who have been administered the second dose of study drug (ie, 5.0 mg dose of USL261) within 24 hours will be assumed to have had a seizure.

### Return to Full Baseline Functionality within 24 Hours after Study Drug Administration (as determined by the caregiver)

a time of return to full baseline functionality recorded within 24 hours of study drug administration or who have been administered the second dose of study drug (ie, 5.0 mg dose of USL261) prior to returning to full functionality will be counted as not having returned to full baseline functionality.

Kaplan-Meier estimates The proportion of subjects who have documented return to full baseline functionality will be

Kaplan-Meier estimates will be used to summarize the time to return to full baseline functionality. Subjects who do not have a time of return to full baseline functionality recorded within 24 hours of study drug administration and have not been administered the second dose of study drug (ie, 5.0 mg dose of USL261) will be censored at the end of the observation period. Subjects who were administered the second dose of study drug (ie, 5.0 mg dose of USL261) prior to returning to full functionality will be censored at the time that the second dose (USL261) was administered. The probabilities of return to full baseline functionality after double-blind study drug administration at each hour with associated standard error and 95% confidence intervals will be presented. The log-rank test will be used to compare the time to return to full baseline functionality between treatment groups. In addition, the hazard ratio for treatment (USL261: placebo) and its 95% CI will be calculated from a Cox proportional hazards model. Kaplan-Meier curves by treatment group will also be presented.

The Cox proportional hazards regression model will be used to evaluate the difference between treatment groups adjusting for the covariates specified in Section 7.6. Interactions between treatment and each covariate will be evaluated at the 0.10 significance level; if not significant, they will be removed from the final model.

#### Analyses for Subjects Receiving 2 Doses of Study Drug 7.6.3.3.

Data from subjects randomized to USL261 and placebo who received the first dose of doubleblind study drug and the second dose of open-label study drug (ie, 5.0 mg dose of USL261) will be used for the analyses of subjects receiving 2 doses of study drug.

### 7.6.3.3.1. Treatment Success of the Second Dose of Study Drug (5.0 mg of USL261)

Treatment Success of the second dose for subjects receiving the second dose of study drug (ie, 5.0 mg of USL261) will be presented for each treatment group. For the active group, this represents two doses of 5.0 mg of USL261. The placebo group has received one dose of 5.0 mg of USL261 (preceded by a dose of placebo). Since the administration of the second dose is not a For this analysis, Treatment Success of the second dose is defined as achieving the following:

• Termination of seizure(s) within 10 minutes after 41.

mg of USL 261 randomized treatment, the analysis includes only subjects whose seizure was not stopped by the

Termination of seizure(s) within 10 minutes after the second dose of study drug (5.0

• No recurrence of seizure(s) beginning 10 minutes after administration of the second dose of study drug (ie, 5.0 mg of USL261) to 6 hours after the second dose of study drug (5.0 mg of USL261)

Subjects whose Subject Workbook indicates seizure termination within 10 minutes of the second dose and who have no seizures recorded with start time > 10 minutes and  $\leq 6$  hours after the second dose of study drug will be considered a Treatment Success of the second dose. Subjects who do not meet either of these criteria will not be considered a Treatment Success of the second dose. Similar derivation rules as used for the primary endpoint will be used for defining Treatment Success of the second dose, with the exception of not including the rule pertaining to the second dose.

Number and percentage will be presented for Treatment Success of the second dose and each component (seizure termination and recurrence) for subjects who received two doses of study drug. The 95% CIs for the proportions will also be presented.

### 7.6.3.3.2. Additional Second Dose Data Presentations / Analyses

A summary of subjects receiving the second dose of study drug by randomized treatment arm will be presented. In addition to the total number of subjects receiving the second dose, counts of subjects receiving the second dose in specific time categories post first dose (0 to <10 minutes, >=10 to  $\leq$ 20 minutes, >20 minutes to  $\leq$ 1 hr, >1 hr to 6 hrs, and >6 hrs) will also be presented.

Kaplan-Meier estimates will be used to summarize the time-to-second dose. Subjects who do not receive the second dose of study drug (ie, 5.0 mg dose of USL261) within 6 hours of the initial study drug administration will be censored at the end of this 6 hour period. The time-to-second dose percentiles (defined based on the data) with associated 95% CIs will be displayed. Kaplan-Meier curves by treatment group will also be presented.

As an additional exploratory analysis, a logistic regression with response treatment success of the second dose will be examined including time from first dose to second dose as a continuous covariate with treatment as an effect.

Kaplan-Meier estimates will also be used to summarize the time-to-next seizure following the second dose. Subjects who do not have another seizure before the end of the 24-hour observation period following the second dose of study drug (ie, 5.0 mg dose of USL261) will be censored at the end of this observation period. The time-to-next seizure following the second dose percentiles (defined based on the data) with associated 95% CIs will be displayed. The probabilities of experiencing the next seizure following the second dose at each hour with associated standard error and 95% confidence intervals will be presented. Kaplan-Meier curves by treatment group will also be presented.

### 7.6.3.4. Treatment Success of all Dose of Study Drug

Treatment Success of all doses will be assessed based upon the Treatment Success of the first dose and Treatment Success of the second dose taken within 6 hours after first dose during the Comparative Phase. If the second dose taken later than 6 hours after first dose, then treatment success of all doses will only be based on the result of treatment success for the first dose.

The same analysis as described in Section 7.6.3.3.1 (Treatment Success of the Second Dose of Study Drug) will be performed for treatment success of all doses.

14 April 2017 32

### 7.6.3.5. Subject and Caregiver Outcome Assessments

### 7.6.3.5.1. SF-12v2

The SF-12v2 is a 12-item questionnaire which will be administered to both the subject and caregiver at Visits 2 and 4. All analyses will be presented separately for the subject and caregiver. Eight domains make up the SF-12v2: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. In addition, the physical functioning, role-physical, bodily pain, and general health domains will be combined to obtain the Physical Health Component Score (PCS); the vitality, social functioning, role-emotional, and mental health domains will be combined to obtain the Mental Health Component Score (MCS). The scores for each domain, the PCS and the MCS range from 0 to 100 where zero indicates the lowest level of health by the scales and 100 indicates the highest level of health.

Summary scores for PCS and MCS for each patient will be computed using published algorithms. Each summary measure is scored and standardized using a t-score transformation, such that a higher score represents better health status, with a mean score of 50 and a standard deviation of 10 in the general population. Missing data on the SR-12v2 will be handled as follows: domain scores will not be calculated for domains in which data are missing. Subsequently, component scores in which domain scores are missing will not be calculated.

Summarization and analysis of SF-12v2 data will be performed for the mITT and the Randomized Safety population. The domain and component scores will be presented for Visit 2 (baseline) and Visit 4/ET, including change from baseline. For each domain and component score a paired t-test will be used to assess the within-group mean change from baseline. An analysis of covariance (ANCOVA), with treatment and baseline as covariates, will be used for between-group comparison of change from baseline for the domain and component scores.

### 7.6.3.5.2. Treatment Satisfaction Questionnaire for Medication (TSQM)

The TSQM is a 14- item questionnaire that will be administered to the subject. The four TSQM scale scores calculated from the questionnaire are: effectiveness, side-effects, convenience, and global satisfaction. The TSQM scale scores are computed by adding the items loading on each factor. The lowest possible score is subtracted from the composite score and divided by the greatest possible score minus the lowest possible score. This will provide a transformed score between 0 and 1 that is then multiplied by 100. If more than one item is missing from each scale, the scale will not be calculated. Calculation of each scale score is provided below.<sup>7</sup>

### **Effectiveness**

$$([Q1 + Q2 + Q3) - 3]/18) * 100$$

If one item is missing then, ([Qx + Qy - 2]/12) \* 100 where x and y = 1, 2, or 3, with

### Side-Effects

If Q4 is 'No' then score = 
$$100$$

Else, 
$$([Q5 + Q6 + Q7 + Q8 - 4]/16) * 100$$

14 April 2017 33

If one item is missing then, ([Qx + Qy + Qz - 3]/12) \* 100 where x, y, and z = 5, 6, 7, or 8, with  $x\neq y\neq z$ .

### Convenience

$$([Q9 + Q10 + Q11) - 3]/18) * 100$$

### Global Satisfaction

$$([Q12 + Q13 + Q14) - 3]/14) * 100$$

2y + 2y + 100 where x and y = 9, 10, or 11.

Where x and y = 9, 10, or 11.

Where x and y = 12, 13, or 14.

Where x and y = 12, 13, or 14.

Where x and y = 12, 13, or 14.

Where x and y = 12, 13, or 14. Summarization and analysis of TSQM data will be performed for the mITT population. The 4 scale scores will be presented for Visit 2 (baseline) and Visit 4/ET, including change from baseline. For each score a paired t-test will be used to assess the within-group mean change from baseline. An analysis of covariance (ANCOVA), with treatment and baseline as covariates will be used for between-group comparison of change from baseline.

## 7.6.3.5.3. Intranasal Therapy Impact Questionnaire (ITIQ)

The ITIQ is a two item questionnaire that is completed by both the subject and caregiver at Visit 4/ET. The level of anxiety change since subject received intranasal therapy is a scale with a range from -7 to 7, and confidence about travelling having a spray the subject can take with them is a scale from 1 to 5. The change in level of anxiety since subject received intranasal therapy will be compared between treatment groups using the t-test. The chi-square will be used to compare treatment groups for confidence about travelling having a spray the subject can take with them.

#### 7.7. **Safety Analyses**

All safety analyses will be presented by phase of the study based on the Safety Population and Randomized Safety Population, unless otherwise specified.

#### Adverse Events (AEs) 7.7.1.

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 16.1. Coding includes SOC and preferred term (PT). All verbatim descriptions and coded terms will be listed for all AEs.

For subjects who screen fail prior to the start of the Test Dose Phase for the reason of an adverse event, the event will be recorded on the Screening Failure Log.

#### 7.731.1. **Pre-treatment AEs**

Pre-treatment AEs will be defined as any AE that started before the study drug administration at Visit 2. Pre-treatment AEs will be flagged out in a listing named as 'Adverse Events'.

#### 7.7.1.2. **Treatment-emergent AEs (TEAEs)**

TEAEs will be categorized as TEAEs during the Test Dose Phase and TEAEs during the Comparative Phase based on the date and time of onset.

Upsher-Smith Laboratories, Inc. Statistical Analysis Plan for Protocol No.: P261-401

The following AEs will be defined as TEAEs during the Test Dose Phase:

- AEs with onset on or after study drug administration at Visit 2 and up to first dose of study drug in Comparative Phase;
- Valiations thereof. • AEs that started prior to study drug administration at Visit 2, but worsened in severity following study drug administration at Visit 2 up to first dose of study drug in Comparative Phase.

The following AEs will be defined as TEAEs during the Comparative Phase:

- AEs with onset on or after the first dose of study drug in Comparative Phase;
- AEs that started prior to study drug administration at Visit 2, but worsened in severity following the first dose of study drug in Comparative Phase.

All AEs will be listed by subject and by MedDRA SOC and PT.

The number of events and the frequency and percentage of subjects with TEAEs/SAEs will be summarized for the Safety Population during the Test Dose Phase and for the Randomized Safety Population during the Comparative Phase. An overall summary of all AEs for Screened Population will also be presented. Summary tables of TEAEs and SAEs will be presented by SOC and PT. At each summary level, a subject will be counted only once for each AE he/she experiences within that level, regardless of how many occurrences of that AE that subject experienced. The percentage of subjects having had at least one TEAE/SAE at each level will be calculated. All the TEAE analysis will also be repeated for the subset of all TEAEs that started within two days of study drug administration.

Tabular summaries will include all TEAEs, TEAEs by age group (< 18 years, ≥18 - <65 years, ≥65 years), TEAEs by severity (mild, moderate, severe), TEAEs by relationship to study drug, TEAEs of interests, serious TEAEs (SAEs) including SAEs leading to permanent discontinuation or death, SAEs by severity, and SAEs by relationship to study drug. If there are any deaths while on study, they will be presented in a listing that includes the AE leading to death, demographic data, details of study treatment, and relationship of the AE leading to death to the study drug. In addition, all TEAEs, SAEs, and AEs leading to discontinuation will be flagged out in the listing of Adverse Events.

In instances where a subject may have multiple TEAEs with differing levels of severity or relatedness, the most severe or most related event, respectively, will be reported for the severity and relatedness tables. For the purpose of analysis, TEAEs with a reported relatedness of "Related", "Possibly Related", "Unlikely Related", or missing the relationship will be classified as related to study drug. TEAEs assessed as "Not Related" will be classified as not related to The following AEs of special interest (AESIs) will be summarized by AESI category:

• Taste and smell disorders

• Acute contact study drug. TEAEs with missing severity will be presented as severe in the tables but will be

- Route of administration

Upsher-Smith Laboratories, Inc. Statistical Analysis Plan for Protocol No.: P261-401

- Depression and suicidality/self-injury
- Abuse-related AEs

Abuse-related TEAEs will be further broken out by the following categories:

- , any extensions or variations thereof. • Drug Abuse, Dependence, Withdrawal and Substance-Related Disorders, Including Diversion
- Euphoria-related Term
- CNS Depressant Effects
- Stimulation and Anxiety Symptoms
- Perceptual Disturbances/Psychotomimetic Effects
- Mood Disorders and Disturbances
- Mental and Cognitive Impairment

Additional summaries will be made for abuse-related treatment-emergent SAEs and abuserelated TEAEs resulted in discontinuation from study drug or the study.

SMQs and/or a USL-defined algorithm will be used to search AESIs. Search strategies are described in Table 5.

**Search Strategy for AESI** Table 5:

| AESI category | Search Strategy |
|---|---|
| Taste and smell disorders | Modified Taste and Smell Disorders SMQ - broad |
| Acute central respiratory depression | Modified Acute Central Respiratory Depression SMQ - broad |
| Depression and suicidality/self-injury | Modified Depression and Suicidality/Self-Injury SMQ – broad |
| Route of administration | USL-defined [Oral Soft Tissue Conditions HLT (Gastrointestinal Disorders SOC); Respiratory Disorders NEC (Respiratory, Thoracic and Mediastinal Disorders SOC); Upper Respiratory Tract Disorders (Exclude Infections) (Respiratory, Thoracic and Mediastinal Disorders SOC)] – excluding overlapping terms with Acute Central Respiratory Depression SMQ and terms unrelated to USL261's nasal route of administration, e.g., terms for conditions in the respiratory tract below the larynx or terms with defined causes |
| Abuse-related AEs | USL-defined algorithm |

Abbreviations: HLT=High Level Term; SMQ=Standardized MedDRA Queries; NEC=Not Elsewhere Classified.

Standard MedDRA Queries (SMQs) defined by the Council for International Organizations of Medical Sciences (CIOMS) Working Group are groupings of terms from one or more MedDRA SOCs that relate to a defined medical condition or area of interest. Modifications of SMQs will be documented. For hierarchical SMQs, the portion of the hierarchy to be used will be that part or those parts determined to be most relevant. A list of AE terms in each category is presented in Appendix 3. Summary tables will be presented by SOC and PT.
In addition, potentially clinically important AESI will be presented for each category of AESI. AE which meets at least one of the following criteria is defined as a potentially clinically important AE:

- AE is a SAE
- AE led to discontinuation
- AE is severe in intensity and related to study drug
- AE required intervention and is related to study drug.

If action taken and other action taken of a AE are not "none", "not applicable", "unknown" "dose not changed", then it will be considered requiring intervention.

#### 7.7.2. **Observer's Assessment of Alertness/Sedation (OAA/S)**

The OAA/S scale is a validated qualitative categorical measure of sedation. The OAA/S Scale is composed of four assessment categories: responsiveness, speech, facial expression, eyes. Responsiveness has possible scores of 1, 2, 3, 4, or 5; speech has scores of 2, 3, 4, or 5; and facial expression and eyes have scores of 3, 4, or 5. The OAA/S Scale is scored in two ways as described below. Descriptive statistics and graphical presentations will be used to present results by time point at Visit 2 for the Safety Population.

#### 7.7.2.1. **Composite Score**

The composite score has a range between 1 (deep sleep) and 5 (alert); the lowest level checked by the study center personnel in any one of the four assessments will be analyzed. The composite score will be set to missing if all 4 of the assessment categories are missing.

Number of subjects with an OAA/S composite score of 1 at Visit 2 will be presented by time point and overall total.

#### 7.7.2.2. **Sum Score**

The sum score is the sum of the 4 assessments. If one of the assessment categories is missing, the sum score will be set to missing.

Summaries for the composite score and sum score will be based on the calculation specified above. However, an imputation approach on each domain score will be employed for the derivation of pharmacodynamic parameters described in the next section. Specifically, for each individual domain score, if a subject who has completely missing data at all timepoints for a single domain, the median domain score of all available data from all other subjects at each timepoint will be used as the domain score for this subject. For subjects with complete missing scores for two or more domains at all timepoints, each domain score will be treated as missing at all timepoints and OAA/S sum and composite scores will not be calculated.

#### 7.7.2.3. Pharmacodynamic (PD) Parameters

The following PD parameters will be calculated by subject using non-compartmental methods for the OAA/S composite score and sum score following midazolam dosing:

**Table 6:** Pharmacodynamic Parameters

| Parameter | Definition |
|---|---|
| AUEC <sub>0-t</sub> | Area under the effect (AUEC) versus time curve, from time 0 to the time of last |
| | measurable value. Calculated using the linear trapezoidal method. |
| AUEC <sub>0-x</sub> | Area under the effect (AUEC) versus time curve, calculated using the linear |
| | trapezoidal method from time 0 to the x time, where $x = 1, 2$ and 4 hours. |
| $E_{max}$ | Maximum observed PD effect. Note – For OAA/S sum and composite scores |
| | this will represent the lowest observed score (as lower scores indicate greater |
| | sedation) |
| Teffect | Time to Peak "E <sub>max</sub> " Effect |

Among these parameters, the calculated OAA/S sum score and composite score will be used for calculating the unadjusted  $E_{max}$ . The  $E_{max}$  will also be adjusted by using change from baseline values of OAA/S composite score and sum score. For parameters AUEC<sub>0-t</sub>, AUEC<sub>0-x</sub> (x=1, 2, 4), the calculation will be based on the change from baseline values of OAA/S composite score and sum score.

Actual time will be used for AUEC calculation. If actual time for pre-dose values is before the Test dose, 0 will be used for time point calculation. If equal to or greater than 50% domain data for a subject is missing, then all their AUEC values (including AUEC<sub>0-last</sub>, AUEC<sub>0-1hr</sub>, AUEC<sub>0-2hr</sub> and AUEC<sub>0-4hr</sub>) will be treated as missing. If less than 50% domain data for a subject is missing, then last observation carried forward approach will be used to impute all missing time points after the last non-missing time point.

Individual PD parameter values will be listed and descriptive statistics will be used to present PD parameters at Visit 2 for the Safety Population.

# 7.7.3. Requirement for Unscheduled ER or EMS Visit

The number and percent of subjects requiring an unscheduled ER or EMS visit within 24 hours after study drug administration in the Comparative Phase will be compared between treatment groups for the Randomized Safety Population using Fisher's Exact Test. In addition, Chi-squared test will be performed as a sensitivity analysis.

# 7.7.4. Brief Smell Identification Test (B-SIT; United States only)

For olfactory examination, the B-SIT final scores and changes from baseline will be presented and plotted by visits. Baseline value is defined as the Visit 2 (pre-dose) value. An analysis of covariance (ANCOVA), with treatment and baseline as covariates, will be used for between-group comparison of change from baseline for the B-SIT final scores.

## 7.7.5. Columbia-Suicide Severity Rating Scale (C-SSRS)

The C-SSRS is collected referencing two time points for suicidal ideation (lifetime, past 6 months) and two time points for suicidal behavior (lifetime, past 5 years) at Visit 1 (screening). For all analyses the 'lifetime' time point will be used for Visit 1 assessments. In addition, a 'Since Last Visit' version will be administered at Visits 2, 3 and 4/ET.

14 April 2017 38

### 7.7.5.1. Suicidal Ideation

The number and percent of subjects with each of the following suicidal ideation scores will be summarized for each visit by treatment group (See Table 7). The highest score for suicide ideation will be used for each subject by visit.

**Table 7:** Suicidal Ideation Scores

| Suicidal ideation | Score |
|---|---|
| Wish to be dead | 1 |
| Non-specific active suicidal thoughts | 2 |
| Active suicidal ideation with any methods (not planned) without intent to act | 3 6 |
| Active suicidal ideation with some intent to act, without specific plan | 4:01 |
| Active suicidal ideation with specific plan and intent | 5 |

Any suicidal ideation regardless of type will also be presented.

Each suicidal ideation severity rating will range from 0 (no ideation present) to 5 (active ideation with plan of intent). Descriptive statistics will be presented for suicidal ideation severity rating at each visit by treatment group.

Descriptive statistics will also be presented for suicidal ideation intensity at each visit by treatment group. The five intensity items (frequency, duration, controllability, deterrents, and reason for ideation) will be combined to create a total, sum score ranging between 0 and 25. If the subject did not have any suicidal ideation, the total score will be 0. If the subject had suicidal ideation and if one intensity item is missing, the total score will not be calculated.

## 7.7.5.2. Suicidal Behavior

The number and percent of the following suicidal behaviors will be summarized for each visit by treatment group.

- Actual attempt
- Engaged in non-suicidal self-injurious behavior
- Aborted attempt
- Interrupted attempts
- Preparatory acts or behavior
- Suicidal behavior
- Any suicidal behavior regardless of type
- Completed suicide

Descriptive statistics will be presented for the following suicidal behaviors for each visit by treatment group.

- Number of attempts
- Aborted attempts

14 April 2017 39

## Interrupted attempts

The number and percent of subjects with any suicidal ideation or behavior will be presented for each visit by treatment group.

The number and percent of patients having normal and abnormal findings (clinically significant vs. not clinically significant) for each body system or assessment will be presented by visit and treatment group for the Safety and Randomized Safety Population

Clinical laboratory parameters for serum chemistry, hematology, and urinalysis will be summarized descriptively for each study visit. Mean and mean change from beautimeasurement minus that summarized descriptively for each study visit. Mean and mean change from baseline values will missing, the observation will not be included in the change from baseline summary. The last value at post-baseline visits will be used for summaries.

Each laboratory result will be classified as low (L), normal (N), and high (H) at each visit according to the laboratory-supplied normal range. The shift from baseline will be presented. Potentially clinically significant (PCS) laboratory abnormalities will be identified using standardized criteria in Appendix 1 prior to database lock and will be presented by for each treatment group. Additional displays of PCS may be presented.

Baseline values are the last available values collected prior to the test-dose.

#### Vital Signs and Oxygen Saturation 7.7.8.

Vital signs (systolic and diastolic blood pressure, pulse, respiration rate, temperature) will be summarized descriptively for each study visit and time point and presented graphically (excluding temperature) for each Visit 2 time point. Mean and mean change from baseline values will be presented for each study visit and time point, excluding temperature. Change from baseline will be calculated as post-baseline measurement minus baseline measurement. If either the baseline or post-baseline value is missing, the observation will not be included in the change from baseline summary. Baseline values are the last available values before Test-Dose administration.

Descriptive statistics and graphical presentations will be used to present results by visit and time point for oxygen saturation for the Safety Population.

The number of subjects meeting the following criteria will be presented by treatment group, by visit, and by time point:

- < 8 breaths per minute after study drug administration
- > 24 breaths per minute after study drug administration
- systolic blood pressure < 85 mm Hg
- a change from baseline in systolic pressure ≥ 40 mm Hg

- diastolic blood pressure < 50 mm Hg
- a change from baseline in diastolic pressure  $\geq 30$  mm Hg
- Pulse rate > 120 beats per minute
- Pulse rate < 50 beats per minute
- a change from baseline in heart rate  $\geq 40$  beats per minute
- oxygen saturation < 90%

Valiations thereof. The caregiver-recorded respiration rate from the Comparative Phase will be presented using descriptive statistics at 15 minutes, 30 minutes, 1 hour, 2 hours, and 4 hours by treatment group and overall total for the Randomized Safety Population. The number of subjects who have < 8 and > 24 breaths per minute will be presented by time point, treatment group, and overall total.

#### 7.7.9. Electrocardiogram (ECG)

Electrocardiogram (ECG) parameters (heart rate, PR interval, RR interval, QRS interval, QT interval, and QTc interval) will be summarized descriptively for each scheduled visit and time point collected for the Safety Population. Mean and mean change from baseline values at Visit 2 will be presented. Change from baseline will be calculated as post-baseline measurement minus baseline measurement. If either the baseline or post-baseline value is missing, the observation will not be included in the change from baseline summary. In addition, counts and percentages for ECG diagnosis (normal or abnormal) at each study visit and time point will also be presented. If the diagnosis was abnormal, counts and percentages for clinical significance will be presented. Baseline values are the last available values before Test-Dose administration.

The number of subjects meeting the following criteria will be presented by treatment group for the Safety Population:

• QTcF interval > 450 msec for males and > 470 msec for females

## OTHER PLANNED ANALYSES 8.

#### Pharmacokinetic (PK) Analyses 8.1.

Pharmacokinetic parameters for individual plasma concentrations will be calculated using a standard non-compartmental approach using appropriate validated PK software (WinNonlin Enterprise version 5.2 or higher). The following PK parameters of midazolam and 1hydroxymidazolam will be calculated from data obtained for the PK Population:

- AUC<sub>0-last</sub> the area under the plasma concentration-time curve from time 0 to the last measurable concentration. Estimation by the linear-up/log-down trapezoidal method is preferred.
- $AUC_{0-x}$  the area under the plasma concentration-time curve from time 0 to time x, where x = 1, 2 and 4 hours.
- C<sub>max</sub> the maximum plasma concentration
- t<sub>max</sub> the time to reach the maximum plasma concentration

 $t_{lag}$  – the time before the first measurable plasma concentration

Due to the limited length of the PK sampling schedule (out to a maximum of 4 hrs post dose), it Pre-dose concentration values reported as below the limit of quantification (BLQ) and missing pre-dose values will be treated as "0" and listed as BLQ. A series of BLQ values that include the pre-dose time point will also be treated as "0" and listed as BLQ. A series of BLQ values that include the pre-dose time point will also be treated as "0" and listed as BLQ. is unlikely that sufficient samples will be available for estimation of the terminal rate constant

With the exception of  $t_{max}$  and  $t_{lag}$ , descriptive statistics by treatment group will include the number of observations (N), mean, standard deviation (SD), coefficient of variation (CV%), geometric mean, and geometric CV%, as well as median, minimum, and maximum for the PK variables. Summary statistics for t<sub>max</sub> and t<sub>lag</sub> will be limited to N, minimum, maximum and median. In addition, summary of PK variables stratified by AED inducer status as well as figures of Midazolam and 1-OH Midazolam concentrations on linear and semi-log scales will also be presented.

A covariate analysis that examines the effect of continuous (age, weight) and, if supported, categorical (gender, race, and age group [adult vs adolescent]) demographic variables on the PK parameters may be conducted.

## Pharmacokinetic/Pharmacodynamic Variables and Analyses 8.2.

Correlations between PK/PD data from the test dose may be evaluated. If conducted, the PK/PD analysis may include correlating the plasma midazolam plus 1-hydroxymidazolam concentrations to respiratory rate, BP, HR, O<sub>2</sub> saturation, and/or sedation based on OAA/S scores. Regression analysis may be used describe the PK/PD relationship, if one exists. For those PD measurements found to correlate to plasma concentrations, the influence of covariates such as gender, AED inducer status, weight, BMI, race, and age group may be explored.

#### CHANGES TO THE PLANNED ANALYSIS 9.

Since the last submission of the P261-401 Statistical Analysis Plan (v2.4) to the FDA (S-0150, 03 March 2015), the following changes were made to the plan (v2.5-v2.9):

- The Brief Smell Identification Test (B-SIT) was added to the list of safety objectives. The plan for analysis of B-SIT data was also added. These changes were made to reflect the changes implemented in Protocol Amendment 4, 20 May 2015.
- The procedures to be completed at Visits 1, 4, and on the monthly telephone followup calls between Visit 3 and Visit 4 were updated to add collection of the number of calls to EMS and ER visits for a seizure cluster or other seizure emergency prior to Visit 1 and during the study. This change was made to reflect the changes implemented in Protocol Amendment 4, 20 May 2015.

- The process for reviewing CSR Reportable protocol deviations and exclusions prior to database lock was clarified to determine if any subject should be excluded from specific analysis populations.
- The subgroup analyses of the primary and secondary endpoints were further clarified to examine consistency as follows:
- The time-frame around the use of enzyme-inducing AEDs was defined as within 14 days before study drug administration. Population PK modeling of deinduction half-life following deinduction half-life following times for strong CYP3A4 inducers, including carbon deinduction half-life following times for strong CYP3A4 inducers, including carbon deinduction half-life following carbon deinduction deindu return to baseline function occurring within approximately 14 days following discontinuation of dosing. Based on these estimates, a subject should be classified as "induced" if they have received an enzyme-inducing AED  $\leq$  14 days prior to administration of USL261.
  - The weight will be categorized based on the median weight for the safety population (< median weight and  $\ge$  median weight). This categorization based on the median weight was chosen to be representative of the population studied.
  - The BMI will be categorized as underweight/normal (< 25), overweight ( $\ge 25$  to <30), and obese 1-3 categories combined ( $\geq$ 30). This categorization was based on standard BMI categories.
  - The subgroups frequency of seizure clusters and benzodiazepine use was removed as these subgroups are based on historic data and may not represent the seizure cluster frequency or benzodiazepine use relative to administration of study drug in the Comparative Phase.
  - The subgroups seizure types (generalized and focal) and seizure etiology were removed.
- For subjects who were rescreened and underwent two Test Dose Visits, baseline will be defined as the last available values before the later Test Dose administration. This clarification was provided to prespecify how baseline is defined in a unique situation.
- An additional exploratory efficacy analysis, "treatment success of all doses of study drug," was included in the plan. This exploratory analysis was added to assess the Treatment Success of the first dose and Treatment Success of the second dose (taken within 6 hours) during the Comparative Phase.
- The definition of a treatment-emergent adverse event (TEAE) in the Test Dose Phase and in the Comparative Phase was clarified. This clarification was made to clearly define the phase in which TEAEs will be reported. However, it does not impact the definition of a TEAE or the total TEAEs reported.
- The AEs of special interest (AESI) and abuse-related AEs were defined.
- Additional detail for the calculation of the following PD parameters: OAA/S sum score, AUEC<sub>0-t</sub>, AUEC<sub>0-x</sub>, and E<sub>max</sub> was added.

An early study termination analysis unrelated to study success or futility was added in the event that the trial has not crossed a boundary for early success or early futility DATA LISTINGS

REFERENCES

1. Cereghino JJ. Identification and treatment of acute repetitive seizures in children and adults. Curr Treat Options Neurol. 2007;9:249-255.

2. Lowenstein DH, Alldredge BK. Status epilepticus. N Engl J Med. 1988-220

3. Glauser TA. Designing practical evidence-based treatment prolonged seizures and status epilepticus. J Children and Status epilepticus epilepti and yet is stopped early before reaching the pre-specified maximum sample size of

# 10.

The mock TLGs will be provided in a separate document.

## 11.

- 5. Utah Department of Health. Interpreting the SF12. 2001 Utah Health Status Survey. 2001: 1-17.
- 6. Web. < http://www.ncbi.nlm.nih.gov/pmc/articles/PMC1434659/>
- 7. Web. <www.qualitymeasures.ahrq.gov
- 8. Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and Reliability of the Observer's Assessment of Alertness/Sedation This document cannot be used to support any Scale: Study with Intravenous Midazolam. J of Clin Psychopharmacology. 1990: 10:

# APPENDIX 1. POTENTIALLY CLINICALLY SIGNIFICANT LABORATORY VALUES

**Potentially Clinically Significant Laboratory Values** Table 8:

| Variable | Units | Values | l III:ak |
|---|---|---|---|
| | | Low | High |
| Haematology | 1 /- | 100 | 1 |
| Haemoglobin | g/L | < 100 | Not applicable |
| | g/L | > 20 decrease | > 20 increase |
| Lymphocytes (Absolute) | 10 <sup>9</sup> /L | from baseline < 0.8 | ULN Not applicab |
| | 10°/L<br>10°/L | < 1.5 | |
| Neutrophils (Absolute) | | | Not applicable |
| Platelet count | 10 <sup>9</sup> /L | < 75 | Not applicable |
| White blood cell (WBC) count | 10 <sup>9</sup> /L | < 3 | Not applicable |
| Serum Chemistry | /* | | |
| Albumin | g/L | < 30 | Not applicab |
| Alkaline phosphotase (AP) | U/L | Not applicable | > 2.5xULN |
| Alanine aminotransferase (ALT) Grade 1 | U/L | Not applicable | > ULN & ≤ 3 |
| Alanine aminotransferase (ALT) Grade 2 | U/L | Not applicable | > 3xULN & : |
| Alanine aminotransferase (ALT) Grade 3 | U/L | Not applicable | > 5xULN & |
| Alanine aminotransferase (ALT) Grade 4 | UVE | Not applicable | > 20xULN |
| Aspartate aminotransferase (AST) Grade 1 | TUK. | Not applicable | $>$ ULN & $\leq 3$ |
| Aspartate aminotransferase (AST) Grade 2 | Ø/Ĺ | Not applicable | > 3xULN & |
| Aspartate aminotransferase (AST) Grade 3 | U/L | Not applicable | > 5xULN & : |
| Aspartate aminotransferase (AST) Grade 4 | U/L | Not applicable | > 20xULN |
| Bicarbonate | mmol/L | ≤ 15.9 | Not applicab |
| Calcium | mmol/L | < 2 | > 2.9 |
| Cholesterol (Total) | mmol/L | Not applicable | > 7.75 |
| Creatinine | umol/L | Not applicable | > 1.5xULN |
| | umol/L | Not applicable | > 2x baseline |
| Gamma glutamyl transferase (GGT) | U/L | Not applicable | > 2.5xULN |
| Glucose | mmol/L | < 3.0 | > 8.9 |
| Phosphorus | mmol/L | < 0.8 | Not applicab |
| Potassium | mmol/L | < 3.0 | > 5.5 |
| Sodium | mmol/L | < 130 | > 150 |
| Total Bilirubin | umol/L | Not applicable | > 1.5xULN |
| (1) | mmol/L | Not applicable | > 3.42 |
| Sodium | mmol/L<br>umol/L | < 130<br>Not applicabl | |

## APPENDIX 2. CLASSIFICATION OF ENZYME INDUCING AEDS

Table 9: **Listing of Non-Enzyme Inducing AEDs** 

| | of Non-Enzymo | 9 and Table 10 do not represent an exhaustive list. reviewed and assigned. 9 Inducing AEDs Inducing AEDs Proposition and any extensions of waite industrial and any extensions where the action and any extensions and any extension and any extensions and extensions are actions and extensions and extensions and extensions are actions and extensions and extensions are actions as a constant and extensions are actions and extensions are actions as a constant action and extensions are actions as a constant and extensions are actions as a constant action and extensions are actions as a constant action and extensions are actions |
|---|---|---|
| AED name | Reference | |
| Acetazolamide | [1] | atio. |
| Chloral Hydrate | [2] | |
| Chlorazepate | [3] | |
| Clonazepam | [4] | |
| Diazepam | [5] | ion |
| Ethosuximide | [6] | 3/1/5 |
| Gabapentin | [7] | The state of the s |
| Lacosamide | [8] | 46. |
| Lamotrigine | [9] | Service of the service of the servic |
| Levetiracetam | [10] | ano |
| Lorazepam | [11] | |
| Midazolam | [12] | ijo, |
| Oxazepam | [13] | |
| Perampanel | [14] | 04 006. |
| Pregabalin | [15] | COX COX |
| Retigabine (ezogabine) | [16] | o atio |
| Гiagabine | [17] | XXX :10 |
| Valproic Acid, | [18] | C,*10, |
| Valproate, Divalproex | | Or any |
| Sodium | 0 | |
| Vigabatrin | [6] | etti. |
| Zonisamide | [19] | |

| AED name | Strength of inducer <sup>a</sup> | Reference |
|---|---|---|
| Carbamazepine | Strong | [20] |
| Clobazam | Weak | [21] |
| Eslicarbazepine | Weak (borderline moderate) | [22] |
| Ethotoin | Strong (assumed from <i>in vitro</i> induction vs. phenytoin) | [23] |
| Felbamate | Weak | [24] |
| Mephenytoin | Strong (assumed from <i>in vitro</i> induction vs. phenytoin) | [23] |
| Oxcarbazepine | Weak (borderline moderate) | [25] |
| Phenobarbital | Strong | [26, 27] |
| Phenytoin | Strong | [20] |
| Primidone | Strong (via phenobarbital major metabolite) | [26, 27] |
| Rufinamide | Weak | [20] |
| Topiramate | Weak (only at doses > 200 mg/day) | [28] |

<sup>&</sup>lt;sup>a</sup> Based on decrease in AUC of CYP3A4 substrate [20]: Weak = 20 - 50% decrease, Moderate = 50 - 80% decrease, Strong =  $\geq 80\%$  decrease

## Washout period required for deinduction following discontinuation of inducing AEDs.

Population PK modeling of deinduction times for strong CYP3A4 inducers, including or variations thereof. carbamazepine, indicates a deinduction half-life following discontinuation of approximately 3-4 days with return to baseline function occurring within approximately 14 days following discontinuation of dosing [29-32]. Based on these estimates, a subject should be classified as "induced" if they have received an enzyme-inducing AED < 14 days prior to administration of USL261.

## References

- 1. Spina, E., F. Pisani, and E. Perucca, *Clinically significant pharmacokinetic drug interactions* with carbamazepine. An update. Clin Pharmacokinet, 1996. 31(3): p. 198-214.
- 2. Perrigo, Chloral Hydrate Mixture. 2006.
- 3. Lundbeck, Tranxene T-Tab (clorazepate dipotassium) [Prescribing Information]. 2009.
- 4. Roche, Klonopin (clonazepam) [Prescribing Information]. 2009.
- 5. Valeant Pharmaceuticals, Diastat Accudial (diazepam) [Prescribing Information]. 2006.
- 6. Riva, R., et al., Pharmacokinetic interactions between antiepileptic drugs. Clinical considerations. Clin Pharmacokinet, 1996. 31(6): p. 470-93.
- 7. Pfizer, Neurontin (gabapentin) [Prescribing Information], 2014.
- 8. UCB, Vimpat (lacosamide) [Prescribing Information]. 2011.
- 9. GlaxoSmithKline, Lamictal (lamotrigine) [Prescribing Information]. 2012.
- 10. UCB, Keppra (levetiracetam) [Prescribing Information]. 2013.
- 11. West-Ward Pharmaceuticals, Ativan (lorazepam) [Prescribing Information]. 2011.
- 12. Hospira, Midazolam Injection, USP [Prescribing Information]. 2009.
- 13. Alphapharm, Alepam (oxazepam) [Prescribing Information]. 2013.
- 14. Eisai, Fycompa (perampanel) [Prescribing Information]. 2013.
- 15. Pfizer, Lyrica (pregabalin) [Prescribing Information]. 2013.
- 16. GlaxoSmithKline, Potiga (ezogabine) [Prescribing Information]. 2013.
- 17. Cephalon, Gabitril (tiagabine hydrochloride) [Prescribing Information]. 2012.
- 18. AbbVie, Depakote (divalproex sodium) [Prescribing Information]. 2015.
- 19. Eisai, Zonegran (zonisamide) [Prescribing Information]. 2012.
- 20. U.S. Food and Drug Administration, Draft Guidance: Drug Interaction Studies Study Design, Data Analysis, Implications for Dosing, and Labeling Recommendations. 2012.
- 21. Lundbeck, ONFI (clobazam) [Prescribing Information]. 2013.
- 22. Sunovion Pharmaceuticals, Aption (eslicarbazepine acetate) [Prescribing Information]. 2013.
- 23. Kobayashi, K., et al., Key structural features of ligands for activation of human pregnane X receptor. Drug Metab Dispos, 2004. 32(4): p. 468-72.
- 24. Meda Pharmaceuticals, Felbatol (felbamate) [Prescribing Information]. 2011.
- 25. Novartis, Trileptal (oxcarbazepine) [Prescribing Information]. 2013.
- 26. Back, D.J., et al., The interaction of phenobarbital and other anticonvulsants with oral contraceptive steroid therapy. Contraception, 1980. 22(5): p. 495-503.
- 27. Ripp, S.L., et al., Use of immortalized human hepatocytes to predict the magnitude of clinical drug-drug interactions caused by CYP3A4 induction. Drug Metab Dispos, 2006. 34(10): p. 1742-8.
- 28. Janssen Pharmaceuticals, Topamax (topiramate) [Prescribing Information]. 2012.

- 29. Baneyx, G., et al., Physiologically based pharmacokinetic modeling of CYP3A4 induction by rifampicin in human: influence of time between substrate and inducer administration. Eur J Pharm Sci, 2014. **56**: p. 1-15.
- 30. Brodie, M.J., et al., Enzyme induction with antiepileptic drugs: cause for concern? Epilepsia,
- 31. Punyawudho, B., et al., Characterization of the time course of carbamazepine deinduction by
- Schaffler, L., B.F. Bourgeois, and H.O. Luders, Rapid reversibility of autoinduction of carbamazepine metabolism after temporary discontinuation. Epilepsia, 1994. **35**(1): p. 195-8. aduction of 1994. 35(1): p. 1. 1

# APPENDIX 3. LIST OF AE TERMS OF SPECIAL INTEREST

# **Table 11:** Abuse-related AEs (MedDRA Preferred Term)

| Drug Abuse, Dependence, Withdrawal and Substa | ance-Related Disorders, Including Diversion |
|---|---|
| Accidental death | Multiple drug overdose intentional |
| Accidental overdose | Nasal necrosis |
| Accidental poisoning | Nasal septum perforation |
| Dependence | Nasal septum ulceration |
| Drug abuser | Needle track marks |
| Drug administered at inappropriate site | Neonatal complications of substance abuse |
| Drug dependence | Overdose |
| Drug detoxification | Poisoning |
| Drug diversion | Polysubstance dependence |
| Drug tolerance | Prescription form tampering |
| Drug tolerance increased | Product tampering |
| Drug toxicity | Product used for unknown indication |
| Drug Withdrawal | Rebound effect |
| Drug withdrawal convulsions | Substance abuse |
| Drug withdrawal headache | Substance abuser |
| Drug withdrawal syndrome | Substance use |
| Intentional drug misuse | Substance-induced mood disorder |
| Intentional overdose | Substance-induced psychotic disorder |
| Multiple drug overdose | Treatment noncompliance |
| Multiple drug overdose accidental Withdrawal Syndrome | |
| Euphoria-related Terms | <i>b</i> |
| Dizziness | Feeling drunk |
| Elevated mood | Feeling of relaxation |
| Euphoric mood | Inappropriate affect |
| Feeling abnormal | |
| CNS Depressant Effects | |
| Fatigue | Sluggishness |
| Lethargy | Somnolence |
| Sedation | Stupor |
| Stimulation and Anxiety Symptoms | |
| Agitation | Hypervigilance |
| Anxiety | Nervousness |
| Energy increased | Psychomotor hyperactivity |
| Feeling jittery | Restlessness |
| Perceptual Disturbances/Psychotomimetic Effects | <u></u> |
| Abnormal dreams | Hallucinations, mixed |
| Acute psychosis | Hostility |
| Aggression | Hypoaesthesia |
| Alice in wonderland syndrome | Ideas of reference |
| Altered state of consciousness | Illogical thinking |
| Altered visual depth perception | Illusion |
| • | |

14 April 2017 49

| Anger | Incoherent |
|---|---|
| Communication disorder | Indifference |
| Confusional state | Jamais vu |
| Consciousness fluctuating | Loose associations |
| Déjà vu | Magical thinking |
| Delirium Delirium | Muscle rigidity |
| Delusion | Nightmare |
| Depersonalisation | Paraesthesia |
| Derailment | Paranoia |
| Derealisation | Paroxysmal perceptual alteration |
| Disinhibition | Psychotic disorder |
| Disorientation | Reactive psychosis |
| Dissociation | Sensory disturbance |
| Dissociative disorder | Sensory level abnormal |
| Dissociative disorder | Somatic delusion |
| Dysarthria | Somatic detasion Somatic hallucination |
| Fear | Staring |
| Flashback | Suspiciousness |
| Flight of ideas | Tangentiality |
| Formication | Thinking apnormal |
| Hallucination | Thought blocking |
| Hallucination, auditory | Thought broadcasting |
| Hallucination, olfactory | Thought insertion |
| Hallucination, synaesthetic | Thought withdrawal |
| Hallucination, tactile | Transient psychosis |
| Hallucination, visual | Transient psychosis |
| Mood Disorders and Disturbances | |
| Abnormal behaviour | Asocial behaviour |
| Affective disorder | Attention-seeking behaviour |
| Affect lability | Belligerence |
| Depressed mood | Blunted affect |
| Depression Superior S | Compulsions |
| Emotional disorder | Confusional arousal |
| Emotional distress | Disturbance in social behaviour |
| Impatience | Feeling of despair |
| Mood altered | Flat effect |
| Mood swings | Impulsive behaviour |
| Personality change | Mania |
| Anhedonia | Panic attack |
| Antisocial behaviour | Panic reaction |
| Apathy | Parasomnia |
| Mental and Cognitive Impairment | |
| Amnesia Mental disorder | |
| Cognitive disorder | Mental status changes |
| Disturbance in attention | Paramnesia |

14 April 2017 50

| Memory impairment | Psychomotor retardation | Psychomotor retardation |
|---|---|---|
| Mental impairment | Retrograde amnesia | Retrograde amnesia |
| Psychomotor skills impaired | Transient global amnesia | |
| Amnestic disorder | Impaired driving ability | Impaired driving ability |
| Anterograde amnesia | Impaired reasoning | Impaired reasoning |
| Balance disorder | Dyslogia | Dyslogia |
| Coordination abnormal | Bradyphrenia | Bradyphrenia |
| Executive dysfunction | Confabulation | Confabulation |
| Judgement impaired | 170 | 1/0 |

**Table 12:** 

| Judgement impaired | | 10 |
|---|---|---|
| Table 12: AEs Related to | Acute Central Respiratory Dep | pression (SMQ) Rejolie |
| System Organ Class | Preferred Term | Lowest Level Term |
| Acute central respiratory depress | Acute central respiratory depression (SMQ) | |
| Cardiac disorders | Cyanosis | Acrocyanosis |
| Cardiac disorders | Cardiac arrest | Arrest cardiac |
| Cardiac disorders | Cardiac arrest | Asystole |
| Cardiac disorders | Cardiac arrest | Asystolia |
| Cardiac disorders | Cardiac arrest | Asystolic |
| Cardiac disorders | Cyanosis | Blue lips |
| Cardiac disorders | Cardiac arrest Cyanosis Cardiac arrest Cordiac arrest | Cardiac arrest |
| Cardiac disorders | Cardiac arrest | Cardiac arrest transient |
| Cardiac disorders | Cardio-respiratory arrest | Cardio-respiratory arrest |
| Cardiac disorders | Cardio-respiratory arrest | Cardiopulmonary arrest |
| Cardiac disorders | Cardiac arrest | Congestive cardioplegia |
| Cardiac disorders | Cyanosis | Cyanosed |
| Cardiac disorders | Cyanosis | Cyanosis |
| Cardiac disorders | Cyanosis | Cyanosis NOS |
| Cardiac disorders | Cyanosis | Cyanosis of lip |
| Cardiac disorders | Cyanosis | Cyanosis peripheral |
| Cardiac disorders | Cyanosis | Cyanotic |
| Cardiac disorders | Cardiac arrest | Heart arrest |
| Cardiac disorders | Cardiac arrest | Hypoxic arrest |
| Cardiac disorders | Cyanosis | Lips cyanosed |
| Cardiac disorders | Cyanosis | Nails cyanosed |
| Cardiac disorders | Cardiac arrest | Standstill cardiac |
| Cardiac disorders | Cardiopulmonary failure | Cardio-respiratory failure |
| Cardiac disorders | Cardio-respiratory distress | Cardio-respiratory distress |
| Cardiac disorders | Cardiopulmonary failure | Cardiopulmonary insufficiency |
| Cardiac disorders | Cardiopulmonary failure | Cardiopulmonary failure |
| Cardiac disorders | Cyanosis | Circumoral cyanosis |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depressi- | on (SMQ) | |
| Cardiac disorders | Cyanosis | Cyanosis aggravated |
| Infections and infestations | Severe acute respiratory syndrome | Severe acute respiratory syndrome |
| Infections and infestations | Severe acute respiratory syndrome | SARS |
| Injury, poisoning and procedural complications | Respiratory fume inhalation disorder | Respiratory fume inhalation disorder NOS |
| Injury, poisoning and procedural complications | Respiratory fume inhalation disorder | Upper respiratory inflammation due to fumes and vapors |
| Injury, poisoning and procedural complications | Respiratory fume inhalation disorder | Upper respiratory inflammation due to fumes and vapours |
| Injury, poisoning and procedural complications | Respiratory fume inhalation disorder | Smoke inhalation |
| Injury, poisoning and procedural complications | Respiratory fume inhalation disorder | Respiratory fume inhalation disorder |
| Injury, poisoning and procedural complications | Postoperative respiratory failure | Postoperative respiratory failure |
| Investigations | Blood gases abnormal | ABGs abnormal |
| Investigations | Blood gases abnormal | Abnormal arterial blood gases |
| Investigations | Breath sounds abnormal | Abnormal chest sounds |
| Investigations | Breath sounds abnormal | Abnormal chest sounds NOS |
| Investigations | Blood gases abnormal | Blood gases abnormal |
| Investigations | Blood gases abnormal | Blood gases NOS abnormal |
| Investigations | Blood pH abnormal | Blood pH abnormal |
| Investigations | Blood pH decreased | Blood pH decreased |
| Investigations | Breath sounds abnormal | Breath sounds decreased |
| Investigations | Respiratory rate decreased | Breathing rate slowed |
| Investigations | Respiratory rate decreased | Breathing slowed |
| Investigations | Breath sounds abnormal | Diminished lung sounds |
| Investigations | Blood pH decreased | Low pH |
| Investigations | Oxygen saturation abnormal | Oxygen saturation abnormal |
| Investigations | Oxygen saturation decreased | Oxygen saturation decreased |
| Investigations | Oxygen saturation decreased | Oxygen saturation low |
| Investigations | PO2 abnormal | Oxygen tension abnormal NOS |
| Investigations | PO2 decreased | Oxygen tension decreased |
| Investigations | PCO2 decreased | Partial pressure CO2 decreased |
| Investigations | PO2 abnormal | Partial pressure O2 abnormal NOS |
| Investigations | PO2 decreased | Partial pressure O2 decreased |
| Investigations | PCO2 decreased | PCO2 decreased |
| Investigations | Blood pH decreased | pH decreased |
| Investigations | Blood pH decreased | pH reduced |
| Investigations | Blood pH decreased | Plasma pH decreased |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depre | ession (SMQ) | |
| Investigations | PO2 abnormal | PO2 abnormal NOS |
| Investigations | PO2 decreased | PO2 decreased |
| Investigations | PCO2 decreased | Reduced CO2 tension |
| Investigations | Respiratory rate decreased | Respiration rate decreased |
| Investigations | Respiratory rate decreased | Respiratory rate decreased |
| Investigations | Respiratory rate decreased | Respiratory rate low |
| Investigations | Breath sounds abnormal | Respiratory sounds decreased |
| Investigations | Blood pH decreased | Serum pH decreased |
| Investigations | Oxygen saturation abnormal | Oximetry abnormal |
| Investigations | Oxygen saturation decreased | Oximetry decreased |
| Investigations | Blood pH decreased | Arterial blood pH decreased |
| Investigations | Blood pH decreased | Venous blood pH decreased |
| Investigations | PCO2 abnormal | PCO2 abnormal |
| Investigations | Breath sounds abnormal | Abnormal chest sound |
| Investigations | PO2 abnormal | PO2 abnormal |
| Investigations | Breath sounds absent | Breath sounds absent |
| Investigations | Breath sounds abnormal | Breath sounds abnormal |
| Investigations | Breath sounds abnormal | Vesicular breathing abnormal |
| Investigations | Venous oxygen saturation decreased | Mixed venous blood saturation decreased |
| Investigations | Venous oxygen saturation abnormal | Mixed venous blood saturation abnormal |
| Investigations | Venous oxygen saturation decreased | SvO2 decreased |
| Investigations | Venous oxygen saturation abnormal | SvO2 abnormal |
| Investigations | Capnogram abnormal | Capnogram abnormal |
| Investigations | End-tidal CO2 abnormal | End-tidal CO2 abnormal |
| Investigations | End-tidal CO2 decreased | End-tidal CO2 decreased |
| Investigations Investigations | Alveolar oxygen partial pressure decreased | Alveolar oxygen partial pressure decreased |
| Investigations | Alveolar oxygen partial pressure abnormal | Alveolar oxygen partial pressure abnormal |
| Investigations | Venous oxygen partial pressure decreased | Venous oxygen partial pressure decreased |
| Investigations | Venous oxygen partial pressure abnormal | Venous oxygen partial pressure abnormal |
| Investigations | Venous oxygen saturation decreased | Venous oxygen saturation decreased |
| Investigations | Venous oxygen saturation abnormal | Venous oxygen saturation abnormal |
| Investigations | Oxygen saturation decreased | Arterial oxygen saturation decreased |
| Investigations | Oxygen saturation abnormal | Arterial oxygen saturation abnormal |
| | | 1 7 5 |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depression (SMQ) | | |
| Investigations | PO2 decreased | Arterial oxygen partial pressure decreased |
| Investigations | PO2 abnormal | Arterial oxygen partial pressure abnormal |
| Investigations | PO2 decreased | PaO2 decreased |
| Investigations | PO2 abnormal | PaO2 abnormal |
| Investigations | Breath sounds abnormal | Coarse breath sounds |
| Nervous system disorders | Central-alveolar hypoventilation | Central-alveolar hypoventilation |
| Nervous system disorders | Hypercapnic coma | Hypercapnic coma |
| Psychiatric disorders | Breath holding | Breath holding |
| Psychiatric disorders | Breath holding | Breath holding attack |
| Psychiatric disorders | Breath holding | Breath holding spells |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | A.R.D.S. |
| Respiratory, thoracic and mediastinal disorders | Respiratory acidosis | Acidosis respiratory |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory failure | Acute on chronic respiratory failure |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Acute respiratory distress syndrome |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory failure | Acute respiratory failure |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Adult RDS |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Adult respiratory distress syndrome |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Adult respiratory stress syndrome |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Air hunger |
| Respiratory, thoracic and mediastinal disorders | Anoxia | Anoxia |
| Respiratory, thoracic and mediastinal disorders | Apnoea | Apnea |
| Respiratory, thoracic and mediastinal disorders | Apnoea | Apnoea |
| Respiratory, thoracic and mediastinal disorders | Apnoeic attack | Apnoea attack |
| Respiratory, thoracic and mediastinal disorders | Apnoeic attack | Apnoeic attack |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | ARDS |
| | | - |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depressi | on (SMQ) | |
| Respiratory, thoracic and mediastinal disorders | Respiratory arrest | Arrest pulmonary |
| Respiratory, thoracic and mediastinal disorders | Respiratory arrest | Arrest respiratory |
| Respiratory, thoracic and mediastinal disorders | Asphyxia | Asphyxia |
| Respiratory, thoracic and mediastinal disorders | Asphyxia | Asphyxiation |
| Respiratory, thoracic and mediastinal disorders | Bradypnoea | Bradypnea |
| Respiratory, thoracic and mediastinal disorders | Bradypnoea | Bradypnoea |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Breath shortness |
| Respiratory, thoracic and mediastinal disorders | Hypopnoea | Breathing abnormally shallow |
| Respiratory, thoracic and mediastinal disorders | Respiratory arrest | Breathing arrested |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Breathing difficult |
| Respiratory, thoracic and mediastinal disorders | Hypopnoea | Breathing shallow |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Breathlessness |
| Respiratory, thoracic and mediastinal disorders | Hypercapnia | Carbon dioxide narcosis |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Central sleep apnoea syndrome |
| Respiratory, thoracic and mediastinal disorders | Cheyne-Stokes respiration | Cheyne-Stokes respiration |
| Respiratory, thoracic and mediastinal disorders | Cyanosis central | Cyanosis central |
| Respiratory, thoracic and mediastinal disorders | Respiratory depression | Depression respiratory |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Difficulty breathing |
| Respiratory, thoracic and mediastinal disorders | Respiratory distress | Distress respiratory |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Dyspnea |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Dyspnea exacerbated |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Dyspnoea |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depress | ion (SMQ) | |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Dyspnoea exacerbated |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Dyspnoea NOS |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Failure respiratory |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Gasping |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Hunger air |
| Respiratory, thoracic and mediastinal disorders | Hypercapnia | Hypercapnia |
| Respiratory, thoracic and mediastinal disorders | Hypercapnia | Hypercaphic |
| Respiratory, thoracic and mediastinal disorders | Hypercapnia | Hypercarbia |
| Respiratory, thoracic and mediastinal disorders | Hypopnoea | Hypopnea |
| Respiratory, thoracic and mediastinal disorders | Hypopnoea Hypoventilation Hypoventilation | Hypopnoea |
| Respiratory, thoracic and mediastinal disorders | Hypoventilation | Hypoventilation |
| Respiratory, thoracic and mediastinal disorders | Hypoxia | Hypoxaemia |
| Respiratory, thoracic and mediastinal disorders | Hypoxia | Hypoxemia |
| Respiratory, thoracic and mediastinal disorders | Нурохіа | Нурохіа |
| Respiratory, thoracic and mediastinal disorders | Нурохіа | Hypoxic |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Increased shortness of breath |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Increased work of breathing |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Labored breathing |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Laboured breathing |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Laboured respiration |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Marked inactivity of chest wall on inspiratory effort |
| Respiratory, thoracic and mediastinal disorders | Hypercapnia | Narcosis carbon dioxide |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depress | ion (SMQ) | |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Obstructive sleep apnoea syndrome |
| Respiratory, thoracic and mediastinal disorders | Orthopnoea | Orthopnea |
| Respiratory, thoracic and mediastinal disorders | Orthopnoea | Orthopnoea |
| Respiratory, thoracic and mediastinal disorders | Respiratory arrest | Pulmonary arrest |
| Respiratory, thoracic and mediastinal disorders | Respiratory gas exchange disorder | Resp gas exchange disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Respiration abnormal | Respiration abnormal |
| Respiratory, thoracic and mediastinal disorders | Cheyne-Stokes respiration | Respiration biot-type |
| Respiratory, thoracic and mediastinal disorders | Cheyne-Stokes respiration | Respiration Cheyne-Stokes-type |
| Respiratory, thoracic and mediastinal disorders | Respiratory depression | Respiration depressed |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Respiration failure |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiration irregularity |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Respiration labored |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Respiration labored |
| Respiratory, thoracic and mediastinal disorders | Нурорпоеа | Respiration spontaneous decreased |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiratory abnormality, unspecified |
| Respiratory, thoracic and mediastinal disorders | Respiratory acidosis | Respiratory acidosis |
| Respiratory, thoracic and mediastinal disorders | Respiratory arrest | Respiratory arrest |
| Respiratory, thoracic and mediastinal disorders | Respiratory depression | Respiratory depression |
| Respiratory, thoracic and mediastinal disorders | Respiratory depth decreased | Respiratory depth decreased |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiratory disorder |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiratory disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Respiratory distress | Respiratory distress |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depress | ion (SMQ) | |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Respiratory distress syndrome adult |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiratory dysfunction NOS |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Respiratory failure |
| Respiratory, thoracic and mediastinal disorders | Respiratory gas exchange disorder | Respiratory gas exchange disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Respiratory insufficiency |
| Respiratory, thoracic and mediastinal disorders | Respiratory paralysis | Respiratory paralysis |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiratory rhythm disorder |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Respiratory system disorder |
| Respiratory, thoracic and mediastinal disorders | Hypercapnia OT applic | Retention carbon dioxide |
| Respiratory, thoracic and mediastinal disorders | Hypopnoea | Shallow breathing |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Shock lung |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Short of breath |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Shortness of breath |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Sleep apnea |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Sleep apnea syndrome |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Sleep apnoea |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Sleep apnoea syndrome |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Sleep apnoea syndromes |
| Respiratory, thoracic and mediastinal disorders | Asphyxia | Strangulation |
| Respiratory, thoracic and mediastinal disorders | Asphyxia | Suffocation |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Surfactant deficiency syndrome adult |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Syndrome adult respiratory distress |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depression | on (SMQ) | |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory distress syndrome | Syndrome respiratory distress adult |
| Respiratory, thoracic and mediastinal disorders | Respiratory disorder | Unspecified disease of respiratory system |
| Respiratory, thoracic and mediastinal disorders | Hypoventilation | Ventilation difficult |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Ventilatory failure |
| Respiratory, thoracic and mediastinal disorders | Respiration abnormal | Respiratory sighs |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory failure | Acute respiratory decompensation |
| Respiratory, thoracic and mediastinal disorders | Respiration abnormal | Respiration abnormal NOS |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Pulmonary failure |
| Respiratory, thoracic and mediastinal disorders | Asphyxia | Injury asphyxiation |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Apnoea syndrome |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Labored respiration |
| Respiratory, thoracic and mediastinal disorders | Apnoeic attack | Apnea attack |
| Respiratory, thoracic and mediastinal disorders | Sleep apuoea syndrome | Apnea syndrome |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Central sleep apnea syndrome |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Obstructive sleep apnea syndrome |
| Respiratory, thoracic and mediastinal disorders | Orthopnoea | Supine dyspnea |
| Respiratory, thoracic and mediastinal disorders | Orthopnoea | Supine dyspnea |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Hypercapnic respiratory failure |
| Respiratory, thoracic and mediastinal disorders | Respiratory gas exchange disorder | Respiratory gas exchange disorder |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Restrictive respiratory insufficiency |
| Respiratory, thoracic and mediastinal disorders | Apnoeic attack | Apneic attack |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Acute dyspnea |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Acute central respiratory depress | sion (SMQ) | |
| Respiratory, thoracic and mediastinal disorders | Dyspnoea | Acute dyspnea |
| Respiratory, thoracic and mediastinal disorders | Cyanosis central | Cyanosis central aggravated |
| Respiratory, thoracic and mediastinal disorders | Respiratory failure | Respiratory failure aggravated |
| Respiratory, thoracic and mediastinal disorders | Acute respiratory failure | Acute respiratory insufficiency |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Hypopnea syndrome |
| Respiratory, thoracic and mediastinal disorders | Sleep apnoea syndrome | Hypopnoea syndrome |
| Respiratory, thoracic and mediastinal disorders | Hypoventilation | Alveolar hypoventilation |
| Surgical and medical procedures | Oxygen supplementation | Oxygen supplementation |

AEs Related to Route of Administration-Oral Soft Tissue Conditions (HLT) **Table 13:** 

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral So | Route of Administration : Oral Soft Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Angina bullosa haemorrhagica | Angina bullosa haemorrhagica |
| Gastrointestinal disorders | Angina bullosa haemorrhagica | Angina bullosa hemorrhagica |
| Gastrointestinal disorders | Aphthous stomatitis | Aphthous stoma |
| Gastrointestinal disorders | Aphthous stomatitis | Aphthous stomatitis |
| Gastrointestinal disorders | Aphthous stomatitis | Aphthous ulcer |
| Gastrointestinal disorders | Aphthous stomatitis | Buccal mucosa aphthous ulceration |
| Gastrointestinal disorders | Aphthous stomatitis | Canker sores oral |
| Gastrointestinal disorders | Aphthous stomatitis | Oral aphthae |
| Gastrointestinal disorders | Aphthous stomatitis | Stomatitis aphthous |
| Gastrointestinal disorders | Aphthous stomatitis | Stomatitis ulcerative aphthous |
| Gastrointestinal disorders | Aphthous stomatitis | Ulcer aphthous |
| Gastrointestinal disorders | Aphthous stomatitis | Ulcer aphthous oral |
| Gastrointestinal disorders | Aphthous stomatitis | Ulcers aphthous oral |
| Gastrointestinal disorders | Aphthous stomatitis | Canker sore lip |
| Gastrointestinal disorders | Aphthous stomatitis | Aphthous ulcer recurrent |
| Gastrointestinal disorders | Aphthous stomatitis | Aphtha |
| Gastrointestinal disorders | Buccal mucosal roughening | Roughness oral |
| Gastrointestinal disorders | Buccal mucosal roughening | Buccal mucosal roughening |
| Gastrointestinal disorders | Buccal mucosal roughening | Rough mouth |
| Gastrointestinal disorders | Burning mouth syndrome | Burning mouth syndrome |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral So | ft Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Chapped lips | Lip rough |
| Gastrointestinal disorders | Chapped lips | Chapped lips |
| Gastrointestinal disorders | Chapped lips | Cracked lips |
| Gastrointestinal disorders | Cheilitis | Angular cheilitis |
| Gastrointestinal disorders | Cheilitis | Angular stomatitis |
| Gastrointestinal disorders | Cheilitis | Cheilitis |
| Gastrointestinal disorders | Cheilitis | Lip redness |
| Gastrointestinal disorders | Cheilitis | Desquamative cheilitis |
| Gastrointestinal disorders | Cheilitis | Rash lips |
| Gastrointestinal disorders | Cheilitis | Irritation lips |
| Gastrointestinal disorders | Cheilitis | Raw lips |
| Gastrointestinal disorders | Cheilitis | Redness corner of mouth |
| Gastrointestinal disorders | Cheilitis | Inflammation lips |
| Gastrointestinal disorders | Cheilitis | Soreness corner mouth |
| Gastrointestinal disorders | Cheilitis | Sores lip |
| Gastrointestinal disorders | Cheilitis | Perleche |
| Gastrointestinal disorders | Cheilitis | Angular cheilosis |
| Gastrointestinal disorders | Cheilitis granulomatosa | Cheilitis granulomatosa |
| Gastrointestinal disorders | Cheilosis | Cheilosis |
| Gastrointestinal disorders | Contact stomatitis | Contact stomatitis |
| Gastrointestinal disorders | Enlarged uvula | Enlarged uvula |
| Gastrointestinal disorders | Gingival blister | Gingival blister |
| Gastrointestinal disorders | Gingival blister | Blisters gum |
| Gastrointestinal disorders | Gingival oedema | Gingival oedema |
| Gastrointestinal disorders | Gingival oedema | Oedema gum |
| Gastrointestinal disorders | Gingival oedema | Gingival edema |
| Gastrointestinal disorders | Gingival oedema | Edema gum |
| Gastrointestinal disorders | Gingival pruritus | Gingival pruritus |
| Gastrointestinal disorders | Gingival pruritus | Itching gum |
| Gastrointestinal disorders | Gingival swelling | Gingival swelling |
| Gastrointestinal disorders | Gingival swelling | Gum swelling |
| Gastrointestinal disorders | Hypoaesthesia oral | Anaesthesia lip |
| Gastrointestinal disorders | Hypoaesthesia oral | Anaesthesia mouth |
| Gastrointestinal disorders | Hypoaesthesia oral | Anaesthesia oral mucosa |
| Gastrointestinal disorders | Hypoaesthesia oral | Anaesthesia tongue |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoaesthesia oral NOS |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoaesthesia tongue |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness circumoral |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral So | oft Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness of mouth angular |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness of tongue |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness oral |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness perioral |
| Gastrointestinal disorders | Hypoaesthesia oral | Oral mucosal anaesthesia |
| Gastrointestinal disorders | Hypoaesthesia oral | Perioral numbness |
| Gastrointestinal disorders | Hypoaesthesia oral | Tongue sensation loss of |
| Gastrointestinal disorders | Hypoaesthesia oral | Tongue tip numbness of |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoaesthesia lips |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoaesthesia gingival |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness mouth |
| Gastrointestinal disorders | Hypoaesthesia oral | Numb mouth |
| Gastrointestinal disorders | Hypoaesthesia oral | Numb lips |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness lips |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoaesthesia gum |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness gum |
| Gastrointestinal disorders | Hypoaesthesia oral | Numbness gingival |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoesthesia gingival |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoesthesia lips |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoesthesia oral |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoesthesia tongue |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoaesthesia oral |
| Gastrointestinal disorders | Hypoaesthesia oral | Hypoesthesia gum |
| Gastrointestinal disorders | Hypoaesthesia oral | Anesthesia lip |
| Gastrointestinal disorders | Hypoaesthesia oral | Anesthesia mouth |
| Gastrointestinal disorders | Hypoaesthesia oral | Anesthesia oral mucosa |
| Gastrointestinal disorders | Hypoaesthesia oral | Anesthesia tongue |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia of mouth |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia of oral mucosa, including tongue |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia oral |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia oral NOS |
| Gastrointestinal disorders | Leukoplakia oral | Oral leukoplakia NOS |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia buccalis |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia labialis |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia lingualis |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia of oral mucosa, incl tongue |
| Gastrointestinal disorders | Leukoplakia oral | Leukoplakia tongue |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral So | ft Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Lip blister | Blister of lip |
| Gastrointestinal disorders | Lip blister | Lip blister |
| Gastrointestinal disorders | Lip blister | Blister lip |
| Gastrointestinal disorders | Lip discolouration | Lip colour altered |
| Gastrointestinal disorders | Lip discolouration | Lip discolouration |
| Gastrointestinal disorders | Lip discolouration | Lip color altered |
| Gastrointestinal disorders | Lip discolouration | Lip discoloration |
| Gastrointestinal disorders | Lip disorder | Lip disorder NOS |
| Gastrointestinal disorders | Lip disorder | Lip disorder |
| Gastrointestinal disorders | Lip disorder | Bumps lip |
| Gastrointestinal disorders | Lip erosion | Lip erosion |
| Gastrointestinal disorders | Lip exfoliation | Lip sloughing |
| Gastrointestinal disorders | Lip exfoliation | Peeling lips |
| Gastrointestinal disorders | Lip exfoliation | Lip exfoliation |
| Gastrointestinal disorders | Lip haematoma | Lip haematoma |
| Gastrointestinal disorders | Lip haematoma | Lip hematoma |
| Gastrointestinal disorders | Lip haemorrhage | Lip haemorrhage |
| Gastrointestinal disorders | Lip haemorrhage Lip haemorrhage | Hemorrhage lips |
| Gastrointestinal disorders | Lip haemorrhage | Bleeding lips |
| Gastrointestinal disorders | Lip haemorrhage | Lip hemorrhage |
| Gastrointestinal disorders | Lip haemorrhage | Haemorrhage lips |
| Gastrointestinal disorders | Lip haemorrhage | Lip bleeding |
| Gastrointestinal disorders | Lip oedema | Edema lip |
| Gastrointestinal disorders | Lip oedema | Lip edema |
| Gastrointestinal disorders | Lip oedema | Lip oedema |
| Gastrointestinal disorders | Lip oedema | Oedema lip |
| Gastrointestinal disorders | Lip pain | Lip pain |
| Gastrointestinal disorders | Lip pain | Lip sore |
| Gastrointestinal disorders | Lip pain | Lip soreness |
| Gastrointestinal disorders | Lip pain | Tender lips |
| Gastrointestinal disorders | Lip pain | Stinging lips |
| Gastrointestinal disorders | Lip pain | Sensitive lips |
| Gastrointestinal disorders | Lip pruritus | Lip pruritus |
| Gastrointestinal disorders | Lip swelling | Lip swelling |
| Gastrointestinal disorders | Lip swelling | Lips swelling non-specific |
| Gastrointestinal disorders | Lip swelling | Swelling lips |
| Gastrointestinal disorders | Lip swelling | Swelling of lips |
| Gastrointestinal disorders | Lip swelling | Swollen lips |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral So | ft Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Lip ulceration | Lip ulcer |
| Gastrointestinal disorders | Lip ulceration | Lip ulceration |
| Gastrointestinal disorders | Lip ulceration | Ulcer lip |
| Gastrointestinal disorders | Melanoplakia oral | Melanoplakia oral |
| Gastrointestinal disorders | Mouth haemorrhage | Hemorrhage mouth |
| Gastrointestinal disorders | Mouth haemorrhage | Hemorrhage mouth Hemorrhage of mouth |
| Gastrointestinal disorders | Mouth haemorrhage | Hemorrhage oral |
| Gastrointestinal disorders | Mouth haemorrhage | Mouth haemorrhage |
| Gastrointestinal disorders | Mouth haemorrhage | Mouth hemorrhage |
| Gastrointestinal disorders | Mouth haemorrhage | Oral haemorrhage |
| Gastrointestinal disorders | Mouth haemorrhage | Oral hemotrhage |
| Gastrointestinal disorders | Mouth haemorrhage | Oral mucosa bleeding |
| Gastrointestinal disorders | Mouth haemorrhage | Oral mucosa ecchymosis |
| Gastrointestinal disorders | Mouth haemorrhage | Oral mucosal petechiae |
| Gastrointestinal disorders | Mouth haemorrhage | Petechiae oral mucosa |
| Gastrointestinal disorders | Mouth haemorrhage | Bleeding mouth |
| Gastrointestinal disorders | Mouth haemorrhage | Haemorrhage mouth |
| Gastrointestinal disorders | Mouth haemorrhage | Haemorrhage of mouth |
| Gastrointestinal disorders | Mouth haemorrhage | Haemorrhage oral |
| Gastrointestinal disorders | Mouth haemorrhage | Mouth bleeding |
| Gastrointestinal disorders | Mouth ulceration | Buccal mucosa ulceration |
| Gastrointestinal disorders | Mouth ulceration | Buccal ulceration |
| Gastrointestinal disorders | Mouth ulceration | Mouth ulcer |
| Gastrointestinal disorders | Mouth ulceration | Mouth ulceration |
| Gastrointestinal disorders | Mouth ulceration | Oral ulceration |
| Gastrointestinal disorders | Mouth ulceration | Stomatitis ulcerative |
| Gastrointestinal disorders | Mouth ulceration | Ulcer buccal |
| Gastrointestinal disorders | Mouth ulceration | Ulcer mouth |
| Gastrointestinal disorders | Mouth ulceration | Ulceration mouth |
| Gastrointestinal disorders | Mouth ulceration | Ulceration of mouth |
| Gastrointestinal disorders | Mouth ulceration | Ulcerative stomatitis |
| Gastrointestinal disorders | Mouth ulceration | Ulcerative stomatitis, acute |
| Gastrointestinal disorders | Mouth ulceration | Mouth ulceration aggravated |
| Gastrointestinal disorders | Odynophagia | Odynophagia |
| Gastrointestinal disorders | Odynophagia | Swallowing painful |
| Gastrointestinal disorders | Oedema mouth | Edema of mouth |
| Gastrointestinal disorders | Oedema mouth | Oedema mouth |
| Gastrointestinal disorders | Oedema mouth | Oral mucosa swollen |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral So | ft Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Oedema mouth | Swollen mouth |
| Gastrointestinal disorders | Oedema mouth | Edema mouth |
| Gastrointestinal disorders | Oedema mouth | Oedema of mouth |
| Gastrointestinal disorders | Oral discharge | Oral discharge |
| Gastrointestinal disorders | Oral discomfort | Burning oral sensation Discomfort in mouth |
| Gastrointestinal disorders | Oral discomfort | Discomfort in mouth |
| Gastrointestinal disorders | Oral discomfort | Lip burning sensation of |
| Gastrointestinal disorders | Oral discomfort | Oral cavity discomfort |
| Gastrointestinal disorders | Oral discomfort | Oral discomfort |
| Gastrointestinal disorders | Oral discomfort | Oral hot feeling |
| Gastrointestinal disorders | Oral discomfort | Burning corner of mouth |
| Gastrointestinal disorders | Oral discomfort | Burninglips |
| Gastrointestinal disorders | Oral discomfort | Burning mouth |
| Gastrointestinal disorders | Oral disorder | Oral soft tissue disorder NOS |
| Gastrointestinal disorders | Oral disorder | Oral mucosal disorder |
| Gastrointestinal disorders | Oral disorder | Oral lesion |
| Gastrointestinal disorders | Oral disorder | Oral soft tissue disorder |
| Gastrointestinal disorders | Oral disorder Oral disorder Oral disorder Oral disorder | Oral disorder |
| Gastrointestinal disorders | Oral disorder | Mouth bump |
| Gastrointestinal disorders | Oral dysaesthesia | Dysesthesia of lips |
| Gastrointestinal disorders | Oral dysaesthesia | Dysesthesia of tongue |
| Gastrointestinal disorders | Oral dysaesthesia | Oral dysaesthesia |
| Gastrointestinal disorders | Oral dysaesthesia | Oral dysesthesia |
| Gastrointestinal disorders | Oral dysaesthesia | Dysaesthesia of lips |
| Gastrointestinal disorders | Oral dysaesthesia | Dysaesthesia of tongue |
| Gastrointestinal disorders | Oral dysaesthesia | Vincent's symptom |
| Gastrointestinal disorders | Oral leukoedema | Oral leukoedema |
| Gastrointestinal disorders | Oral lichen planus | Oral lichen planus |
| Gastrointestinal disorders | Oral mucosa atrophy | Oral mucosa atrophy |
| Gastrointestinal disorders | Oral mucosa erosion | Oral mucosa erosion |
| Gastrointestinal disorders | Oral mucosal blistering | Blistering of mouth |
| Gastrointestinal disorders | Oral mucosal blistering | Oral mucosa blister |
| Gastrointestinal disorders | Oral mucosal blistering | Oral mucosa blistering |
| Gastrointestinal disorders | Oral mucosal blistering | Oral mucosal blistering |
| Gastrointestinal disorders | Oral mucosal discolouration | Oral mucosa discolouration |
| Gastrointestinal disorders | Oral mucosal discolouration | Oral mucosal discolouration |
| Gastrointestinal disorders | Oral mucosal discolouration | Oral mucosal discoloration |
| Gastrointestinal disorders | Oral mucosal eruption | Oral mucosal eruption |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral S | oft Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Oral mucosal erythema | Oral mucosa redness |
| Gastrointestinal disorders | Oral mucosal erythema | Oral redness |
| Gastrointestinal disorders | Oral mucosal erythema | Redness mouth |
| Gastrointestinal disorders | Oral mucosal erythema | Oral mucosal erythema |
| Gastrointestinal disorders | Oral mucosal erythema | Palatal erythema |
| Gastrointestinal disorders | Oral mucosal exfoliation | Oral mucosal sloughing |
| Gastrointestinal disorders | Oral mucosal exfoliation | Sloughing of buccal mucosa |
| Gastrointestinal disorders | Oral mucosal exfoliation | Sloughing of mouth |
| Gastrointestinal disorders | Oral mucosal exfoliation | Gingival sloughing |
| Gastrointestinal disorders | Oral mucosal exfoliation | Peeling mouth |
| Gastrointestinal disorders | Oral mucosal exfoliation | Desquamation mouth |
| Gastrointestinal disorders | Oral mucosal exfoliation | Sloughing gums |
| Gastrointestinal disorders | Oral mucosal exfoliation | Sloughing gingival |
| Gastrointestinal disorders | Oral mucosal exfoliation | Peeling gingival |
| Gastrointestinal disorders | Oral mucosal exfoliation | Peeling gum |
| Gastrointestinal disorders | Oral mucosal exfoliation | Desquamation gum |
| Gastrointestinal disorders | Oral mucosal exfoliation | Desquamation gingival |
| Gastrointestinal disorders | Oral mucosal exfoliation | Oral mucosal exfoliation |
| Gastrointestinal disorders | Oral mucosal hypertrophy | Oral mucosal hypertrophy |
| Gastrointestinal disorders | Oral pain | Mouth pain |
| Gastrointestinal disorders | Oral pain | Oral angular pain |
| Gastrointestinal disorders | Oral pain | Oral mucosa pain |
| Gastrointestinal disorders | Oral pain | Oral pain |
| Gastrointestinal disorders | Oral pain | Pain mouth |
| Gastrointestinal disorders | Oral pain | Pain oral |
| Gastrointestinal disorders | Oral pain | Sore mouth |
| Gastrointestinal disorders | Oral pain | Sensitive mouth |
| Gastrointestinal disorders | Oral pain | Tender mouth |
| Gastrointestinal disorders | Oral pain | Stinging mouth |
| Gastrointestinal disorders | Oral pain | Soreness roof of mouth |
| Gastrointestinal disorders | Oral papule | Oral papule |
| Gastrointestinal disorders | Oral pruritus | Intraoral pruritus |
| Gastrointestinal disorders | Oral pruritus | Itching mouth |
| Gastrointestinal disorders | Oral pruritus | Oral pruritus |
| Gastrointestinal disorders | Oral submucosal fibrosis | Oral submucosal fibrosis |
| Gastrointestinal disorders | Oral submucosal fibrosis | Oral submucous fibrosis, including of tongue |
| Gastrointestinal disorders | Oral submucosal fibrosis | Oral submucous fibrosis, incl of tongue |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral So | ft Tissue Conditions (HLT) | |
| Gastrointestinal disorders | Oral toxicity | Oral toxicity |
| Gastrointestinal disorders | Palatal disorder | Palatal disorder |
| Gastrointestinal disorders | Palatal disorder | Palatal lesion |
| Gastrointestinal disorders | Palatal disorder | Palatal nodule |
| Gastrointestinal disorders | Palatal disorder | Soft palate disorder |
| Gastrointestinal disorders | Palatal dysplasia | Soft palate disorder Palatal dysplasia |
| Gastrointestinal disorders | Palatal oedema | Palatine arch swollen |
| Gastrointestinal disorders | Palatal oedema | Oedema uvula |
| Gastrointestinal disorders | Palatal oedema | Edema uvula |
| Gastrointestinal disorders | Palatal oedema | Palatal oedema |
| Gastrointestinal disorders | Palatal oedema | Palatal edema |
| Gastrointestinal disorders | Palatitis | Palatitis |
| Gastrointestinal disorders | Paraesthesia oral | Circumoral paresthesia |
| Gastrointestinal disorders | Paraesthesia oral | Mouth paresthesia |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia circumoral |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia mouth |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia oral NOS |
| Gastrointestinal disorders | Paraesthesia oral Paraesthesia oral Paraesthesia oral | Paraesthesia tongue |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia circumoral |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia mouth |
| Gastrointestinal disorders | Paraesthesia oral | Tongue abnormal feeling of |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia lips |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia gingival |
| Gastrointestinal disorders | Paraesthesia oral | Tingling mouth |
| Gastrointestinal disorders | Paraesthesia oral | Tingling lips |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia lips |
| Gastrointestinal disorders | Paraesthesia oral | Tingling tongue |
| Gastrointestinal disorders | Paraesthesia oral | Tingling gum |
| Gastrointestinal disorders | Paraesthesia oral | Tingling gingival |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia gum |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia gingival |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia gum |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia oral |
| Gastrointestinal disorders | Paraesthesia oral | Paresthesia tongue |
| Gastrointestinal disorders | Paraesthesia oral | Paraesthesia oral |
| Gastrointestinal disorders | Paraesthesia oral | Perioral tingling |
| Gastrointestinal disorders | Paraesthesia oral | Perioral paraesthesia |
| Gastrointestinal disorders | Paraesthesia oral | Perioral paresthesia |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration : Oral Soft Tissue Conditions (HLT) | | |
| Gastrointestinal disorders | Pigmentation buccal | Pigmentation buccal |
| Gastrointestinal disorders | Pigmentation lip | Lip pigmental spot |
| Gastrointestinal disorders | Pigmentation lip | Lip pigmentation |
| Gastrointestinal disorders | Pigmentation lip | Pigmentation lip |
| Gastrointestinal disorders | Pyostomatitis vegetans | Pyostomatitis vegetans |
| Gastrointestinal disorders | Stomatitis | Buccal inflammation |
| Gastrointestinal disorders | Stomatitis | Mouth irritation |
| Gastrointestinal disorders | Stomatitis | Mucositis oral |
| Gastrointestinal disorders | Stomatitis | Stomatitis |
| Gastrointestinal disorders | Stomatitis | Sores mouth |
| Gastrointestinal disorders | Stomatitis | Sores roof of mouth |
| Gastrointestinal disorders | Stomatitis | Raw mouth |
| Gastrointestinal disorders | Stomatitis | Irritation roof of mouth |
| Gastrointestinal disorders | Stomatitis | Chapped mouth |
| Gastrointestinal disorders | Stomatitis | Inflammation of mouth |
| Gastrointestinal disorders | Stomatitis Stomatitis Stomatitis Stomatitis Stomatitis Stomatitis | Mouth broke out |
| Gastrointestinal disorders | Stomatitis | Inflammation under tongue |
| Gastrointestinal disorders | Stomatitis | Oral mucosal irritation |
| Gastrointestinal disorders | Stomatitis | Vesicular stomatitis |
| Gastrointestinal disorders | Stomatitis | Gingivostomatitis |
| Gastrointestinal disorders | Stomatitis | Pseudomembranous stomatitis |
| Gastrointestinal disorders | Stomatitis haemorrhagic | Stomatitis haemorrhagic |
| Gastrointestinal disorders | Stomatitis haemorrhagic | Stomatitis hemorrhagic |
| Gastrointestinal disorders | Stomatitis necrotising | Cancrum oris |
| Gastrointestinal disorders | Stomatitis necrotising | Mouth necrosis |
| Gastrointestinal disorders | Stomatitis necrotising | Necrosis mouth |
| Gastrointestinal disorders | Stomatitis necrotising | Noma |
| Gastrointestinal disorders | Stomatitis necrotising | Stomatitis necrotising |
| Gastrointestinal disorders | Stomatitis necrotising | Stomatitis necrotizing |
| Gastrointestinal disorders | Uvulitis | Uvulitis |

**AEs Related to Route of Administration-Respiratory Disorders NEC (HLT)** 

| | Gastrointestinal disorders | Uvulitis | Uvulitis |
|---|---|---|---|
| | Table 14: AEs Related to | Route of Administration-Respi | ratory Disorders NEC (HLT) |
| CUR | System Organ Class | Preferred Term | Lowest Level Term |
| 800 | Route of Administration: Respiratory Disorders NEC (HLT) | | |
| This doc | Respiratory, thoracic and mediastinal disorders | Allergic cough | Allergic cough |
| | Respiratory, thoracic and mediastinal disorders | Choking | Choked on food |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respirat | tory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Choking | Choking |
| Respiratory, thoracic and mediastinal disorders | Choking | Choke on medication |
| Respiratory, thoracic and mediastinal disorders | Choking sensation | Choking sensation |
| Respiratory, thoracic and mediastinal disorders | Choking sensation | Choking sensation (excl psychogenic and dysphagia) |
| Respiratory, thoracic and mediastinal disorders | Choking sensation | Pharynx closed sensation of |
| Respiratory, thoracic and mediastinal disorders | Choking sensation | Pharynx strangled sensation of |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough increased |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough nonproductive |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough resembling asthma |
| Respiratory, thoracic and mediastinal disorders | Cough Cough Cough Cough | Coughing |
| Respiratory, thoracic and mediastinal disorders | Cough | Dry cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Irritant cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Irritative cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Nocturnal cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Persistent dry cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Persistent non-productive cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough aggravated |
| Respiratory, thoracic and mediastinal disorders | Cough | Coughing after drug inhalation |
| Respiratory, thoracic and mediastinal disorders | Cough | Drug-induced cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Smoker's cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Paroxysmal cough |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respirat | tory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Cough | Acute cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Chronic cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Persistent cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Painful cough |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough ineffective |
| Respiratory, thoracic and mediastinal disorders | Cough | Cough weak |
| Respiratory, thoracic and mediastinal disorders | Cough decreased | Cough decreased |
| Respiratory, thoracic and mediastinal disorders | Dry throat | Dry throat |
| Respiratory, thoracic and mediastinal disorders | Dry throat | Pharynx dry |
| Respiratory, thoracic and mediastinal disorders | Dry throat Dysphonia Dysphonia | Throat dry |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Distorted voice |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Disturbance in loudness |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Dysphonia |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Hoarse voice |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Hoarseness |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Hoarseness of voice |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Phonation difficulty |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Resonance disorder |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Vocal tone disorder |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Vocal volume disorder |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Voice alteration |
| Respiratory, thoracic and mediastinal disorders | Dysphonia | Voice disturbance |

| Preferred Term | Lowest Level Term |
|---|---|
| ory Disorders NEC (HLT) | |
| Dysphonia | Voice disturbance, unspecified |
| Dysphonia | Voice lowered |
| Dysphonia | Hypophonia |
| Dysphonia | Rhinolalia |
| Haemoptysis | Blood streaked sputum |
| Haemoptysis | Coughing blood |
| Haemoptysis | Haemoptysis |
| Haemoptysis | Hemoptysis |
| Haemoptysis Ot applic | Sputum bloody |
| Hiccups | Hiccough |
| Hiccups Carroll | Hiccup |
| Hiccups | Hiccups |
| Hiccups | Singultation |
| Hiccups | Singultous |
| Hiccups | Singultus |
| Hiccups | Intractable hiccups |
| Increased bronchial secretion | Airway secretion excessive |
| Increased bronchial secretion | Bronchial secretion excessive |
| Increased bronchial secretion | Bronchorrhea |
| Increased bronchial secretion | Bronchorrhoea |
| Increased bronchial secretion | Excessive bronchial secretion |
| Increased bronchial secretion | Tracheo-bronchial secretion excess |
| | Dysphonia Dysphonia Dysphonia Dysphonia Dysphonia Haemoptysis Haemoptysis Haemoptysis Haemoptysis Hiccups Hiccups Hiccups Hiccups Hiccups Hiccups Increased bronchial secretion |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respirat | ory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Increased bronchial secretion | Increased bronchial secretion |
| Respiratory, thoracic and mediastinal disorders | Increased upper airway secretion | Throat secretion increased |
| Respiratory, thoracic and mediastinal disorders | Increased upper airway secretion | Phlegm |
| Respiratory, thoracic and mediastinal disorders | Increased upper airway secretion | Increased upper airway secretion |
| Respiratory, thoracic and mediastinal disorders | Increased viscosity of bronchial secretion | Sputum viscosity increased |
| Respiratory, thoracic and mediastinal disorders | Increased viscosity of bronchial secretion | Increased viscosity of bronchial secretion |
| Respiratory, thoracic and mediastinal disorders | Increased viscosity of nasal secretion | Increased viscosity of nasal secretion |
| Respiratory, thoracic and mediastinal disorders | Increased viscosity of nasal secretion | Thick nasal mucus |
| Respiratory, thoracic and mediastinal disorders | Laryngeal discomfort | Laryngeal discomfort |
| Respiratory, thoracic and mediastinal disorders | Laryngeal discomfort | Pharyngolaryngeal discomfort |
| Respiratory, thoracic and mediastinal disorders | Laryngeal pain | Laryngeal pain |
| Respiratory, thoracic and mediastinal disorders | Laryngeal pain | Larynx burning pain of |
| Respiratory, thoracic and mediastinal disorders | Laryngeal pain | Larynx pain |
| Respiratory, thoracic and mediastinal disorders | Laryngeal pain | Pharyngolaryngeal pain |
| Respiratory, thoracic and mediastinal disorders | Mouth breathing | Jaw breathing |
| Respiratory, thoracic and mediastinal disorders | Mouth breathing | Mouth breathing |
| Respiratory, thoracic and mediastinal disorders | Nasal discharge discolouration | Nasal discharge discolouration |
| Respiratory, thoracic and mediastinal disorders | Nasal discharge discolouration | Nasal discharge discoloration |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Discomfort in nose |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal burning |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal cavity strange sensation of |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal irritation |
| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respirat | tory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal itching |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal passage irritation |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal soreness |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Sore nose |
| Respiratory, thoracic and mediastinal disorders | Nasal discomfort | Nasal discomfort |
| Respiratory, thoracic and mediastinal disorders | Nasal flaring | Nasal flaring |
| Respiratory, thoracic and mediastinal disorders | Nasal obstruction | Nasal obstruction |
| Respiratory, thoracic and mediastinal disorders | Nasal obstruction | Nasal obstruction increased |
| Respiratory, thoracic and mediastinal disorders | Nasopharyngeal reflux | Nasopharyngeal reflux |
| Respiratory, thoracic and mediastinal disorders | Nocturnal dyspnoea | Nocturnal dyspnoea |
| Respiratory, thoracic and mediastinal disorders | Nocturnal dysphoea | Nocturnal dyspnea |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal blistering | Oropharyngeal blistering |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal discomfort | Pharynx discomfort |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal discomfort | Pharynx ill sensation of |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal discomfort | Pharynx strange sensation of |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal discomfort | Oropharyngeal discomfort |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Pain pharynx |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Pain throat |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Sore throat |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Sore throat NOS |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Throat pain |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal pain | Throat sore |

| Oropharyngeal pain Oropharyngeal pain Oropharyngeal pain | Chronic sore throat Oropharyngeal pain |
|---|---|
| Oropharyngeal pain | |
| | Oropharyngeal pain |
| Oropharyngeal plaque | |
| | Mouth plaque |
| Oropharyngeal plaque | Plaque mouth |
| Oropharyngeal plaque | Oropharyngeal plaque |
| Oropharyngeal scar | Oropharyngeal scar |
| Paranasal sinus discomfort | Paranasal sinus discomfort |
| Productive cough | Productive cough |
| Productive cough | Sputum |
| Productive cough | Expectoration |
| Respiratory tract oedema | Respiratory tract oedema |
| Respiratory tract oedema | Airway oedema |
| Respiratory tract oedema | Airway edema |
| Respiratory tract oedema | Respiratory tract edema |
| Rhinalgia | Nasal stinging |
| Rhinalgia | Stinging of nose |
| Rhinalgia | Rhinalgia |
| Rhinalgia | Nasal pain |
| Rhinorrhoea | Nasal discharge |
| Rhinorrhoea | Nasal discharge watery excessive |
| Rhinorrhoea | Rhinorrhea |
| Rhinorrhoea | Rhinorrhoea |
| | Oropharyngeal plaque Oropharyngeal scar Paranasal sinus discomfort Productive cough Productive cough Productive cough Respiratory tract oedema Respiratory tract oedema Respiratory tract oedema Respiratory tract oedema Rhinalgia Rhinalgia Rhinalgia Rhinorrhoea Rhinorrhoea Rhinorrhoea |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respira | tory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Runny nose |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Nasal mucus increased |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Mucus nasal increased |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Gustatory rhinorrhoea |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Sniffles |
| Respiratory, thoracic and mediastinal disorders | Rhinorrhoea | Gustatory rhinorthea |
| Respiratory, thoracic and mediastinal disorders | Sneezing | Paroxysmal sneeze |
| Respiratory, thoracic and mediastinal disorders | Sneezing | Sneezing |
| Respiratory, thoracic and mediastinal disorders | Sneezing | Sneezing excessive |
| Respiratory, thoracic and mediastinal disorders | Snoring Snoring Snoring | Snore |
| Respiratory, thoracic and mediastinal disorders | Snoring | Snoring |
| Respiratory, thoracic and mediastinal disorders | Sputum decreased | Sputum decreased |
| Respiratory, thoracic and mediastinal disorders | Sputum discoloured | Sputum discolored |
| Respiratory, thoracic and mediastinal disorders | Sputum discoloured | Sputum discoloured |
| Respiratory, thoracic and mediastinal disorders | Sputum increased | Sputum excretion increased |
| Respiratory, thoracic and mediastinal disorders | Sputum increased | Sputum increased |
| Respiratory, thoracic and mediastinal disorders | Sputum retention | Sputum excretion difficulty |
| Respiratory, thoracic and mediastinal disorders | Sputum retention | Sputum expectoration difficult |
| Respiratory, thoracic and mediastinal disorders | Sputum retention | Sputum sticking sensation of |
| Respiratory, thoracic and mediastinal disorders | Sputum retention | Sputum retention |
| Respiratory, thoracic and mediastinal disorders | Suffocation feeling | Suffocation feeling |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Burning in throat |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respirat | tory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Local throat irritation |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Pharyngo-oral irritation |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Pharynx burning sensation of |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Pharynx irritated sensation of |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Pharynx itchy sensation of |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Throat burning sensation of |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Throat irritation |
| Respiratory, thoracic and mediastinal disorders | Throat irritation | Itehy throat |
| Respiratory, thoracic and mediastinal disorders | Throat lesion | Throat lesion |
| Respiratory, thoracic and mediastinal disorders | Throat tightness | Constriction throat |
| Respiratory, thoracic and mediastinal disorders | Throat tightness | Throat constriction |
| Respiratory, thoracic and mediastinal disorders | Throat tightness | Throat tightness |
| Respiratory, thoracic and mediastinal disorders | Upper anway necrosis | Upper airway necrosis |
| Respiratory, thoracic and mediastinal disorders | Upper airway obstruction | Upper airway obstruction |
| Respiratory, thoracic and mediastinal disorders | Upper airway resistance syndrome | Upper airway resistance syndrome |
| Respiratory, thoracic and mediastinal disorders | Upper respiratory tract congestion | Upper respiratory tract congestion |
| Respiratory, thoracic and mediastinal disorders | Upper respiratory tract inflammation | Upper respiratory tract inflammation |
| Respiratory, thoracic and mediastinal disorders | Upper respiratory tract inflammation | Acute upper respiratory tract inflammation |
| Respiratory, thoracic and mediastinal disorders | Upper respiratory tract irritation | Upper respiratory tract irritation |
| Respiratory, thoracic and mediastinal disorders | Upper-airway cough syndrome | Posterior nasal drip |
| Respiratory, thoracic and mediastinal disorders | Upper-airway cough syndrome | Postnasal drip |
| Respiratory, thoracic and mediastinal disorders | Upper-airway cough syndrome | Chronic post nasal drip |

Statistical Analysis Plan for Protocol No.: P261-401

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Respir | Route of Administration: Respiratory Disorders NEC (HLT) | |
| Respiratory, thoracic and mediastinal disorders | Upper-airway cough syndrome | Upper-airway cough syndrome |
| Respiratory, thoracic and mediastinal disorders | Yawning | Yawn |
| Respiratory, thoracic and mediastinal disorders | Yawning | Yawning |
| Respiratory, thoracic and mediastinal disorders | Yawning | Yawning excessive |

Table 15: AEs Related to Route of Administration-Upper Respiratory Tract Disorders (HLT) (Exclude Infections)

System Organ Class

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | r Respiratory Tract Disorders (HLT) ( | Exclude Infections) |
| Respiratory, thoracic and mediastinal disorders | Adductor vocal cord weakness | Adductor vocal cord weakness |
| Respiratory, thoracic and mediastinal disorders | Adenoidal disorder | Adenoidal disorder |
| Respiratory, thoracic and mediastinal disorders | Adenoidal hypertrophy | Adenoid vegetations |
| Respiratory, thoracic and mediastinal disorders | Adenoidal hypertrophy | Adenoidal hypertrophy |
| Respiratory, thoracic and mediastinal disorders | Allergic pharyngitis | Allergic pharyngitis |
| Respiratory, thoracic and mediastinal disorders | Allergic sinusitis | Allergic sinusitis |
| Respiratory, thoracic and mediastinal disorders | Allergic sinusitis | Seasonal sinusitis |
| Respiratory, thoracic and mediastinal disorders | Chronic eosinophilic rhinosinusitis | Chronic eosinophilic rhinosinusitis |
| Respiratory, thoracic and mediastinal disorders | Chronic hyperplastic eosinophilic sinusitis | Chronic hyperplastic eosinophilic sinusitis |
| Respiratory, thoracic and mediastinal disorders | Croup noninfectious | Croup noninfectious |
| Respiratory, thoracic and mediastinal disorders | Dysaesthesia pharynx | Dysaesthesia pharynx |
| Respiratory, thoracic and mediastinal disorders | Dysaesthesia pharynx | Dysesthesia pharynx |
| Respiratory, thoracic and mediastinal disorders | Dysaesthesia pharynx | Laryngopharyngeal dysesthesia |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT) | (Exclude Infections) |
| Respiratory, thoracic and mediastinal disorders | Dysaesthesia pharynx | Laryngopharyngeal dysaesthesia |
| Respiratory, thoracic and mediastinal disorders | Eosinophilic rhinitis | Eosinophilic rhinitis |
| Respiratory, thoracic and mediastinal disorders | Epiglottic cyst | Epiglottic cyst |
| Respiratory, thoracic and mediastinal disorders | Epiglottic erythema | Epiglottic erythema |
| Respiratory, thoracic and mediastinal disorders | Epiglottic mass | Epiglottic mass |
| Respiratory, thoracic and mediastinal disorders | Epiglottic oedema | Epiglottic oedema |
| Respiratory, thoracic and mediastinal disorders | Epiglottic oedema | Epiglottic edema |
| Respiratory, thoracic and mediastinal disorders | Epiglottis ulcer | Epiglottis ulcer |
| Respiratory, thoracic and mediastinal disorders | Epistaxis Epistaxis | Bleeding nose |
| Respiratory, thoracic and mediastinal disorders | Epistaxis Epistaxis | Epistaxis |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Haemorrhage nasal |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Hemorrhage nasal |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Nasal bleeding |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Nasal mucus blood tinged |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Nose bleed |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Nose bleeds |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Nosebleed |
| Respiratory, thoracic and mediastinal disorders | Epistaxis | Chronic epistaxis |
| Respiratory, thoracic and mediastinal disorders | Intranasal hypoaesthesia | Intranasal numbness |
| Respiratory, thoracic and mediastinal disorders | Intranasal hypoaesthesia | Intranasal hypoaesthesia |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT) | (Exclude Infections) |
| Respiratory, thoracic and mediastinal disorders | Intranasal hypoaesthesia | Intranasal hypoesthesia |
| Respiratory, thoracic and mediastinal disorders | Intranasal paraesthesia | Intranasal paraesthesia |
| Respiratory, thoracic and mediastinal disorders | Intranasal paraesthesia | Intranasal paresthesia |
| Respiratory, thoracic and mediastinal disorders | Laryngeal cyst | Laryngeal cyst |
| Respiratory, thoracic and mediastinal disorders | Laryngeal disorder | Laryngeal disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Laryngeal disorder | Unspecified disease of larynx |
| Respiratory, thoracic and mediastinal disorders | Laryngeal disorder | Laryngeal disorder |
| Respiratory, thoracic and mediastinal disorders | Laryngeal dyspnoea | Laryngeal dyspnoea |
| Respiratory, thoracic and mediastinal disorders | Laryngeal dyspnoea | Laryngeal dyspnea |
| Respiratory, thoracic and mediastinal disorders | Laryngeal erythema | Laryngeal erythema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haematoma | Laryngeal haematoma |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haematoma | Laryngeal hematoma |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haematoma | Glottic haematoma |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haematoma | Glottic hematoma |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haemorrhage | Laryngeal haemorrhage |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haemorrhage | Laryngeal hemorrhage |
| Respiratory, thoracic and mediastinal disorders | Laryngeal haemorrhage | Laryngeal bleeding |
| Respiratory, thoracic and mediastinal disorders | Laryngeal hypertrophy | Laryngeal hypertrophy |
| Respiratory, thoracic and mediastinal disorders | Laryngeal infiltration | Laryngeal infiltration NOS |
| Respiratory, thoracic and mediastinal disorders | Laryngeal infiltration | Laryngeal infiltration |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT | ) (Exclude Infections) |
| Respiratory, thoracic and mediastinal disorders | Laryngeal inflammation | Laryngeal inflammation |
| Respiratory, thoracic and mediastinal disorders | Laryngeal inflammation | Laryngeal mucositis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal leukoplakia | Laryngeal leukoplakia |
| Respiratory, thoracic and mediastinal disorders | Laryngeal leukoplakia | Laryngeal leucoplakia |
| Respiratory, thoracic and mediastinal disorders | Laryngeal mass | Laryngeal mass |
| Respiratory, thoracic and mediastinal disorders | Laryngeal necrosis | Laryngeal necrosis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal necrosis | Laryngeal chondronecrosis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal obstruction | Laryngeal obstruction |
| Respiratory, thoracic and mediastinal disorders | Laryngeal obstruction | Subglottic obstruction |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedeina | Edema glottis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Edema larynx |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Edema of larynx |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Edema vocal cord |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Glottic edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Glottic oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Laryngeal edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Laryngeal oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Larynx edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Larynx oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Oedema of larynx |
| | • | • |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Uppe | r Respiratory Tract Disorders (HL | T) (Exclude Infections) |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Subglottic edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Subglottic oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Vocal cord edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Vocal cord oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Oedema glottis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Oedema larynx |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Oedema vocal cord |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Aryepiglottis edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema Laryngeal oedema | Aryepiglottis oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Acute laryngeal edema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal oedema | Acute laryngeal oedema |
| Respiratory, thoracic and mediastinal disorders | Laryngeal polyp | Laryngeal polyp |
| Respiratory, thoracic and mediastinal disorders | Laryngeal stenosis | Laryngeal stenosis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal stenosis | Laryngeal stricture |
| Respiratory, thoracic and mediastinal disorders | Laryngeal stenosis | Stenosis of larynx |
| Respiratory, thoracic and mediastinal disorders | Laryngeal stenosis | Subglottic stenosis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal stenosis | Supraglottic stenosis |
| Respiratory, thoracic and mediastinal disorders | Laryngeal ulceration | Laryngeal ulceration |
| Respiratory, thoracic and mediastinal disorders | Laryngeal ulceration | Larynx ulcer |
| Respiratory, thoracic and mediastinal disorders | Laryngeal ulceration | Larynx ulceration |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT | (F) (Exclude Infections) |
| Respiratory, thoracic and mediastinal disorders | Laryngeal ventricle prolapse | Laryngeal ventricle prolapse |
| Respiratory, thoracic and mediastinal disorders | Laryngitis allergic | Laryngitis allergic |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm | Glottic spasm |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm | Laryngeal spasm |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm | Laryngismus |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm | Laryngospasm |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm | Larynx muscle hypersensitive |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm | Spasm glottis |
| Respiratory, thoracic and mediastinal disorders | Laryngospasm Larynx irritation | Spasm larynx |
| Respiratory, thoracic and mediastinal disorders | Larynx irritation | Larynx irritation |
| Respiratory, thoracic and mediastinal disorders | Larynx irritation | Larynx itching |
| Respiratory, thoracic and mediastinal disorders | Maxillary sinus pseudocyst | Maxillary sinus pseudocyst |
| Respiratory, thoracic and mediastinal disorders | Nasal cavity mass | Nasal cavity mass |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Congestion nasal |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Nasal congestion |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Nasal stuffiness |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Nose congestion |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Rhinitis medicamentosa |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Rhinitis medicamentous |
| Respiratory, thoracic and mediastinal disorders | Nasal congestion | Nasal mucosal swelling |

| gestion |
|--------------|
| estion |
| Valial |
| ORSON |
| OS S |
| of |
| on |
| mmation |
| flammation |
| ophy |
| scolouration |
| scoloration |
| llor |
| sorder NOS |
| sorder |
| ythema |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT | (Exclude Infections) |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal disorder | Nasal mucosal hyperaemia |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal disorder | Nasal mucosal ulcer |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal disorder | Nasal mucosal hyperemia |
| Respiratory, thoracic and mediastinal disorders | Nasal mucosal hypertrophy | Nasal mucosal hypertrophy |
| Respiratory, thoracic and mediastinal disorders | Nasal necrosis | Nasal mucosal necrosis |
| Respiratory, thoracic and mediastinal disorders | Nasal necrosis | Nasal necrosis |
| Respiratory, thoracic and mediastinal disorders | Nasal necrosis | Necrosis nasal |
| Respiratory, thoracic and mediastinal disorders | Nasal necrosis | Nasal septal mucosa necrosis |
| Respiratory, thoracic and mediastinal disorders | Nasal odour OR | Nasal odour |
| Respiratory, thoracic and mediastinal disorders | Nasal odour | Nasal odor |
| Respiratory, thoracic and mediastinal disorders | Nasal oedema | Nasal oedema |
| Respiratory, thoracic and mediastinal disorders | Nasal oedema | Nose edema |
| Respiratory, thoracic and mediastinal disorders | Nasal oedema | Nose oedema |
| Respiratory, thoracic and mediastinal disorders | Nasal oedema | Nasal turbinate edema |
| Respiratory, thoracic and mediastinal disorders | Nasal oedema | Nasal edema |
| Respiratory, thoracic and mediastinal disorders | Nasal oedema | Nasal turbinate oedema |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Nasal polyp |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Nasal polyps |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Polyp of nasal cavity |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Polyps nasal |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT | (Exclude Infections) |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Unspecified nasal polyp |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Hyperplastic nasal polyp |
| Respiratory, thoracic and mediastinal disorders | Nasal polyps | Choanal polyp |
| Respiratory, thoracic and mediastinal disorders | Nasal septum disorder | Nasal septum disorder |
| Respiratory, thoracic and mediastinal disorders | Nasal septum disorder | Nasal septum disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Nasal septum disorder | Nasal septal erythema |
| Respiratory, thoracic and mediastinal disorders | Nasal septum perforation | Nasal septum perforation |
| Respiratory, thoracic and mediastinal disorders | Nasal septum perforation | Perforation nasal septum |
| Respiratory, thoracic and mediastinal disorders | Nasal septum ulceration | Nasal septum ulceration |
| Respiratory, thoracic and mediastinal disorders | Nasal turbinate abnormality | Nasal turbinate abnormality |
| Respiratory, thoracic and mediastinal disorders | Nasal turbinate hypertrophy | Hypertrophy of nasal turbinates |
| Respiratory, thoracic and mediastinal disorders | Nasal turbinate hypertrophy | Nasal turbinate hypertrophy |
| Respiratory, thoracic and mediastinal disorders | Nasal turbinate hypertrophy | Concha bullosa |
| Respiratory, thoracic and mediastinal disorders | Nasal ulcer | Nasal ulcer |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal spasm | Oropharyngeal spasm |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal spasm | Spasm oropharyngeal |
| Respiratory, thoracic and mediastinal disorders | Oropharyngeal swelling | Oropharyngeal swelling |
| Respiratory, thoracic and mediastinal disorders | Paranasal cyst | Paranasal sinus mucocoele |
| Respiratory, thoracic and mediastinal disorders | Paranasal cyst | Paranasal cyst |
| Respiratory, thoracic and mediastinal disorders | Paranasal cyst | Paranasal sinus mucocele |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Uppe | r Respiratory Tract Disorders (HLT) | (Exclude Infections) |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus haematoma | Maxillary sinus haematoma |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus haematoma | Maxillary sinus hematoma |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus haematoma | Paranasal sinus haematoma |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus haematoma | Paranasal sinus hematoma |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus hypersecretion | Paranasal sinus hypersecretion |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus hypersecretion | Nasal sinus discharge |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus mucosal hypertrophy | Paranasal sinus mucosal hypertrophy |
| Respiratory, thoracic and mediastinal disorders | Paranasal sinus necrosis | Paranasal sinus necrosis |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal cyst | Pharyngeal cyst |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal disorder | Pharyngeal disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal disorder | Unspecified disease of pharynx |
| Respiratory, thoracic and mediastinal disorders | Pharyngcal disorder | Nasopharyngeal disorder |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal disorder | Pharyngeal disorder |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal dyskinesia | Pharyngeal dyskinesia |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal enanthema | Pharyngeal enanthema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal erosion | Pharyngeal erosion |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal erythema | Pharynx redness of |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal erythema | Red throat |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal erythema | Pharyngeal erythema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal erythema | Uvular erythema |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper Respiratory Tract Disorders (HLT) (Exclude Infections) | | |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal exudate | Pharyngeal exudate |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal fistula | Pharyngeal fistula |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haematoma | Pharyngeal haematoma |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haematoma | Pharyngeal hematoma |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Haemorrhage from throat |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Haemorrhage pharyngeal |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Hemorrhage from throat |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Pharyngeal haemorrhage |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Hemorrhage pharyngeal |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Pharyngeal hemorrhage |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Oropharyngeal hemorrhage |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal haemorrhage | Oropharyngeal haemorrhage |
| Respiratory, thoracic and mediastinal disorders | Rharyngeal haemorrhage | Pharyngeal bleeding |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal hypertrophy | Pharyngeal hypertrophy |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal hypoaesthesia | Pharyngeal hypoaesthesia |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal hypoaesthesia | Numbness throat |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal hypoaesthesia | Pharyngeal hypoesthesia |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal inflammation | Pharyngeal inflammation |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal inflammation | Pharyngeal mucositis |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal lesion | Pharyngeal lesion |

| System Organ Class Preferred Term | | Lowest Level Term |
|---|---|---|
| Route of Administration: Uppe | er Respiratory Tract Disorders (HLT | Γ) (Exclude Infections) |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal leukoplakia | Pharyngeal leukoplakia |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal mass | Pharyngeal mass |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal mucosa atrophy | Pharyngeal mucosa atrophy |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal necrosis | Pharyngeal necrosis |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Edema pharynx |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Oedema pharynx |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Pharyngeal oedema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Pharynx edema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Throat edema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Throat oedema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oederna | Throat swelling |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Throat swelling non-specific |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Throat swelling NOS |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Pharyngeal edema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal oedema | Pharynx oedema |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal polyp | Pharyngeal polyp |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal stenosis | Pharyngeal stenosis |
| Respiratory, thoracic and mediastinal disorders | Pharyngeal ulceration | Pharyngeal ulceration |
| Respiratory, thoracic and mediastinal disorders | Reflux laryngitis | Laryngopharyngeal reflux |
| Respiratory, thoracic and mediastinal disorders | Reflux laryngitis | Reflux laryngitis |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper | Respiratory Tract Disorders (HLT) | (Exclude Infections) |
| Respiratory, thoracic and mediastinal disorders | Rhinitis allergic | Allergic rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis allergic | Allergic rhinitis (excl hay fever) |
| Respiratory, thoracic and mediastinal disorders | Rhinitis allergic | Atopic rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis allergic | Rhinitis allergic |
| Respiratory, thoracic and mediastinal disorders | Rhinitis allergic | Rhinitis allergic atopic |
| Respiratory, thoracic and mediastinal disorders | Rhinitis allergic | Rhinitis allergic NOS |
| Respiratory, thoracic and mediastinal disorders | Rhinitis atrophic | Atrophic rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis atrophic | Ozena |
| Respiratory, thoracic and mediastinal disorders | Rhinitis atrophic | Rhinitis atrophic |
| Respiratory, thoracic and mediastinal disorders | Rhinitis atrophic | Dry rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis hypertrophic | Rhinitis hypertrophic |
| Respiratory, thoracic and mediastinal disorders | Rhinitis perennial | Perennial allergic rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis perennial | Perennial rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis perennial | Rhinitis perennial |
| Respiratory, thoracic and mediastinal disorders | Rhinitis seasonal | Allergic rhinitis due to pollen |
| Respiratory, thoracic and mediastinal disorders | Rhinitis seasonal | Rhinitis seasonal |
| Respiratory, thoracic and mediastinal disorders | Rhinitis seasonal | Seasonal allergic rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis seasonal | Seasonal rhinitis |
| Respiratory, thoracic and mediastinal disorders | Rhinitis ulcerative | Rhinitis ulcerative |
| Respiratory, thoracic and mediastinal disorders | Rhinolithiasis | Rhinolithiasis |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper Respiratory Tract Disorders (HLT) (Exclude Infections) | | |
| Respiratory, thoracic and mediastinal disorders | Rhinolithiasis | Nasal calculus |
| Respiratory, thoracic and mediastinal disorders | Sinus congestion | Nasal sinus congestion |
| Respiratory, thoracic and mediastinal disorders | Sinus congestion | Sinus congestion |
| Respiratory, thoracic and mediastinal disorders | Sinus disorder | Sinus disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Sinus disorder | Sinus disorder |
| Respiratory, thoracic and mediastinal disorders | Sinus perforation | Perforation of sinus |
| Respiratory, thoracic and mediastinal disorders | Sinus perforation | Sinus perforation |
| Respiratory, thoracic and mediastinal disorders | Sinus polyp | Antral polyp (of maxillary sinus) |
| Respiratory, thoracic and mediastinal disorders | Sinus polyp | Maxillary sinus polyp |
| Respiratory, thoracic and mediastinal disorders | Sinus polyp | Sinus polyp |
| Respiratory, thoracic and mediastinal disorders | Sinus polyp degeneration | Polypoid sinus degeneration |
| Respiratory, thoracic and mediastinal disorders | Sinus polyp degeneration | Sinus polyp degeneration |
| Respiratory, thoracic and mediastinal disorders | Sinusitis noninfective | Sinusitis noninfective |
| Respiratory, thoracic and mediastinal disorders | Stridor | Stridor |
| Respiratory, thoracic and mediastinal disorders | Stridor | Stridor inspiratory |
| Respiratory, thoracic and mediastinal disorders | Tonsillar atrophy | Tonsillar atrophy |
| Respiratory, thoracic and mediastinal disorders | Tonsillar atrophy | Submerged tonsil |
| Respiratory, thoracic and mediastinal disorders | Tonsillar disorder | Chronic tonsillar disease |
| Respiratory, thoracic and mediastinal disorders | Tonsillar disorder | Tonsillar disorder |
| Respiratory, thoracic and mediastinal disorders | Tonsillar disorder | Cryptic tonsil |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper Respiratory Tract Disorders (HLT) (Exclude Infections) | | |
| Respiratory, thoracic and mediastinal disorders | Tonsillar haemorrhage | Tonsillar haemorrhage |
| Respiratory, thoracic and mediastinal disorders | Tonsillar haemorrhage | Tonsillar hemorrhage |
| Respiratory, thoracic and mediastinal disorders | Tonsillar haemorrhage | Tonsillar bleeding |
| Respiratory, thoracic and mediastinal disorders | Tonsillar hypertrophy | Tonsillar hypertrophy |
| Respiratory, thoracic and mediastinal disorders | Tonsillar hypertrophy | Enlarged tonsils |
| Respiratory, thoracic and mediastinal disorders | Tonsillar inflammation | Tonsillar inflammation |
| Respiratory, thoracic and mediastinal disorders | Tonsillar ulcer | Tonsillar ulcer |
| Respiratory, thoracic and mediastinal disorders | Tonsillolith | Tonsillolith |
| Respiratory, thoracic and mediastinal disorders | Vasomotor rhinitis | Vasomotor rhinitis |
| Respiratory, thoracic and mediastinal disorders | Velopharyngeal incompetence | Velopharyngeal incompetence |
| Respiratory, thoracic and mediastinal disorders | Vocal cord atrophy | Vocal cord atrophy |
| Respiratory, thoracic and mediastinal disorders | Vocal cord cyst | Vocal cord cyst |
| Respiratory, thoracic and mediastinal disorders | Vocal cord disorder | Vocal cord disorder NOS |
| Respiratory, thoracic and mediastinal disorders | Vocal cord disorder | Vocal cord dysfunction |
| Respiratory, thoracic and mediastinal disorders | Vocal cord disorder | Vocal cord disorder |
| Respiratory, thoracic and mediastinal disorders | Vocal cord inflammation | Vocal cord inflammation |
| Respiratory, thoracic and mediastinal disorders | Vocal cord leukoplakia | Vocal cord leukoplakia |
| Respiratory, thoracic and mediastinal disorders | Vocal cord polyp | Polyp of vocal cord |
| Respiratory, thoracic and mediastinal disorders | Vocal cord polyp | Vocal cord polyp |
| Respiratory, thoracic and mediastinal disorders | Vocal cord thickening | Singers nodules |

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Route of Administration: Upper Respiratory Tract Disorders (HLT) (Exclude Infections) | | |
| Respiratory, thoracic and mediastinal disorders | Vocal cord thickening | Vocal cord thickening |
| Respiratory, thoracic and mediastinal disorders | Vocal cord thickening | Vocal cord nodule |

Table 16: AEs Related to Taste and Smell Disorders (SMQ)

| System Organ Class | Preferred Term | Lowest Level Term |
|---|---|---|
| Taste and Smell Disorders (SMQ) | ) | ans. |
| Nervous system disorders | Dysgeusia | After taste |
| Nervous system disorders | Ageusia | Ageusia |
| Nervous system disorders | Parosmia | Altered smell sensation |
| Nervous system disorders | Anosmia | Anosmia |
| Nervous system disorders | Dysgeusia | Dysgeusia |
| Nervous system disorders | Parosmia | Dysosmia |
| Nervous system disorders | Parosmia Parosmia | Dysosmia NOS |
| Nervous system disorders | Parosmia Parosmia Hypogeusia Hellveingtion gustory | Faint odor of sulfur |
| Nervous system disorders | Hypogeusia | Gustatory sense diminished |
| Psychiatric disorders | Hallucination, gustatory | Hallucination gustatory |
| Psychiatric disorders | Hallucination, olfactory | Hallucination olfactory |
| Psychiatric disorders | Hallucination, gustatory | Hallucination, gustatory |
| Psychiatric disorders | Hallucination, olfactory | Hallucination, olfactory |
| Nervous system disorders | Parosmia | Hyperosmia |
| Nervous system disorders | Hypogeusia | Hypogeusia |
| Nervous system disorders | Anosmia | Loss of smell |
| Nervous system disorders | Ageusia | Loss of taste |
| Psychiatric disorders | Hallucination, olfactory | Olfactory hallucination |
| Nervous system disorders | Dysgeusia | Parageusia |
| Nervous system disorders | Parosmia | Parosmia |
| Nervous system disorders | Parosmia | Perversion olfactory |
| Nervous system disorders | Parosmia | Smell alteration |
| Nervous system disorders | Parosmia | Smell change |
| Nervous system disorders | Anosmia | Smell loss |
| Nervous system disorders | Parosmia | Smell perversion |
| Nervous system disorders | Parosmia | Smelly sensation |
| Nervous system disorders | Parosmia | Strange smell sensation |
| Nervous system disorders | Dysgeusia | Taste abnormality |
| Nervous system disorders | Ageusia Taste absent | |

| System Organ Class Preferred Term | | Lowest Level Term |
|---|---|---|
| Taste and Smell Disorders (SMQ) | | |
| Nervous system disorders | Dysgeusia | Taste alteration |
| Nervous system disorders | Dysgeusia | Taste altered |
| Nervous system disorders | Dysgeusia | Taste bitter |
| Nervous system disorders | Dysgeusia | Taste bitter-salty |
| Nervous system disorders | Dysgeusia | Taste changed |
| Nervous system disorders | Hypogeusia | Taste diminished |
| Nervous system disorders | Dysgeusia | |
| Nervous system disorders | Dysgeusia | Taste disturbance Taste garlic |
| Nervous system disorders | Ageusia | Taste loss |
| Nervous system disorders | Dysgeusia | Taste metallice |
| Nervous system disorders | Dysgeusia | Taste peculiar |
| Nervous system disorders | Dysgeusia | Taste perversion |
| Nervous system disorders | Dysgeusia | Taste salty |
| Nervous system disorders | Dysgeusia | Taste sour |
| Nervous system disorders | Dysgeusia | Taste sweet |
| Nervous system disorders | Dysgeusia | Bilious taste |
| Nervous system disorders | Parosmia | Cacosmia |
| Nervous system disorders | Hyposmia | Hyposmia |
| Nervous system disorders | Dysgeusia Parosmia Hyposmia Parosmia Olfactory part disorder | Faint odour of sulfur |
| Nervous system disorders | Olfactory nerve disorder | Olfactory nerve disorder |
| Investigations | Olfactory test abnormal | Olfactory test abnormal |
| Investigations | Olfactory test abnormal | Olfactory acuity test abnormal |
| Nervous system disorders | Hyposmia | Diminished sense of smell |
| Investigations | Gustometry abnormal | Gustometry abnormal |
| General disorders and administration site conditions Nervous system disorders | Product taste abnormal | Medication after taste |
| Nervous system disorders | Parosmia Phantosmia | |
| Nervous system disorders | Parosmia Olfactism | |
| Nervous system disorders | Hypergeusia Hypergeusia | |
| Nervous system disorders | Dysgeusia Chalky taste | |

AEs Related to Depression and Suicidality/Self-Injury-Depression (SMQ) (Exclude Suicide/Self-Injury)

| | ivervous system disorders | Trypergeusia | | Trypergeusia |
|---|---|---|---|---|
| | Nervous system disorders | Dysgeusia | | Chalky taste |
| Table 17: AEs Related to Depression and Suicidality/Self-Injury-Depr | | | -Injury-Depression (SMQ) | |
| | (Exclude Suicide/Self-Injury) | | | |
| *OC/1/ | Preferred Term Depression and Suicide/Self-Injury: Depression (SMQ) (Exclude Suicide/Self-Injury) Activation syndrome | | | rm |
| is | | | | e/Self-Injury) |
| KI. | Activation syndrome | | | me |
| Adjustment disorder with depressed mood | | | Adjustment disorder with depressed mood | |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SMC | Q) (Exclude Suicide/Self-Injury) |
| Adjustment disorder with depressed mood | Adjustment reaction with brief depressive reaction |
| Adjustment disorder with depressed mood | Adjustment reaction with prolonged depressive reaction |
| Adjustment disorder with mixed anxiety and depressed mood | Adjustment disorder with mixed anxiety and depressed mood |
| Agitated depression | Agitated depression |
| Agitated depression | Depression agitated |
| Anhedonia | Anhedonia |
| Anhedonia | Loss of all pleasure |
| Antidepressant therapy | Antidepressant therapy |
| Childhood depression | Childhood depression |
| Decreased interest | Decreased interest |
| Decreased interest | Loss of all interest |
| Decreased interest | Loss of interest |
| Decreased interest | Reduced interest in usual activities |
| Depressed mood | Chronic depressive mood |
| Depressed mood | Dejection emotional |
| Depressed mood | Depressed mood |
| Depressed mood | Emotional dejection |
| Depressed mood | Feeling blue |
| Depressed mood | Feeling down |
| Depressed mood | Feeling sad |
| Depressed mood | Low mood |
| Depressed mood | Mood depression |
| Depressed mood | Mood depressions |
| Depressed mood | Unhappiness |
| Depression Depression | Acute depression |
| Depression | Anxiety depression |
| Depression | Anxiodepressive syndrome |
| Depression | Anxious depression |
| Depression | Atypical depressive disorder |
| Depression | Brief depressive reaction |
| Depression | Chronic depression |
| Depression | Depressed reaction |
| Depression | Depressed state |
| Depression | Depression |
| Depression | Depression aggravated |
| Depression | Depression functional |
| Depression | Depression mental |
| | • |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SM | Q) (Exclude Suicide/Self-Injury) |
| Depression | Depression NOS |
| Depression | Depression reactive |
| Depression | Depression worsened |
| Depression | Depressive disorder |
| Depression | Depressive episode |
| Depression | Depressive illness |
| Depression | Depressive reaction |
| Depression | Depressive state |
| Depression | Depressive stupor |
| Depression | Exogenous depression |
| Depression | Mixed anxiety & depressive |
| Depression | Reactive depression |
| Depression | Recurrent depressive disorder |
| Depression | Unipolar depression |
| Depression | Unipolar depressive illness |
| Depression postoperative | Depression postoperative |
| Depression postoperative | Postoperative depression |
| Depressive symptoms | Depressive symptoms |
| Depressive symptoms | Depressive symptoms aggravvated |
| Dysphoria | Dysphoria |
| Dysthymic disorder | Chronic depressive personality disorder |
| Dysthymic disorder | Depression neurotic |
| Dysthymic disorder | Depressive neurosis |
| Dysthymic disorder | Depressive personality disorder |
| Dysthymic disorder | Dysthymia |
| Dysthymic disorder | Dysthymic disorder |
| Dysthymic disorder | Neurotic depression |
| Electroconvulsive therapy | Bilateral ECT |
| Electroconvulsive therapy | ECT |
| Electroconvulsive therapy | ECT (electro-convulsive therapy) |
| Electroconvulsive therapy | Electroconvulsive therapy |
| Electroconvulsive therapy | Modified ECT |
| Electroconvulsive therapy | Unilateral ECT |
| Electroconvulsive therapy | Unmodified ECT |
| Feeling guilty | Feeling guilty |
| Feeling guilty | Feeling remorse |
| Feeling of despair | Feeling of despair |
| Feelings of worthlessness | Feelings of worthlessness |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression | n (SMQ) (Exclude Suicide/Self-Injury) |
| Major depression | Depression endogenous |
| Major depression | Depression psychotic |
| Major depression | Depressive type psychosis |
| Major depression | Endogenous depression |
| Major depression | Involutional depression |
| Major depression | Involutional melancholia |
| Major depression | Major depression |
| Major depression | Major depressive disorder aggravated |
| Major depression | Major depressive disorder NOS |
| Major depression | Major depressive disorder with melancholic features |
| Major depression | Major depressive disorder, recurrent episode |
| Major depression | Major depressive disorder recurrent episode, in full remission |
| Major depression | Major depressive disorder, single episode |
| Major depression | Major depressive disorder, single episode in full remission |
| Major depression | Major depressive illness |
| Major depression | Melancholia |
| Major depression | Melancholic depression |
| Major depression | Psychosis depressive |
| Major depression | Psychotic depression |
| Menopausal depression | Depression perimenopausal |
| Menopausal depression | Depression postmenopausal |
| Menopausal depression | Menopausal depression |
| Menopausal depression | Postmenopausal depression |
| Post stroke depression | Post stroke depression |
| Postictal depression | Postictal depression |
| Postpartum depression | Baby blues |
| Postpartum depression | Depression puerperal |
| Postpartum depression | Postnatal blues |
| Postpartum depression | Postnatal depression (excl psychosis) |
| Postpartum depression | Postpartum depression |
| Postpartum depression | Puerperal depression |
| Postpartum depression | Transitory postpartum mood disturbance |
| Affect lability | Affect lability |
| Affect lability | Affective incontinence |
| Affect lability | Emotional incontinence |
| Affect lability | Emotional instability |
| Affect lability | Emotional lability |

| Alcohol poisoning | Preferred Term | Lowest Level Term |
|---|---|---|
| Affect lability Alcohol abuse Alcohol poisoning Acute alcoholic intoxication in alcoholism, continuou drinking behavior Acute alcoholic intoxication in alcoholism, episodic drinking behavior Acute alcoholic intoxication in alcoholism, in remission Alcohol poisoning Acute alcoholic intoxication in alcoholism, unspecific drinking behavior Acute alcoholic intoxication acute Alcohol poisoning Toxic effect of alcohol | Depression and Suicide/Self-Injury: Depression | n (SMQ) (Exclude Suicide/Self-Injury) |
| Affect lability Alcohol abuse Alcohol intoxication in alcoholism, episodic drinking behaviour Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol intoxication in alcoholism, unspecific drinking behaviour Alcohol poisoning Alcohol intoxication acute Alcohol intoxication Alcohol intoxication Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poi | Affect lability | Instability emotional |
| Affect lability Affect lability Affect lability Affect lability Affect lability Alcohol abuse Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Acute alcoholic intoxication in alcoholism, continuou drinking behavior Acute alcoholic intoxication in alcoholism, episodic drinking behavior Acute alcoholic intoxication in alcoholism, episodic drinking behavior Acute alcoholic intoxication in alcoholism, in remission Alcohol poisoning Acute alcoholic intoxication in alcoholism, unspecific drinking behavior Acute alcoholic intoxication in alcoholism, unspecific drinking behavior Acute alcoholic intoxication in alcoholism, unspecific drinking behavior Acute alcoholic intoxication in alcoholism, unspecific drinking behavior Acute alcoholic intoxication in alcoholism, unspecific drinking behavior Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol intoxication acute Alcohol poisoning Toxic effect of ethyl alcohol | Affect lability | Labile affect |
| Affect lability Pseudobulbar affect Alcohol abuse Alcohol poisoning | Affect lability | Lability emotional |
| Alcohol abuse Al | Affect lability | Mental lability symptom |
| Alcohol abuse Alcohol abuse Alcohol abuse Alcohol abuse, continuous drinking behavior Alcohol abuse Alcohol abuse, continuous drinking behavior Alcohol abuse Alcohol abuse, episodic drinking behavior Alcohol abuse Alcohol abuse, episodic drinking behavior Alcohol abuse Alcohol abuse, in remission Alcohol abuse Alcohol abuse, unspecified drinking behavior Alcohol abuse Alcohol abuse Alcohol abuse, unspecified drinking behavior Alcohol abuse Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Acute alcoholic intoxication in alcoholism, continuou drinking behavior Alcohol poisoning Acute alcoholic intoxication in alcoholism, episodic drinking behavior Alcohol poisoning Acute alcoholic intoxication in alcoholism, in remission Alcohol poisoning Acute alcoholic intoxication in alcoholism, unspecific drinking behavior Alcohol poisoning Acute alcoholic intoxication in alcoholism, unspecific drinking behavior Alcohol poisoning | Affect lability | Pseudobulbar affect |
| Alcohol abuse Alcohol abuse, continuous drinking behavior Alcohol abuse Alcohol abuse, episodic drinking behaviour Alcohol abuse Alcohol abuse, episodic drinking behaviour Alcohol abuse Alcohol abuse, episodic drinking behaviour Alcohol abuse Alcohol abuse, in remission Alcohol abuse, in remission Alcohol abuse, in remission Alcohol abuse, in remission Alcohol abuse, in remission Alcohol poisoning Acute alcoholic intoxication Acute alcoholic intoxication in alcoholism, continuou drinking behavior Alcohol poisoning Acute alcoholic intoxication in alcoholism, episodic drinking behavior Alcohol poisoning Acute alcoholic intoxication in alcoholism, in remission Alcohol poisoning Acute alcoholic intoxication in alcoholism, unspecific drinking behavior Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol intoxication acute Alcohol poisoning | Alcohol abuse | Alcohol abuse |
| Alcohol abuse Alcohol abuse, continuous drinking behaviour Alcohol abuse Alcohol abuse, episodic drinking behaviour Alcohol abuse Alcohol abuse, episodic drinking behaviour Alcohol abuse Alcohol abuse, in remission Alcohol abuse Alcohol abuse, unspecified drinking behaviour Alcohol abuse Alcohol abuse, unspecified drinking behaviour Alcohol abuse Alcohol abuse, unspecified drinking behaviour Alcohol abuse Alcohol abuse, unspecified drinking behaviour Alcohol abuse Alcohol abuse, unspecified drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, episodic drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, episodic drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, in remission Alcohol poisoning Acute alcoholic intoxication in alcoholism, unspecific drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, unspecific drinking behaviour Alcohol poisoning Alcohol poisoning Alcohol intoxication Alcohol poisoning Alcohol intoxication Alcohol poisoning Alcohol intoxication Alcohol poisoning | Alcohol abuse | Alcohol abuse chronic |
| Alcohol abuse Alcohol abuse, episodic drinking behavior Alcohol abuse Alcohol abuse, episodic drinking behaviour Alcohol abuse Alcohol abuse, in remission Alcohol abuse Alcohol abuse, unspecified drinking behavior Alcohol abuse Alcohol abuse, unspecified drinking behavior Alcohol abuse Alcohol abuse Alcohol abuse, unspecified drinking behaviour Alcohol abuse Alcohol abuse Alcohol abuse of alcohol Alcohol poisoning Acute alcoholic intoxication in alcoholism, episodic drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, episodic drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, in remission Alcohol poisoning Acute alcoholic intoxication in alcoholism, unspecific drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, unspecific drinking behaviour Alcohol poisoning | Alcohol abuse | Alcohol abuse, continuous drinking behavior |
| Alcohol abuse Alcohol poisoning Acute alcoholic intoxication in alcoholism, continuou drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, episodic drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, episodic drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, in remission Acute alcoholic intoxication in alcoholism, unspecific drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, unspecific drinking behaviour Alcohol poisoning Alcohol poisoning Alcohol intoxication Alcohol poisoning Alcohol intoxication Alcohol poisoning | Alcohol abuse | Alcohol abuse, continuous drinking behaviour |
| Alcohol abuse Alcohol poisoning Acute alcoholic intoxication in alcoholism, continuou drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, episodic drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, episodic drinking behaviour Alcohol poisoning Acute alcoholic intoxication in alcoholism, in remission Alcohol poisoning Acute alcoholic intoxication in alcoholism, unspecific drinking behaviour Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol intoxication Alcohol poisoning | Alcohol abuse | Alcohol abuse, episodic drinking behavior |
| Alcohol abuse Alcohol abuse, unspecified drinking behavior Alcohol abuse Alcohol abuse Alcohol abuse Alcohol abuse Alcohol abuse Alcohol abuse Alcohol abuse Alcohol poisoning Acute alcoholic intoxication Alcohol poisoning | Alcohol abuse | Alcohol abuse, episodic drinking behaviour |
| Alcohol abuse Alcohol abuse Nondependent abuse of alcohol Alcohol poisoning | Alcohol abuse | Alcohol abuse, in remission |
| Alcohol abuse Alcohol poisoning | Alcohol abuse | Alcohol abuse, unspecified drinking behavior |
| Alcohol poisoning | Alcohol abuse | Alcohol abuse, unspecified drinking behaviour |
| Alcohol poisoning Toxic effect of alcohol Toxic effect of ethyl alcohol | Alcohol abuse | Nondependent abuse of alcohol |
| Alcohol poisoning | Alcohol poisoning | Acute alcoholic intoxication |
| Alcohol poisoning Alcohol intoxication Alcohol intoxication acute Alcohol poisoning Toxic effect of alcohol Toxic effect of ethyl alcohol | | Acute alcoholic intoxication in alcoholism, continuous drinking behavior |
| Alcohol poisoning Toxic effect of alcohol Toxic effect of ethyl alcohol | Alcohol poisoning | Acute alcoholic intoxication in alcoholism, continuous drinking behaviour |
| Alcohol poisoning Toxic effect of alcohol Toxic effect of ethyl alcohol | Alcohol poisoning | Acute alcoholic intoxication in alcoholism, episodic drinking behavior |
| Alcohol poisoning Toxic effect of alcohol Toxic effect of ethyl alcohol | Alcohol poisoning | Acute alcoholic intoxication in alcoholism, episodic drinking behaviour |
| drinking behavior Alcohol poisoning Acute alcoholic intoxication in alcoholism, unspecified drinking behaviour Alcohol poisoning Alcohol intoxication Alcohol intoxication acute Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Drunkenness Alcohol poisoning Alcohol poisoning Toxic effect of alcohol Toxic effect of ethyl alcohol | Alcohol poisoning | reduce dicononic intoxication in dicononism, in |
| Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol intoxication Alcohol poisoning Alcohol intoxication acute Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Drunkenness Alcohol poisoning Alcohol poisoning Toxic effect of ethyl alcohol Toxic effect of ethyl alcohol | | Acute alcoholic intoxication in alcoholism, unspecified drinking behavior |
| Alcohol poisoning Alcohol intoxication Alcohol poisoning Alcohol intoxication acute Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Drunkenness Alcohol poisoning Toxic effect of alcohol Alcohol poisoning Toxic effect of ethyl alcohol | | Acute alcoholic intoxication in alcoholism, unspecified drinking behaviour |
| Alcohol poisoning Alcohol intoxication acute Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Drunkenness Alcohol poisoning Toxic effect of alcohol Alcohol poisoning Toxic effect of ethyl alcohol | Alcohol poisoning | |
| Alcohol poisoning Alcohol poisoning Alcohol poisoning Alcohol poisoning Drunkenness Alcohol poisoning Toxic effect of alcohol Alcohol poisoning Toxic effect of ethyl alcohol | - 0 | |
| Alcohol poisoning Alcohol poisoning Drunkenness Alcohol poisoning Toxic effect of alcohol Alcohol poisoning Toxic effect of ethyl alcohol | | |
| Alcohol poisoning Alcohol poisoning Toxic effect of alcohol Toxic effect of ethyl alcohol | | * |
| Alcohol poisoning Toxic effect of alcohol Alcohol poisoning Toxic effect of ethyl alcohol | | |
| Alcohol poisoning Toxic effect of ethyl alcohol | | |
| | 1 0 | |
| | Alcohol poisoning | Toxic effect of fusel oil |
| Alcohol poisoning Toxic effect of isopropyl alcohol | | |
| Alcohol poisoning Toxic effect of methyl alcohol | | |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SMC | (2) (Exclude Suicide/Self-Injury) |
| Alcohol poisoning | Toxic effect of unspecified alcohol |
| Alcohol problem | Alcohol problem |
| Alcohol problem | Alcohol problem NOS |
| Alcohol rehabilitation | Alcohol rehabilitation |
| Alcoholism | Alcohol addiction |
| Alcoholism | Alcohol craving |
| Alcoholism | Alcohol dependence syndrome |
| Alcoholism | Alcoholic relapse |
| Alcoholism | Alcoholism |
| Alcoholism | Alcoholism (excl psychosis) |
| Alcoholism | Chronic alcoholism |
| Alcoholism | Dipsomania |
| Apathy | Ambition loss of |
| Apathy | Apathy |
| Apathy | Avolition |
| Apathy | Initiative loss of |
| Apathy | Lack of motivation |
| Apathy | Loss of ambition |
| Apathy | Loss of initiative |
| Blunted affect | Affective blunting |
| Blunted affect | Blunted affect |
| Constricted affect | Constricted affect |
| Constricted affect | Restricted affect |
| Crying | Crying |
| Crying | Crying abnormal |
| Crying | Crying uncontrollable |
| Crying | High-pitched crying |
| Crying | Inconsolable crying |
| Crying | Persistent crying |
| Crying | Uncontrollable crying |
| Crying | Weeping |
| Crying | Weepy |
| Disturbance in attention | Attention concentration difficulty |
| Disturbance in attention | Attention impaired |
| Disturbance in attention | Attentiveness decreased |
| Disturbance in attention | Concentration (mental) abnormal |
| Disturbance in attention | Concentration ability impaired |
| Disturbance in attention | Concentration impaired |
| | ı |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression (SM | Q) (Exclude Suicide/Self-Injury) |
| Disturbance in attention | Concentration impairment |
| Disturbance in attention | Concentration loss |
| Disturbance in attention | Disturbance in attention |
| Disturbance in attention | Impairment of attention |
| Disturbance in attention | Mental concentration decreased |
| Disturbance in attention | Mental concentration difficult |
| Disturbance in attention | Mental concentration difficulty |
| Disturbance in attention | Mental concentration impaired |
| Disturbance in attention | Poor concentration |
| Disturbance in attention | Simple disturbance of activity and attention |
| Disturbance in attention | Vigilance decreased |
| Dyssomnia | Dysfunctions associated with sleep stages or arousal from sleep |
| Dyssomnia | Dyssomnia |
| Dyssomnia | Dyssomnia NOS |
| Emotional distress | Embarrassment |
| Emotional distress | Emotional distress |
| Emotional distress | Humiliation |
| Emotional distress | Mental distress |
| Emotional distress | Suffering |
| Emotional poverty | Emotional poverty |
| Emotional poverty | Emotional withdrawal |
| Emotional poverty | Lack of feeling emotions |
| Emotional poverty | Poverty emotional |
| Emotional poverty | Withdrawal emotional |
| Hypersomnia | Hypersomnia |
| Hypersomnia | Idiopathic hypersomnia |
| Hypersomnia | Persistent disorder of initiating or maintaining wakefulness |
| Hypersomnia | Primary hypersomnia |
| Hypersomina | Sleep excessive |
| Hypersonnia | Transient disorder of initiating or maintaining wakefulness |
| Hyposomnia | Hyposomnia |
| Impaired self-care | Impaired self-care |
| Initial insomnia | Initial insomnia |
| Initial insomnia | Trouble falling asleep |
| Intentional product misuse | Intentional drug misuse |
| Intentional product misuse | Intentional misuse |
| | • |

| Intentional product use issue | |
|---|---|
| Intentional product misuse Intentional product misuse Intentional product misuse Intentional product use issue Intentional use beyond labelled duration Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional use of illicit drugs Intentional use for unlabeled indication Intentional use of illicit drugs Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use beyond labeled administration Intentional use beyond labeled undication Inte | |
| Intentional product misuse Intentional product use issue Intentional use beyond labeled administration Intentional product use issue Intentional use beyond labeled administration Intentional product use issue Intentional use by incorrect pour Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Listless Listless Listless Maternal use of illicit drugs Maemal use of illicit drugs Maemal use of illicit drugs Memory impairment Memory | |
| Intentional product use issue Intentional use beyond labelled duration Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Listless Listless Listless Listless Maternal use of illicit drugs Mammal use of illicit drugs Memory impairment | |
| Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional use of illicit drugs Intentional use for unlabeled indication Intentional use beyond labeled duration Intentional use beyond labeled indication Intentional use beyond la | |
| Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional use of illicit drugs Intentional use for unlabeled indication Intentional use beyond labeled duration Intentional use beyond labeled indication Intentional use for unlabeled indication Intentional use for unl | *. |
| Intentional product use issue Intentional use beyond labeled administration Intentional product use issue Intentional use beyond labeled duration Intentional product use issue Intentional use beyond labelled administration Intentional product use issue Intentional use beyond labelled duration Intentional product use issue Intentional use by incorrect route Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional use of illicit drugs Intentional use for unlabeled indication Intentional use for unlabeled indica | :(0) |
| Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Listless Listless Listless Listless Maternal use of illicit drugs Memory impairment Memory impairment Memory impairment Memory deficit Memory impairment Memory disturbance Memory impairment | 13/ |
| Intentional product use issue Intentional use by incorrect route Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Listless Listless Listless Listless Maternal use of illicit drugs Memory impairment | duration |
| Intentional product use issue Intentional product use issue Intentional product use issue Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Listless Listless Listless Listless Maternal use of illicit drugs Memory impairment Memory imp | , |
| Intentional product use issue Intentional use beyond labelled duration Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Listless Listless Listless Listless Listless Maternal use of illicit drugs Memory impairment | n duration |
| Intentional product use issue Intentional use by incorrect route Intentional product use issue Intentional use for unlabeled indication Intentional product use issue Intentional use for unlabeled indication Listless Listless Listless Listless Maternal use of illicit drugs Memory impairment Middle insomnia Middle insomnia Middle insomnia Nocturnal awakening | |
| Intentional product use issue Intentional use for unlabeled indication Listless Listless Listless Listless Maternal use of illicit drugs Maternal use of illicit drugs Memory impairment Forgetfulness Memory impairment Memory deficit Memory impairment Memory deficit Memory impairment Memory disturbance Memory impairment Middle insomnia Arousal night Middle insomnia Middle insomnia Middle insomnia Nocturnal awakening | |
| Listless Listless Listless Maternal use of illicit drugs Memory impairment Middle insomnia Arousal night Middle insomnia Middle insomnia Middle insomnia Middle insomnia | |
| Listless Listless Listless Maternal use of illicit drugs Memory impairment Middle insomnia Arousal night Middle insomnia Middle insomnia Middle insomnia Middle insomnia | |
| Maternal use of illicit drugs Memory impairment Middle insomnia Middle insomnia Middle insomnia Middle insomnia Middle insomnia | |
| Maternal use of illicit drugs Memory impairment Middle insomnia Middle insomnia Middle insomnia Middle insomnia Middle insomnia | |
| Memory impairmentForgetfulnessMemory impairmentHypomnesiaMemory impairmentMemory deficitMemory impairmentMemory disturbanceMemory impairmentMemory disturbance (excl dementia)Memory impairmentMemory impairmentMemory impairmentMemory impairmentMemory impairmentShort-term memory impairmentMiddle insomniaArousal nightMiddle insomniaMiddle insomniaMiddle insomniaNocturnal awakening | |
| Memory impairment Memory impairment Memory impairment Memory impairment Memory disturbance Memory disturbance (excl dementia) Memory impairment Middle insomnia Middle insomnia Middle insomnia Middle insomnia Nocturnal awakening | |
| Memory impairment Memory impairment Memory deficit Memory disturbance Memory disturbance (excl dementia) Memory impairment Arousal night Middle insomnia Middle insomnia Middle insomnia Nocturnal awakening | |
| Memory impairment Arousal night Middle insomnia Middle insomnia Middle insomnia Middle insomnia Nocturnal awakening | |
| Memory impairment Memory impairment Memory impairment Memory impairment Memory impairment Short-term memory impairment Middle insomnia Middle insomnia Middle insomnia Nocturnal awakening | |
| Memory impairment Memory impairment Short-term memory impairment Middle insomnia Middle insomnia Middle insomnia Nocturnal awakening | |
| Memory impairment Middle insomnia Middle insomnia Middle insomnia Middle insomnia Nocturnal awakening | |
| Memory impairment Middle insomnia Middle insomnia Middle insomnia Middle insomnia Nocturnal awakening | |
| Middle insomnia Middle insomnia Nocturnal awakening | |
| Middle insomnia Nocturnal awakening | |
| Middle insomnia Sleep maintenance insomnia | |
| Mood altered Affect alteration | |
| Mood altered Affect altered | |
| Mood altered Altered mood | |
| Mood altered Bad mood | |
| Mood altered Mood alteration NOS | |
| Mood altered Mood altered | |
| Mood altered Mood change | |
| Mood swings Mood swings | |
| Mood swings Mood variable | |
| Morose Morose | |

| Neglect of personal appearance Neglect of personal appearance Neglect of personal appearance Neglect of personal appearance Poor quality sleep Sleep restless Poor quality sleep Poor quality sleep Poor quality sleep Poor quality sleep Posychomotor hyperactivity Psychomotor hyperacti | ida/Salf_Injury) |
|---|---|
| Negative thoughts Neglect of personal appearance Personal appearance Poor quality sleep Sleep restless Poor quality sleep Poor qua | iuc/Scii-iiijui y) |
| Neglect of personal appearance Poor quality sleep Sleep restless Poor quality sleep Psychomotor hyperactivity Psychomot | |
| Neglect of personal appearance Neglect of personal appearance Neglect of personal appearance Neglect of personal appearance Poor quality sleep Sleep restless Poor quality sleep Psychomotor hyperactivity Psychomotor hy | hts |
| Neglect of personal appearance Personal appearance Poor quality sleep Psychomotor hyperactivity Psychomotor hyper | rsonal neglect of |
| Neglect of personal appearance Poor quality sleep Poor sleep Wakefulness Psychomotor hyperactivity Motor activity of Muscular hyperactivity | on appearance . |
| Neglect of personal appearance Poor quality sleep Poor sleep Poor quality sleep Poor sleep Poor quality sleep Sleep restless Paulity motor Psychomotor hyperactivity Psychomotor hypera | onal appearance |
| Poor quality sleep Poor quality sleep Poor quality sleep Poor quality sleep Poor quality sleep Sleep restless Poor quality sleep Sleep unwell Poor quality sleep Wakefulness Psychomotor hyperactivity Motor activity of Muscular hyperactivity Psychomotor hyperactivity | rance neglect of |
| Poor quality sleep Poor quality sleep Sleep restless Poor quality sleep Sleep unwell Poor quality sleep Wakefulness Psychomotor hyperactivity Psychomotor hyperactivity Psychomotor hyperactivity Behaviour hyper Psychomotor hyperactivity Motor activity of Muscular hyperactivity Psychomotor hyperactivity Muscular hyperactivity | SO, |
| Poor quality sleep Poor quality sleep Poor quality sleep Poor quality sleep Poor quality sleep Psychomotor hyperactivity Motor activity of Muscular hyperactivity Muscular hyperactivity | ep ;oll |
| Poor quality sleep Poor quality sleep Poor quality sleep Psychomotor hyperactivity Motor activity of Muscular hyperactivity Psychomotor hyperactivity Muscular hyperactivity | "SUS" |
| Poor quality sleep Psychomotor hyperactivity Motor activity of Muscular hyperactivity Muscular hyperactivity | ot o |
| Psychomotor hyperactivity Motor activity of Muscular hyperactivity Psychomotor hyperactivity Muscular hyperactivity | tm |
| Psychomotor hyperactivity Motor activity of Muscular hyperactivity Muscular hyperactivity | 20.0 |
| Psychomotor hyperactivity Motor activity of Muscular hyperactivity Psychomotor hyperactivity Psychomotor hyperactivity Muscular hyperactivity | exaggerated |
| Psychomotor hyperactivity Motor activity Psychomotor hyperactivity Muscular hyperactivity | |
| Psychomotor hyperactivity Motor activity of Muscular hyperactivity | - U |
| Psychomotor hyperactivity Motor activity Psychomotor hyperactivity Muscular hyperactivity | |
| Psychomotor hyperactivity Psychomotor hyperactivity Psychomotor hyperactivity Psychomotor hyperactivity Psychomotor hyperactivity Motor activity Psychomotor hyperactivity Muscular hyperactivity | |
| Psychomotor hyperactivity Psychomotor hyperactivity Psychomotor hyperactivity Motor activity of Muscular hyperactivity | ity |
| Psychomotor hyperactivity Muscular hyper | |
| | exaggerated |
| . (8) | ractivity |
| Psychomotor hyperactivity Overactive | - |
| Psychomotor hyperactivity Overactivity | |
| Psychomotor hyperactivity Psychomotor ag | gitation |
| Psychomotor hyperactivity Psychomotor es | ceitability |
| Psychomotor hyperactivity Psychomotor hyperactivity | yperactivity |
| Psychomotor retardation Psychomotor re | tardation |
| Psychosocial support Psychosocial co | ounseling |
| Psychosocial support Psychosocial su | |
| Psychotherapy Art therapy | |
| Psychotherapy Cognitive psycl | notherapy |
| Psychotherapy Couples psycho | otherapy |
| Psychotherapy Family psychot | herapy |
| Psychotherapy Group psychoth | |
| Psychotherapy Hippotherapy | |
| Psychotherapy Interpersonal ps | sychotherapy |
| Psychotherapy Play therapy | |
| Psychotherapy Psychotherapy | |

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Depression ( | SMQ) (Exclude Suicide/Self-Injury) |
| Psychotherapy | Supportive psychotherapy |
| Self esteem decreased | Self esteem decreased |
| Substance-induced mood disorder | Stimulant-induced mood disorder |
| Substance-induced mood disorder | Substance-induced mood disorder |
| Tearfulness | Tearfulness |
| Terminal insomnia | Awakening early |
| Terminal insomnia | Early morning awakening |
| Terminal insomnia | Terminal insomnia |

AEs Related to Depression and Suicidality/Self-Injury-Suicide/Self-Injury **Table 18:** (SMQ)

| Preferred Term | Lowest Level Term |
|---|---|
| Depression and Suicide/Self-Injury: Suicide/Self-Injury | |
| Columbia suicide severity rating scale abnormal | Columbia suicide severity rating scale abnormal |
| Completed suicide | Accomplished suicide |
| Completed suicide | Completed suicide |
| Completed suicide | Suicide |
| Completed suicide | Suicide (accomplished) |
| Depression suicidal | Depression suicidal |
| Depression suicidal | Suicidal depression |
| Depression suicidal Depression suicidal Intentional overdose | Deliberate overdose |
| Intentional overdose | Drug overdose deliberate self-inflicted |
| Intentional overdose | Intentional overdose |
| Intentional overdose | Multiple drug overdose intentional |
| Intentional overdose | Non-accidental overdose |
| Intentional overdose | Overdose deliberate self-inflicted |
| Intentional overdose | Overdose intentional |
| Intentional self-injury | Deliberate self-harm |
| Intentional self-injury | Deliberate self-injury |
| Intentional self-injury | Intentional self-injury |
| Intentional self-injury | Parasuicide |
| Intentional self-injury | Repeated parasuicide |
| Intentional self-injury | Self inflicted laceration |
| Intentional self-injury | Self mutilation |
| Attempted suicide | Deliberate poisoning |
| Attempted suicide | Poisoning deliberate |
| Poisoning deliberate | Poisoning deliberate |

| Depression and Suicide/Self-Injury: Suicide/Self-Injury (SMQ) Poisoning deliberate Self injurious behaviour Self-injurious behaviour Self-injurious ideation Self-injurious ideation Self-injurious ideation Suicidal behaviour Suicidal ideation | ent |
|---|---|
| Self injurious behaviour Self injurious behaviour Self-injurious ideation Self-injurious ideation Self-injurious ideation Thoughts of self harm Preparatory actions toward imminent suicidal behaviour Suicidal ideation Suicidal ideation | ent |
| Self injurious behaviour Self-injurious ideation Self-injurious ideation Self-injurious ideation Thoughts of self harm Suicidal behaviour Preparatory actions toward imminent suicidal behaviour Suicidal ideation | ent |
| Self injurious behaviour Self injurious behaviour Self injurious behaviour Self injurious behaviour Self-injurious ideation Self-injurious ideation Self-injurious ideation Thoughts of self harm Suicidal behaviour Preparatory actions toward imminent suicidal behaviour Suicidal ideation Suicidal intention | nt |
| Self injurious behaviour Self-injurious ideation Self-injurious ideation Self-injurious ideation Thoughts of self harm Suicidal behaviour Preparatory actions toward imminent suicidal behaviour Suicidal ideation Suicidal ideation | |
| Self-injurious ideation Self-injurious ideation Thoughts of self harm Suicidal behaviour Preparatory actions toward imminent suicidal Suicidal behaviour Suicidal ideation | |
| Self-injurious ideation Suicidal behaviour Preparatory actions toward imminent suicidal behaviour Suicidal ideation Suicidal ideation | tent |
| Suicidal behaviour Suicidal ideation | 1/5 |
| Suicidal behaviour Suicidal ideation Suicidal intention | 20, |
| Suicidal behaviour Suicidal behaviour Suicidal behaviour Suicidal behaviour Suicidal behaviour Suicidal ideation Suicidal ideation Suicidal ideation Suicidal ideation Suicidal ideation Suicidal ideation Suicidal ideation Suicidal ideation | al behav |
| Suicidal behaviour Suicidal behaviour Suicidal behaviour Suicidal ideation Suicidal ideation Suicidal ideation Suicidal ideation Suicidal ideation Life weariness Suicidal ideation | al |
| Suicidal behaviour Suicidal ideation Active suicidal ideation Suicidal ideation Death wishes Suicidal ideation Life weariness Suicidal ideation | |
| Suicidal ideation Suicidal ideation Death wishes Suicidal ideation Life wearings Suicidal ideation Passive suicidal ideation Suicidal intention | |
| Suicidal ideation Suicidal ideation Life weariness Suicidal ideation Suicidal intention | |
| Suicidal ideation | |
| Suicidal ideation | |
| Suicidal ideation Suicidal ideation Suicidal intention Suicidal ideation | |
| Suicidal ideation Suicidal ideation Suicidal intention Suicidal ideation | |
| 0::11:1 | |
| Suicidal ideation Suicidal plans Suicidal ideation Suicidal tendency Suicide attempt Attempted suicide | |
| Suicidal ideation Suicidal tendency Suicide attempt Attempted suicide | |
| Suicide attempt Attempted suicide | |
| Suicide attempt Suicide attempt | |
| Suicide attempt other than overdose | |
| Suicide attempt Unsuccessful suicide | |
| Suicide attempt Unsuccessful suicide Unsuccessful suicide | |